### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for Protocol 207966: Study<br>Evaluating the Efficacy, Safety, and Tolerability of Long-<br>acting Cabotegravir Plus Long-acting Rilpivirine<br>administered every 8 weeks in Virologically Suppressed<br>HIV-1-infected Adults |
| <b>Compound Number</b> | : | GSK1265744 |
| Effective Date | : | 17-JAN-2019 |

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 207966
- This RAP will be provided to the study team members to convey the content of the Week 24/Week 48/Week 96/End of Study: Statistical Analysis Complete (SAC) deliverable.

# Author(s)

| Author | | Date |
|---|---|---|
| Lead | | |
| | | 15-JAN-2019 |
| Principal Statistici | an (Infectious Diseases, Clinical Statistics) | |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Review Confirmations**

(Method: E-mail)

| Reviewer | Date |
|---|---|
| Clinical Development Director (ViiV Healthcare) | 16-JAN-2019 |
| PPD PPD | |
| Clinical Development Director (ViiV Healthcare) | 15-JAN-2019 |
| PPD | |
| Manager, Programming (Infectious Diseases, Clinical Programming) | 15-JAN-2019 |
| PPD | 16-JAN-2019 |
| SERM Director (CMO GCSP SERM) | 10-JAIN-2019 |
| Director, Clinical Pharmacology (Clinical Pharmacology CPKMS) | 16-JAN-2019 |
| PPD | |
| Clinical Development Manager (Translational Medicine, ViiV Sci Med Office) | 16-JAN-2019 |
| PPD | |
| Manager, Health Outcomes, ViiV Sci Med Office) | 16-JAN-2019 |

# Clinical Statistics and Clinical Programming Line Approvals: (Method: Pharma TMF eSignature)

| Approver | Date |
|---|---|
| PPD | |
| Manager, Statistics (Infectious Diseases, Clinical Statistics) Delegated by PPD | 17-JAN-2019 |
| Director, Statistics (Infectious Diseases, Clinical Statistics) | |
| Director, Programming (Infectious Diseases, Clinical Programming) | 17-JAN-2019 |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 7 |
| 2. | SUM | MARY OF KEY PROTOCOL INFORMATION | 8 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | |
| 3. | PLAN | NED ANALYSES | 13 |
| | 3.1. | IDMC Analyses | |
| | 3.2. | Final Analyses | 14 |
| 4. | | YSIS POPULATIONS | |
| | 4.1. | Protocol Deviations | 15 |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | 47 |
| | | /ENTIONS | |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | |
| | 5.3.<br>5.4. | Multicentre Studies | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | |
| | | 5.4.1. Covariates and Other Strata | |
| | 5.5. | | |
| | 5.5. | Multiple Comparisons and Multiplicity | |
| | | <ul><li>5.5.1. Primary Comparison of Interest</li><li>5.5.2. Other Comparisons of Interest</li></ul> | |
| | 5.6. | Other Considerations for Data Analyses and Data Handling | 22 |
| | 5.0. | Conventions | 22 |
| 6. | STUD | OY POPULATION ANALYSES | 23 |
| ٥. | 6.1. | Overview of Planned Study Population Analyses | |
| | 6.2. | Prior and Concomitant Medications | 25 |
| _ | | | |
| 7. | | CACY ANALYSES | |
| | 7.1. | Primary Efficacy Analyses | |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | |
| | | 7.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.1.5. Statistical Analyses / Methods | |
| | 7.0 | 7.1.5.1. Statistical Methodology Specification | |
| | 7.2. | Secondary Efficacy Analyses | |
| | | 7.2.1. Endpoints | |
| | | 7.2.2. Summary Measure | |
| | | 7.2.3. Population of Interest | |
| | | 7.2.4. Strategy for Intercurrent (Post-Randomization) Events 7.2.5. Statistical Analyses / Methods | |
| | | 7.2.5. Statistical Analyses / Methods | |
| | | 1,4,5,1, | |

| | 7.3. | Exploratory Efficacy Analyses | 32 |
|---|---|---|---|
| 8. | SAFE | TY ANALYSES | 34 |
| | 8.1. | Adverse Events Analyses | 34 |
| | | 8.1.1. Analyses for Injection Site Reaction Adverse Events from | |
| | | Study Drug Injection | |
| | 8.2. | Adverse Events of Special Interest Analyses | |
| | 8.3. | Clinical Laboratory Analyses | |
| | 8.4. | Other Safety Analyses | 36 |
| 9. | PHAR | MACOKINETIC ANALYSES | 37 |
| | 9.1. | Endpoint / Variables | |
| | | 9.1.1. Drug Concentration Measures | |
| | 9.2. | Overview of Planned Analyses | |
| | 9.3. | Statistical Analyses / Methods | 38 |
| 10. | POPU | LATION PHARMACOKINETIC ANALYSES | 38 |
| 11. | PHAR | MACOKINETIC / PHARMACODYNAMIC ANALYSES | 38 |
| | 11.1. | Overview of Planned Analyses | 39 |
| | 11.2. | Statistical Analyses / Methods | 39 |
| 12. | HEAL | TH OUTCOMES ANALYSES | 40 |
| | 12.1. | Endpoint / Variables | |
| | 12.2. | Summary Measure | 41 |
| | 12.3. | Population of Interest | 41 |
| | 12.4. | Strategy for Intercurrent (Post-Randomization) Events | 41 |
| | 12.5. | Statistical Analyses / Methods | |
| | | 12.5.1. Statistical Methodology Specification | 42 |
| 13. | VIROL | .OGY | 44 |
| 14 | RFFF | RENCES | 45 |
| 15. | | NDICES | 46 |
| | 15.1. | Appendix 1: Protocol Deviation Management and Definitions for Per | 46 |
| | | Protocol Population | |
| | 15.0 | 15.1.1. Exclusions from Per Protocol Population | |
| | 15.2. | 15.2.1. Protocol Defined Schedule of Events for Q4W Arm | |
| | | 15.2.1. Protocol Defined Schedule of Events for Q4W Arm | |
| | 15.3. | Appendix 3: Assessment Windows | |
| | 13.3. | 15.3.1. Definitions of Assessment Windows for Analyses | |
| | | 15.3.2. Definitions of Assessment Windows for Analyses | 00 |
| | | than Health Outcome and PK | 67 |
| | | 15.3.3. Assessment Window for Phase Conclusion | <mark>70</mark> |
| | | 15.3.4. Assessment Window for Health Outcome Data | <mark>70</mark> |
| | | 15.3.4.1. PIN / HAT-QoL / HIVTSQs / HIVTSQc / | |
| | | ACCEPT / Preference | |
| | | 15.3.4.2. Reasons for Continuation/Switch | |
| | | 15.3.5. Assessment Window for PK Concentration Data | |
| | | 15.3.6. Multiple Assessments within an Assessment Window | |
| | 15.4. | Appendix 4: Study Phases and Treatment State | 74 |

| | 15.4.1. | Study Phases | .74 |
|---|---|---|---|
| | | Treatment State | |
| | | 15.4.2.1. Treatment States for AE Data | |
| | 15.4.3. | Study Period | .77 |
| 15.5. | <b>Appendix</b> | 5: Data Display Standards & Handling Conventions | .79 |
| | 15.5.1. | Reporting Process | |
| | 15.5.2. | Reporting Standards | |
| | 15.5.3. | Reporting Standards for Pharmacokinetic | .80 |
| 15.6. | <b>Appendix</b> | 6: Derived and Transformed Data | |
| | 15.6.1. | General | .81 |
| | 15.6.2. | Study Population | .82 |
| | 15.6.3. | Efficacy | .84 |
| | 15.6.4. | Safety | .87 |
| | 15.6.5. | Pharmacokinetic | .92 |
| | 15.6.6. | Health Outcomes | .93 |
| | | Virology | |
| 15.7. | | 7: Reporting Standards for Missing Data | |
| | | Premature Withdrawals | |
| | 15.7.2. | Handling of Missing Data | |
| | | 15.7.2.1. Handling of Missing and Partial Dates | |
| | | 15.7.2.2. Handling of Missing data for Statistical Analysis | |
| 15.8. | | 8: Values of Potential Clinical Importance | |
| 15.9. | | 9: Snapshot Algorithm Details | |
| | | 10: Variables Defined for Time to Event Analysis | |
| | | 11: Identification of Adverse Events of Special Interest | |
| 15.12. | | 12: IDMC | |
| | | Adhoc CVF IDMC Analyses | |
| 15 40 | 15.12.2. | Week 24 IDMC Analyses | 135 |
| 15.13. | | 13: Abbreviations & Trademarks | |
| | | Abbreviations | |
| 15 11 | | Trademarks | |
| 15.14. | | 14: List of Data Displays | |
| | | Data Display Numbering | |
| | | Deliverables | |
| | | List of Data Displays for Week 24 IDMC and Week 24 | 139 |
| | 13.14.4. | Planned Analyses | 140 |
| | | 15.14.4.1. Study Population Tables | 140<br>141 |
| | | 15.14.4.2. Efficacy Tables | |
| | | 15.14.4.3. Efficacy Figures | |
| | | 15.14.4.4. Safety Tables | |
| | | 15.14.4.5. Safety Figures | |
| | | 15.14.4.6. Pharmacokinetic Tables | |
| | | 15.14.4.7. Pharmacokinetic Figures | |
| | | 15.14.4.8. Virology Tables | |
| | | 15.14.4.9. ICH Listings | |
| | | 15.14.4.10. Non-ICH Listings | |
| | 15.14.5. | List of Data Displays for Week 48/96/End-of-Study | |
| | | Planned Analyses | 157 |
| | | 15.14.5.1. Study Population Tables | |
| | | 15.14.5.2. Efficacy Tables | |
| | | 15.14.5.3. Efficacy Figures | |

# 2019N406358\_00 207966

| 15.14.5.4. Safety Tables | 171 |
|-----------------------------------------------------------|-----|
| 15.14.5.5. Safety Figures | |
| 15.14.5.6. Pharmacokinetic Tables | |
| 15.14.5.7. Pharmacokinetic Figures | 186 |
| 15.14.5.8. Pharmacokinetic / Pharmacodynamic Tables | 188 |
| 15.14.5.9. Pharmacokinetic / Pharmacodynamic Figures | 189 |
| 15.14.5.10. Health Outcomes Tables | 192 |
| 15.14.5.11. Health Outcomes Figures | 200 |
| 15.14.5.12. Virology Tables | 202 |
| 15.14.5.13. ICH Listings | 204 |
| 15.14.5.14. Non-ICH Listings | 210 |
| 15.15. Appendix 15: Example Mock Shells for Data Displays | 214 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|---|---|---|
| 2017N326521_00 | 17-JUL-2017 | Original |
| 2017N326521_01 | 14-SEP-2017 | The primary purpose of protocol amendment # 1 is to revise the study sample size to randomize approximately 1020 participants including 510 participants per arm based on a non-inferiority margin of 4% between the CAB LA + RPV LA Q8W and Q4W arms. |
| 2017N326521_02 | 03-Jul-2018 | The primary reasons for amendment #2 are to: |
| | | <ul> <li>Add the additional interim analysis of data when all<br/>subjects have completed the Week 24 visit, with the<br/>intent of expediting the submission of study results to<br/>Health Authorities;</li> </ul> |
| | | Change the objective for assessing the preference for CAB LA + RPV LA every 8 weeks or CAB LA + RPV LA every 4 weeks LA compared to oral antiretroviral (ARV) and the preference for CAB LA + RPV LA every 8 weeks compared to CAB LA + RPV LA every 4 weeks from an exploratory objective to a secondary objective. A change to the supporting version of the Preference questionnaire administered to participants at Week 48 (or withdrawal) is also acknowledged; |
| | | <ul> <li>Add revisions and clarifications for the administration<br/>of health outcomes questionnaires;</li> </ul> |
| | | <ul> <li>Extend exclusion criterion #28 to also exclude<br/>hereditary coagulation and platelet disorders such as<br/>haemophilia or Von Willebrand Disease;</li> </ul> |
| | | <ul> <li>Update exclusion criterion #11 to indicate that CD4+<br/>counts &lt;200 cells/µL are not exclusionary;</li> </ul> |
| | | <ul> <li>Offer clarification that withdrawal assessments will be<br/>performed for any participant who withdraws<br/>prematurely from the Maintenance or Extension<br/>Phase. Additional guidance for participants<br/>withdrawing at Week 52 or Week 100 has been<br/>added;</li> </ul> |
| | | <ul> <li>Offer guidance to monitor medications that are<br/>dependent on OAT1 and OAT3 transport upon<br/>concomitant exposure with CAB;</li> </ul> |
| | | <ul> <li>Specify that 2-hour post-dose ECG should be<br/>performed at Day 1 and Week 48 only for<br/>participants receiving CAB LA + RPV LA as it is not<br/>required to perform 2-hour post-dose ECG for those<br/>receiving oral CAB + RPV at Day 1;</li> </ul> |

| Revision Chronology: | |
|---|---|
| | <ul> <li>Exclude language that previously indicated hormonal contraception may be susceptible to interaction with the study drugs. The lack of a demonstrated interaction with a representative contraceptive supports use of CAB and RPV across a broad range of estrogen and progestin or progestin only hormonal contraceptives;</li> <li>Add minor clarifications and corrections to typographical errors/formatting to protocol text.</li> </ul> |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 2 [(Dated: 03/JUL/2018)].

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To demonstrate the non-inferior<br>antiviral activity of CAB LA + RPV LA<br>every 8 weeks (every two months)<br>compared to CAB LA + RPV LA every<br>4 weeks (monthly) over 48 weeks in<br>suppressed HIV-1 infected<br>antiretroviral therapy (ART)-<br>experienced participants | Proportion of participants with plasma HIV-RNA greater than or equal to 50 copies/mL as per Food and Drug Administration (FDA) Snapshot algorithm at Week 48 (Intent-to-Treat Exposed [ITT-E] population) |
| Secondary Objectives | Secondary Endpoints |
| To demonstrate the antiviral and immunologic activity of CAB LA + RPV LA every 8 weeks compared to CAB LA + RPV LA every 4 weeks | <ul> <li>Proportion of participants with plasma HIV-1 RNA &lt;50 c/mL (c/mL) at Week 24, Week 48 and Week 96 using the FDA Snapshot algorithm (Intent-to-Treat Exposed [ITT-E] population)</li> <li>Proportion of participants with protocol-defined confirmed virologic failure (CVF) through Week 24, Week 48 and Week 96</li> <li>Proportion of participants with HIV-RNA greater than or equal to 50 c/mL as per FDA Snapshot algorithm at Week 24 and Week 96</li> <li>Absolute values and changes from Baseline in viral load and CD4+ cell counts over time including Week 48 and Week 96</li> </ul> |
| To evaluate the safety and tolerability<br>of CAB LA + RPV LA every 8 weeks<br>compared to CAB LA + RPV LA every | <ul> <li>Incidence and severity of AEs and laboratory<br/>abnormalities over time including Week 24, Week 48 and<br/>Week 96</li> </ul> |
| 4 weeks | <ul> <li>Proportion of participants who discontinue treatment due<br/>to AEs over time including Week 24, Week 48 and Week</li> </ul> |

| Objectives | Endpoints |
|---|---|
| | 96 |
| | <ul> <li>Change from Baseline in laboratory parameters over time<br/>including Week 48 and Week 96</li> </ul> |
| To assess viral resistance in participants experiencing protocoldefined confirmed virologic failure | <ul> <li>Incidence of treatment emergent genotypic and<br/>phenotypic resistance to CAB, RPV through Week 24,<br/>Week 48 and Week 96</li> </ul> |
| To characterize CAB and RPV concentrations and population pharmacokinetics and identify | <ul> <li>Plasma PK parameters for CAB LA and RPV LA (when<br/>evaluable, Ctrough, concentrations post dose [~Cmax],<br/>and area under the curve [AUC])</li> </ul> |
| important determinants of variability | <ul> <li>Demographic parameters including, but not limited to,<br/>age, sex, race, body weight, body mass index, and<br/>relevant laboratory parameters will be evaluated as<br/>potential predictors of inter- and intra-participant<br/>variability for pharmacokinetic parameters</li> </ul> |
| <ul> <li>To assess preference for CAB LA + RPV LA every 8 weeks or CAB LA + RPV LA every 4 weeks LA compared to oral antiretroviral (ARV)</li> <li>To assess preference for CAB LA+ RPV LA every 8 weeks compared to CAB LA + RPV LA every 4 weeks</li> </ul> | <ul> <li>Preference for CAB LA + RPV LA every 8 weeks and<br/>CAB LA + RPV LA every 4 weeks compared to oral ARV<br/>and preference for CAB LA + RPV LA every 8 weeks<br/>compared to CAB LA + RPV LA every 4 weeks will be<br/>assessed using a preference questionnaire at week 48<br/>(or Withdrawal).</li> </ul> |
| To assess patient reported health-related quality of life, treatment satisfaction, injection tolerability, and treatment acceptance. | <ul> <li>Change from Baseline (Day 1) in HRQoL at Week 24, and Week 48 (or Withdrawal)</li> <li>Change from baseline (Day 1) in total "treatment satisfaction" score, and individual item scores of the HIV Treatment Satisfaction Status Questionnaire (HIVTSQs) at Week 24, and 48, (or Withdrawal)</li> <li>Change in treatment satisfaction over time using the HIV Treatment Satisfaction Change Questionnaire HIVTSQc at Week 48 (or Withdrawal).</li> <li>Change from Week 8 in Dimension scores ("Colored In Individual item scores assessing pain during injection, anxiety before and after injection, willingness to be injected in the future and overall satisfaction with mode of administration over time will be assessed using the Perception of Injection questionnaire (PIN) at Weeks 24, and 48 (or Withdrawal)</li> <li>Change from Baseline (Day 1) in treatment acceptance at Week 24 and Week 48 (or Withdrawal) will be assessed using the "General acceptance" dimension of the Chronic Treatment Acceptance (ACCEPT) questionnaire</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To evaluate the antiviral and immunologic effects, safety and tolerability, and viral resistance of CAB LA + RPV LA for all participants in the Extension Phase. | <ul> <li>Proportion of participants with plasma HIV-1 RNA &lt;50 c/mL over time</li> <li>Proportion of participants with confirmed virologic failure over time</li> <li>Incidence of treatment emergent genotypic and phenotypic resistance to CAB and RPV in over time</li> <li>Incidence and severity of AEs and laboratory</li> </ul> |

| Objectives | Endpoints |
|---|---|
| | <ul> <li>abnormalities over time</li> <li>Proportion of participants who discontinue treatment due to AEs over time</li> <li>Absolute values and changes in laboratory parameters over time</li> <li>Incidence of disease progression (HIV-associated conditions, acquired immunodeficiency syndrome [AIDS] and death)</li> </ul> |
| To explore the effect of patient<br>characteristics on virologic and<br>immunologic responses to CAB LA+<br>RPV LA every 8 weeks compared to<br>CAB LA + RPV LA every 4 weeks | <ul> <li>Proportion of participants by patient subgroup(s) (e.g., by age, gender, BMI, race, HIV-1 subtype, Baseline CD4+, type of oral treatment [NNRTI, PI, or INSTI], duration prior CAB LA and RPV LA exposure [0 weeks, 1-24 weeks, &gt; 24 weeks]) with HIV-RNA greater than or equal to 50 c/mL, and with protocol-defined confirmed virologic failure over time including Week 48 and Week 96 using the Snapshot algorithm for the ITT-E population</li> <li>Change from Baseline in CD4+ cell counts by subgroups at Week 48 and Week 96</li> </ul> |
| To explore relationship(s) between<br>plasma concentrations of CAB and<br>RPV and pharmacodynamic<br>endpoints. | Relationship between plasma CAB and RPV concentrations and virologic, immunologic responses, and/or occurrence of adverse events [AEs] over time. |
| <ul> <li>To assess reason for switching using a single question.</li> <li>To assess reason for continuation using a single question</li> </ul> | <ul> <li>For patients randomized from oral SOC, the reasons for willingness to switch ART at baseline (Day 1) will be assessed</li> <li>For patients randomized from CAB LA + RPV LA every 4 weeks in ATLAS, the reasons for willingness to continue long-acting ART at baseline (Day 1) will be assessed</li> </ul> |

# 2.3. Study Design



N=1020, randomized 1:1 to each arm and stratified by prior CAB+RPV Exposure

# SOC Patients not transitioning from the ATLAS study must be on uninterrupted current regimen (either the initial or second cART regimen) for at least 6 months prior to Screening. Documented evidence of at least two plasma HIV-1 RNA measurements <50 c/mL in the 12 months prior to Screening: one within the 6 to 12 month window, and one within 6 months prior to Screening. No history of virologic failure. No evidence of viral resistance based on the presence of any resistance-associated major INI, or NNRTI mutation (except K103N) from prior genotype assay results. No current or prior history of etravirine use.

†Optional Extension Phase to continue randomized CAB LA + RPV LA Q4W or Q8W at Wk 100 ¥Participants who withdraw from IM arm must go into 52 week long term follow up phase if randomized regimen is not yet locally approved and commercially available.

| Design<br>Features | <ul> <li>Study 207966 (Antiretroviral Therapy as Long Acting Suppression every 2 Months-ATLAS-2M) is a Phase IIIb, randomized, open-label, active-controlled, multicenter, parallel-group, non-inferiority study designed to assess the antiviral activity and safety of CAB LA + RPV LA administered every 4 weeks compared CAB LA + RPV LA administered every 8 weeks in approximately 1020 adult HIV-1 infected patients.</li> <li>The ATLAS-2M study comprises a Screening Phase (up to 35 days), and a Maintenance Phase (Day 1 to Week 100), followed by an Extension Phase (post Week 96). Additionally, any participant who receives at least a single dose of CAB LA and/or RPV LA and discontinues the CAB LA + RPV LA regimen will enter the Long-term Follow-up Phase and will initiate highly active antiretroviral therapy (HAART) for 52 weeks after the last dose of CAB LA and/or RPV LA, or until the assigned CAB LA + RPV LA regimen is locally approved and commercially available.</li> <li>Two groups of patients who fulfill eligibility requirements will be randomized (1:1) at Day 1 to receive CAB LA + RPV LA Q4W, or CAB LA + RPV LA Q8W regimen for at least 100 weeks:</li> <li>Group 1: Patients randomized from current ART Standard of Care (SOC) therapy</li> <li>Group 2: Patients currently receiving CAB LA + RPV LA Q4W</li> </ul> |
|---|---|
| Dosing | <ul> <li>Group 1: oral therapy with CAB 30 mg + RPV 25 mg once daily at Day 1 for 28 days (±3 days) to determine individual safety and tolerability, followed by CAB LA + RPV LA Q4W or CAB LA + RPV LA Q8W (as randomized at Day 1)</li> <li>Group 2: CAB LA + RPV LA Q4W or CAB LA + RPV LA Q8W (as randomized at Day 1)</li> </ul> |
| Time & Events | Refer to Appendix 2: Schedule of Activities |

| Overview of Study Design and Key Features | |
|---|---|
| Treatment<br>Assignment | Randomized (1:1) at Day 1 to receive CAB LA + RPV LA Q4W or CAB LA + RPV LA Q8W |
| | GSK RandAll NG used to generate randomization schedules |
| | <ul> <li>Stratified Randomization by prior CAB+RPV exposure (0 weeks, 1 to 24 weeks, &gt;24 weeks)</li> </ul> |
| Interim | Futility analysis at (approx.) 50% of subjects completing Week 24 |
| Analysis | Continuous time monitoring of confirmed virologic failure (CVF) in the Q8W randomized arm until all participants complete Week 24 visit |
| | The main analysis will be conducted to evaluate the primary objective of the protocol at Week 48. |
| | Preliminary analyses at Week 24 and analyses at Week 96 |
| | Further data cuts and analyses may be conducted as necessary in order to support regulatory submissions and publications. |

# 2.4. Statistical Hypotheses / Statistical Analyses

The study is designed to demonstrate that the antiviral effect of Q8W dosing with CAB LA + RPV LA is non-inferior to Q4W dosing CAB LA + RPV LA in subjects stably suppressed on an oral SOC regimen or Q4W CAB LA + RPV LA regimen prior to randomization. Non-inferiority in the proportion of participants with HIV-1 RNA  $\geq$ 50 c/mL at Week 48 (defined by the US FDA snapshot algorithm) can be concluded if the upper bound of a two-sided 95% confidence interval for the difference between the two treatment arms (Q8W – Q4W) is less than 4%.

If  $f_{Q8W}$  is the snapshot failure rate for Q8W CAB LA + RPV LA, and  $f_{Q4W}$  is the snapshot failure rate for Q4W CAB LA + RPV LA then the null (H<sub>0</sub>) and alternative (Ha) hypotheses can be written as follows:

$$H_0$$
:  $f_{O8W} - f_{O4W} \ge 4\% \text{ vs } H_a$ :  $f_{O8W} - f_{O4W} < 4\%$ 

#### 3. PLANNED ANALYSES

Analyses will be conducted to support Independent Data Monitoring Committee (IDMC) review of study data. At least three analyses will be conducted to evaluate the objectives of the protocol after all subjects have completed their visits at Week 24, Week 48 and Week 96, respectively. Prior to Week 48 analysis complete, the Week 24 results will be restricted to only those study team members and GSK/ViiV Healthcare senior management who need to be involved in the analysis and interpretation of the results for reporting to regulatory authorities. Details on protection against operation bias for Week 48 analysis are documented in the Study Results Dissemination Plan (SRDP) for this study. There is no planned hypothesis testing on the treatment difference at Week 24 and no decisions will be made based on the Week 24 results. Details of the planned displays for Week 24 analyses are provided in Section 15.14.4. Further data cuts and analyses may be conducted as necessary in order to support regulatory submissions and publications (first publication at Week 48). The Week 48 analysis will be primary and no results will be shared publicly until Week 48 analysis is complete. A final End-of-Study analysis will be conducted when all subjects have completed the study.

# 3.1. IDMC Analyses

An IDMC will be instituted to ensure external objective medical and/or statistical review of efficacy and safety to protect the ethical interests and well-being of subjects and to protect the scientific validity of this study.

The IDMC will evaluate accumulating efficacy, tolerability, safety and PK of CAB LA + RPV LA Q8W during the study. An interim futility analysis will be performed for the IDMC to evaluate the efficacy of CAB LA + RPV LA Q8W prior to the final analyses.

The interim futility analysis will be performed with the intent of having approximately 50% of participants reaching Week 24 and providing sufficient lead time to allow the IDMC to review the data prior to any participants reaching the Week 48 visit. A futility rule based on Bayesian posterior predictive probability approach will be applied to assess the probability that the CAB LA + RPV LA Q8W injectable regimen demonstrates non-inferiority to the CAB LA + RPV LA Q4W regimen at Week 24, given the partial data set. The sponsor will remain blinded to this analysis.

In addition, the IDMC may also monitor the incidence of participants meeting Confirmed Virologic Failure (CVF) criteria before all subjects have completed Week 24 to ensure that subjects are not being sub-optimally treated in the CAB LA + RPV LA Q8W arm.

Full details of the analyses, estimated timing, and the decision criteria that will be used to determine regimen performance will be pre-specified in the IDMC Charter.

A list of outputs required for each IDMC analysis will be provided in the IDMC Charter. Data handing methods and derived data definitions will be the same as detailed in this RAP, unless otherwise stated.

# 3.2. Final Analyses

The primary analysis will be conducted to evaluate the primary objective of the protocol at Week 48. These analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed Week 48 and had a re-test for HIV-1 RNA if necessary.
- 2. All required database cleaning activities have been completed and database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to Ramos NG procedures.

Two secondary analyses will be conducted at Week 24 and Week 96 and a final End-of-Study analysis will be conducted when all subjects have completed the study as defined in the protocol.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | <ul> <li>Comprised of all subjects screened for inclusion in the study.</li> <li>Subjects may be re-screened once, for which they will receive a new subject number.</li> </ul> | Study Population |
| | <ul> <li>receive a new subject number.</li> <li>For disposition displays, except for the listing of subjects who were rescreened, only the latest re-screening data will be included. All screening data will be summarized or listed for other displays.</li> </ul> | |
| Randomized | <ul> <li>All subjects who were randomly assigned to treatment in the study.</li> <li>In this study, the randomized population includes all enrolled participants, i.e. the randomized population is equivalent to the enrolled population.</li> <li>This population will be based on the treatment the participant was randomized to.</li> </ul> | Study Population |
| Safety | <ul> <li>All randomized subjects who received at least one dose of study treatment.</li> <li>Participants will be assessed according to actual treatment received.</li> </ul> | Safety |
| Intent-to-Treat<br>Exposed (ITT-E) | <ul> <li>All randomized subjects who received at least one dose of study treatment.</li> <li>Subjects will be assessed according to their randomized treatment, regardless of the treatment they received.</li> </ul> | <ul><li>Study Population</li><li>Efficacy</li><li>Health Outcomes</li></ul> |
| Per-Protocol<br>(PP) | <ul> <li>All subjects in the ITT-E population with the exception of major protocol violators.</li> <li>Protocol deviations that would exclude participants from the PP population are defined in Section 4.1 (Protocol Deviations) and Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population).</li> </ul> | Efficacy (Sensitivity Analysis) |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Pharmacokinetic (PK) | All subjects who received CAB and / or RPV and underwent PK sampling during the study and provide at least 1 non-missing CAB and / or RPV plasma concentration value (Non-quantifiable [NQ] values will be considered as non-missing values). | • PK |
| Confirmed<br>Virologic Failure<br>(CVF) | All subjects in the ITT-E population who met Confirmed Virologic Failure (CVF) criteria. | Virology Efficacy |
| Long-term Follow-<br>up (LTFU) | All subjects receiving at least one dose of CAB LA and/or RPV LA who have discontinued the CAB LA + RPV LA regimen and have either at least one Long-term Follow-up phase clinic visit (i.e. have at least one long-term follow-up visit shown in the study database, LTFU month 1, LTFU month 3, etc) or have filled out the LTFU phase conclusion form. | <ul><li>Safety</li><li>Study Population</li></ul> |
| Week 24 Futility | <ul> <li>All subjects in the ITT-E population who started study treatment at least 168 days prior to the IDMC cut-off date (in order to account for subjects who withdrew early but would have reached Week 24)</li> <li>The IDMC cut-off date is the predicted Week 24 visit date</li> </ul> | IDMC Futility Analysis (i.e. IDMC Week 24 Analyses) |
| | (Last Subject Last Visit) corresponding to the time at which approximately 50% of subjects have completed Week 24. | |
| Oral Lead-in | All subjects who received at least one dose of study treatment during the oral lead-in period in ATLAS-2M | <ul><li>Safety</li><li>Study Population</li></ul> |
| | study. | Efficacy |
| Q4W ATLAS | All subjects in the ITT-E population who were randomized to Q4W arm in ATLAS. | Health Outcomes |
| SOC | All subjects in the ITT-E population who either were randomized to SOC arm in ATLAS or did not participate in ATLAS. List of Data Displays which details the population used for each display. | Health Outcomes |

Refer to Section 15.14: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population).

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG Randomization System Data Displays for Reporting | | | Reporting |
| Code | Description | Description | Order in TLF |
| Α | Q8W | Q8W | 1 |
| В | Q4W | Q4W | 2 |
| C/A | Oral followed by Q8W | Q8W | 1 |
| C/B | Oral followed by Q4W | Q4W | 2 |

#### Notes:

Unless stated otherwise, data displays will present two treatment group columns (Q8W and Q4W), where
treatment sequence C/A is pooled with sequence A and treatment sequence C/B is pooled with sequence B. The
detailed treatment sequence descriptors (i.e. C/A and C/B) may be used in selected data listings. Treatment C
refers to oral CAB + oral RPV, used for oral lead-in for subjects entering the study with no prior CAB+RPV
exposure.

Treatment comparisons will be displayed as follows using the descriptors as specified:

1. Q8W vs Q4W

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-treatment (see Table 8) assessment with a non-missing value, including those from unscheduled visits. 'Pre-treatment' here refers to prior to the study treatment (i.e. CAB and/or RPV) in this study.

Electrocardiograms (ECGs) are to be performed in triplicate on Day 1 visit. The baseline value for an ECG parameter will be the mean of the last pre-treatment set of assessments from the same date, so long as at least one of the triplicate assessments is available.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

#### 5.3. Multicentre Studies

Data will be summarized for all centres combined. Country will be treated as an exploratory subgroup for analyses of the primary efficacy endpoint as described in Section 7.1.5.1 and secondary efficacy endpoint (HIV-1 RNA <50 c/mL) as described in Section 7.2.5.1. Some countries may be combined for exploratory subgroup analyses with consideration due to the number of participants enrolled.

# 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

The list of covariates and other strata may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates and other strata of clinical interest may also be considered.

| Category | Details |
|---|---|
| Strata | Randomization Strata: |
| | For the proportion of participants with plasma HIV-1 RNA ≥ 50 c/mL per FDA Snapshot algorithm at Week 48 (primary endpoint), a stratified analysis with Cochran-Mantel Haenszel weights will be used to adjust the primary treatment comparison for the randomization strata corresponding to prior exposure to CAB+RPV (0 weeks, 1-24 weeks, >24 weeks). A similar approach will be used to adjust the analysis of the proportion of participants with HIV-1 RNA <50 c/mL (per the FDA's Snapshot algorithm) at Week 48 (key secondary endpoint) and repeat analyses of these endpoints at Week 96. |
| | See Section 7.1.5.1 for additional details on the statistical analysis methodology. |
| Other<br>Subgroups /<br>Covariates | See details in Section 5.4.2 |

# 5.4.2. Examination of Subgroups

The following is a list of subgroups that may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be combined prior to un-blinding the trial.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.
- For subgroup analysis, per European Medicines Agency Guideline on the investigation of subgroups in confirmatory clinical trials (EMA, 2014), factors defining a subgroup population may be put in three categories:

EMA Subgroup Category 1: Factors with strong reason to expect a heterogeneous response to treatment. In this case separate trials should usually be planned. There are no factors falling into this category in this study.

EMA Subgroup Category 2: Factors with at least some biological plausibility or external evidence such that a heterogeneous response might be hypothesized. In this study, stratified randomization strata, key demographic factors, Baseline CD4, CDC stage will be fall into this category. For these factors, subgroup analyses will be performed but likely underpowered so that a formal proof of efficacy will not be available individually

in all subgroups. If consistent findings across multiple comparisons were observed then these analyses would still be suggestive of a generalizable finding from the overall population.

EMA Subgroup Guideline Category 3: Factor with good argumentation why homogeneity of response to treatment is plausible. The impact of factors falling into this category will be explored.

• Additional covariates of clinical interest may also be considered.

| Category | Covariates and / or Subgroups |
|---|---|
| EMA Subgroup Category 2: | |
| Randomization Strata | Prior exposure to CAB+RPV (0 weeks, 1-24 weeks, >24 weeks) For analysis purposes, randomization strata will be rederived using |
| | eCRF data, even if this differs from the strata captured in RAMOS NG. |
| | All statistical analyses will adjust for the above randomization strata, unless stated otherwise. Treatment-by-Strata interactions will be assessed as specified in the analysis sections. |
| Demographic and Baseline | • Age: |
| Characteristic Subgroups | <ul> <li>&lt; 35, 35 - &lt; 50, ≥ 50</li> <li>For the statistical modelling, '&lt; 35' and '35 - &lt; 50' will be consolidated i.e. the following age group will be used:</li> <li>&lt; 50, ≥ 50</li> </ul> |
| | For the summary of demographic characteristics, the following age groups will also be presented: |
| | <ul> <li>≤ 18, 19 - 64, ≥ 65 (FDAAA requirement)</li> <li>18 - 64, 65 - 84, ≥ 85 (EMA requirement)</li> </ul> |
| | Race: |
| | White, Non-White Non-White Non-White Non-White |
| | <ul> <li>Black/African American, Non-Black/African American</li> <li>For the statistical modelling, only White vs Non-White is</li> </ul> |
| | considered. |
| | Sex at birth: |
| | o Female |
| | o Male |
| | Country (not used for statistical modelling) |
| | o Argentina |
| | o Australia |
| | o Canada |
| | <ul><li>France</li><li>Germany</li></ul> |
| | o Italy |
| | Korea, Republic of |
| | o Mexico |
| | <ul> <li>Russian Federation</li> </ul> |

| Category | Covariates and / or Subgroups |
|---|---|
| | South Africa |
| | o Spain |
| | o Sweden |
| | <ul> <li>United States</li> </ul> |
| | Baseline CD4+ cell count (cells/mm³): |
| | ○ <350 |
| | o 350 - < 500 |
| | ○ ≥ 500 |
| | Baseline HIV-1 RNA (c/mL): |
| | <50 |
| | o ≥ 50 |
| | Derived Baseline Centers for Disease Control and Prevention (CDC) estagen; |
| | (CDC) category: |
| | <ul><li>Stage I</li><li>Stage II</li></ul> |
| | Stage III Prior Exposure to CAB+RPV: |
| | Prior Exposure to CAB+RPV. O weeks |
| | o veeks<br>o ≥1 weeks |
| | This subgroup will be used in efficacy analysis, in addition to |
| | the redrived randomization strata (prior exposure to |
| | CAB+RPV: 0, 1-24, and >24 weeks). It will also be used in |
| | health outcomes analysis. In other types of analysis, only the |
| | rederived randomization strata will be used. |
| | Baseline BMI (kg/m²) |
| | o <30 |
| | o ≥30 |
| | Baseline Third Agent Class: |
| | <ul> <li>None (for subjects with prior exposure to CAB+RPV in</li> </ul> |
| | ATLAS, i.e. subjects transitioned from ATLAS) |
| | o NNRTI |
| | o INI |
| | o PI |
| EMA Subgroup Category 3: | |
| Additional subgroup/covariates for | PK/PD efficacy analysis will be performed for participants without prior |
| PK/PD efficacy analysis | exposure to CAB + RPV. |
| | Wook 8 CAR/PD\/ Trough DK concentration /i.e. are does DK |
| | Week 8 CAB/RPV Trough PK concentration (i.e. pre-dose PK concentration at nominal visit of Week 8) |
| | concentration at nominal visit of vvectory |
| | The above covariate will be dichotomized into two subgroup factors |
| | as follows: |
| | o ≤ first Quartile vs > first quartile, |
| | o ≤ Median vs > Median |
| | The concentration will also be treated as earth-ways well-blade |
| | The concentration will also be treated as continuous variable in |
| | logistic regression modelling analysis (i.e. the concentration data will be log <sub>2</sub> transformed in this analysis so that, for assessing the effect, |
| | De 1092 transionned in this analysis 50 that, for assessing the effect, |

| Category | Covariates and / or Subgroups |
|---|---|
| | one unit increase of the point estimate of log2 PK concentration is equivalent to 'doubling the concentration' in the original value). |
| | Length of First CAB/RPV Injection Needle (<2, ≥2 inches) |
| Additional subgroup/covariates for PK/PD safety analysis | For the plot of Maximum Change from Baseline(CFB) in ALT/Total Bilirubin versus Last Trough CAB/RPV PK Concentrations, Last CAB/RPV Trough PK Concentration is the most recent trough PK concentration prior or equal to the date of the lab assessment with maximum CFB during the maintenance phase. For the Plot of Maximum Toxicity Grades of Most Frequently Reported Study Drug ISR adverse events (AEs) versus Last Trough CAB/RPV PK Concentrations, Last CAB/RPV Trough PK Concentration is the most recent trough PK concentration prior or equal to the earliest onset date of the most frequently reported Study Drug ISR AE with maximum toxicity grade, during the maintenance phase. If a participant has no Study Drug ISR AE most commonly reported, then the last trough value during the maintenance phase will be used for the plot. |
| Additional subgroup for common drug-related study drug injection site reaction (ISR) with maximum toxicity grade | <ul> <li>For each preferred term of the common drug-related study drug ISR with maximum toxicity grade (pain, induration, nodules and any other study drug ISR with &gt;=5% subjects in either treatment arm) during the maintenance phase:</li> <li>Needle Length for Last CAB Injection prior to and including the onset date of the earliest corresponding drug-related CAB ISR with maximum toxicity grade during the maintenance phase: ≤1.5, &gt;1.5 to &lt;2, ≥2 inches</li> <li>Needle Length for Last RPV Injection prior to and including the onset date of the earliest corresponding drug-related RPV ISR with maximum toxicity grade during the Maintenance Phase: ≤1.5, &gt;1.5 to &lt;2, ≥2 inches</li> <li>Note: If there is no ISR of interest reported during maintenance phase for a subject, the needle length of last injection during maintenance phase will be used in the summary.</li> </ul> |

# 5.5. Multiple Comparisons and Multiplicity

# 5.5.1. Primary Comparison of Interest

The primary analysis will be based on the ITT-E population. The primary comparison will be made at a one-sided 2.5% level of significance. Treatment with Q8W will be declared non-inferior to Q4W if the upper end of a two-sided 95% confidence interval for the difference between the two groups (Q8W – Q4W) in the proportion of participants with HIV-1 RNA  $\geq$ 50 c/mL at Week 48 (defined by the US FDA snapshot algorithm) lies below 4%.

The primary comparison of interest is the comparison between Q8W (CAB LA + RPV LA Q8W) and Q4W (CAB LA + RPV LA Q4W) for the primary endpoint in the ITT-E population. This analysis will be adjusted for by the re-derived randomization strata based on eCRF data.

#### 5.5.2. Other Comparisons of Interest

If the primary comparison of interest (Section 5.5.1) using the ITT-E population demonstrates non-inferiority of Q8W compared to Q4W then the following key secondary comparisons will be tested:

- Treatment with Q8W will be declared non-inferior to Q4W with respect to the proportion of participants with HIV-1 RNA < 50 c/mL at Week 48 (defined by the US FDA snapshot algorithm) if the lower end of a two-sided 95% confidence interval for the difference between in rates (Q8W Q4W) lies above -10% using the ITT-E population
- Superiority of Q8W compared to Q4Wwith respect to change from baseline HIVTSQs total score at Week 48 using the ITT-E population and a two-sided 5% level of significance. Refer to Section 12.5.1 for details.

For the primary endpoint treatment comparison at Week 48, no multiple comparison adjustment is necessary for testing non-inferiority followed by superiority (conditional on achieving a significant test for non-inferiority) since testing follows a pre-specified sequence of hypothesis such that if the first hypothesis tested is not significant, all subsequent tests will not be performed. This fixed sequence procedure controls the type I error rate at the nominal level. The primary endpoint treatment comparison at Week 48 will also be performed using the PP population and the results will be compared for consistency with the results from the ITT-E population.

In addition to the primary and the key secondary comparisons, the comparisons between two treatment arms for ACCEPT (general acceptance score), PIN (Domain scores (CCI)), and Individual Items Scores (CCI)), HAT-QoL (Life satisfaction, HIV medications, disclosure worries) and HIVTSQc (Treatment Satisfaction score) at timepoints through Week 48 will also be performed as supportive analyses.

Lastly, for the IDMC interim analyses, since the statistical stopping guidelines will not result in early stopping for positive efficacy findings, these interim treatment comparisons will not inflate the Type I error rate for the primary treatment comparison.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 15.3 | Appendix 3: Assessment Windows |
| 15.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |

| Section | Component |
|---------|-------------------------------------------------------------------|
| 15.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 15.6 | Appendix 6: Derived and Transformed Data |
| 15.7 | Appendix 7: Reporting Standards for Missing Data |
| 15.8 | Appendix 8: Values of Potential Clinical Importance |
| 15.9 | Appendix 9: Snapshot Algorithm Details |
| 15.10 | Appendix 10: Variables Defined for Time to Event Analysis |
| 15.11 | Appendix 11: Identification of Adverse Events of Special Interest |
| 15.12 | Appendix 12: IDMC |

#### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and oral study treatment accountability will be based on GSK Core Data Standards.

Table 1 provides an overview of the planned study population analyses, with details of the planned displays are presented in Appendix 14: List of Data Displays.

Table 1 Overview of Planned Study Population Analyses

| Display Type | Data Dis | plays Generated |
|------------------------------------|-----------------|-----------------|
| | Table | Listing |
| Randomization | | |
| Randomization [1] | | <b>Y</b> [2] |
| Subject Disposition | | |
| Study Populations [3] | Υ | |
| Study Recruitment [3] | Υ | |
| Reasons for Screening Failures [3] | Υ | Y |
| Rescreened Subjects [3] | | Y |
| Age Ranges | Υ | |
| Subject Disposition | <b>Y</b> [4][5] | |
| Reasons for Withdrawal | <b>Y</b> [4][5] | Y |
| IP Discontinuation | Y | Y |
| Important Protocol Deviations | Y | Y |

| Display Type | Data Displays Generated | |
|---|---|---|
| | Table | Listing |
| Deviations leading to exclusion from PP | Y | Υ |
| Inclusion and Exclusion Criteria Deviations | Y | Υ |
| Demography and Baseline | | |
| Demographics Characteristics [6] | Y | Υ |
| Race & Racial Combinations [7] | Y | Υ |
| Hepatitis Status at Entry | Y | |
| Baseline CDC Classification of HIV infection (2014) | Y | |
| Baseline Cardiovascular Risk Assessments | Y | |
| Distribution of CD4+ Cell Counts at Screening and Baseline | Y | |
| Prior Exposure to CAB+RPV | Y | |
| HIV-1 Risk Factors | Y | |
| Medical Conditions, Concomitant Medications & Antiretrov | iral Therapy | |
| Medical Conditions (Current/Past) [8] | Y | |
| Medical Conditions: Sub-conditions (Current/Past) [9, 10] | Υ | |
| Concomitant Medications (non-ART) | Y[10] | |
| Prior ART Medications | Y | Υ |
| Concomitant ART Medications during Maintenance Phase | | Υ |
| ART Medications Received during LTFU Phase | | Υ |
| Lipid Modifying Agents (Baseline and during Maintenance Phase) | Y | |
| Substance use at Entry | Y | |
| Medical History of Seizure | | Υ |
| Other | <u>.</u> | |
| Oral Study Treatment Accountability [11] | | Υ |

#### NOTES:

- T = Tables, L = Listings, Y = Display Generated,
- 1. Base on Randomized population.
- 2. One listing of participants randomized but not treated, and one listing of randomized and actual strata and treatment assignment.
- 3. All Subjects screened population.
- 4. Participants who have not been recorded as either completing or withdrawing from the study will be categorized as "Ongoing at time of the analysis" for summary purposes.
- 5. Analysis of subject disposition will be performed for each Study Phase separately, as well as for overall study conclusion.
- 6. Age and ethnicity collected at Screening; weight and height collected at Baseline.
- 7. The five high level FDA race categories and designated Asian subcategories will be summarised along with all combinations of high level categories which exist in the data. The nine race categories collected will be summarised along with categories for mixed race. A by-subject listing of race will also be produced.
- 8. Medical conditions will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).
- 9. Sub conditions are Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, and Nervous System Conditions.
- 10. summarised by, Ingredient combinations.
- 11. Dispensation information (dates and number of tablets dispensed and returned).

#### 6.2. Prior and Concomitant Medications

Non-ART and/or ART Medications will be classified by categories shown in Table 2. The same medication may be classified by more than one categories. For example, if the Non-ART medication was started after the maintenance treatment start date and was stopped at nominal Week 104 visit while subject was still receiving study treatment, this medication would be considered both 'concomitant during maintenance' and 'concomitant during extension'.

Table 2 Derived Data for Non-ART Medications/ART Medications

| | Definition |
|---|---|
| Prior | ART Medication Taken ≤ Maintenance Treatment Start Date |
| | Non-ART Medication Taken < Maintenance Treatment Start Date |
| Concomitant | For subjects continuing into Extension Phase: |
| during<br>Maintenance | Maintenance Treatment Start Date ≤ Non-ART Medication Taken < Date of Nominal Week 100 Visit |
| | Maintenance Treatment Start Date < ART Medication Taken ≤ Date of Nominal Week 100 Visit |
| | For subjects not continuing into Extension Phase <sup>[a]</sup> : |
| | Maintenance Treatment Start Date ≤ Non-ART Medication Taken < LTFU ART Start Date |
| | Maintenance Treatment Start Date < ART Medication Taken < LTFU ART Start Date |
| Concomitant | For subjects continuing into Extension Phase <sup>[a]</sup> : |
| during Extension | Date of Nominal Week 100 Visit ≤ Non-ART Medication Taken < LTFU ART Start Date |
| | Date of Nominal Week 100 Visit < ART Medication Taken < LTFU ART Start Date |
| Received during<br>Long-term Follow- | For subjects Who received at least one CAB and/or RPV injection and have started LTFU ART: |
| up | Non-ART/ART Medication Taken ≥ LTFU ART Start Date |

#### NOTES:

- Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for medications. Use the rules in this table if medication date is completely missing.
- [a] If subjects have missing LFTU ART start date, only the lower bound will be considered in the derivation.

#### 7. EFFICACY ANALYSES

# 7.1. Primary Efficacy Analyses

#### 7.1.1. Endpoint / Variables

Proportion of participants with plasma HIV-1 RNA ≥50 c/mL as per Food and Drug Administration (FDA) Snapshot algorithm at Week 48 (Intent-to-Treat Exposed [ITT-E] population); see Section 15.9 for additional details.

#### 7.1.2. Summary Measure

Difference in the proportion of participants with HIV-1 RNA ≥50 c/mL at Week 48 (defined by the US FDA snapshot algorithm) between each treatment group (Q8W – O4W).

### 7.1.3. Population of Interest

The primary efficacy analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

#### 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

As defined by the Snapshot algorithm, HIV-1 RNA  $\geq$  50 c/mL is determined by the last available HIV-1 RNA measurement while the participant is on treatment within the analysis visit window of interest.

Participants without on-treatment HIV-1 RNA data for the visit of interest and who discontinue treatment for reasons not related to adverse event while having HIV-1 RNA  $\geq 50$  c/mL at time of discontinuation or who change study treatment not permitted per protocol before the analysis window are classified as having HIV-1 RNA  $\geq 50$  c/mL.

#### 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 14: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

### 7.1.5.1. Statistical Methodology Specification

#### **Endpoint**

Proportion of Participants with plasma HIV-1 RNA ≥ 50 c/mL at Week 48 using the Snapshot algorithm for the ITT-E population. Subjects with 'HIV-1 RNA ≥ 50 c/mL' per Snapshot algorithm include those who had plasma HIV-1 RNA ≥ 50 c/mL at Week 48, who discontinued for lack of efficacy, who discontinued for other reasons while not <50 c/mL, or who changed ART.</li>

#### **Snapshot Dataset**

- Virologic outcome ('HIV-1 RNA <50 c/mL' or 'HIV-1 RNA ≥ 50 c/mL') per Snapshot algorithm is determined by the last available on-treatment HIV-1 RNA measurement within the analysis visit window of interest (please refer to analysis window defined in Table 10). In addition, subjects who discontinue for reasons not related to adverse event with on-treatment HIV-1 RNA result at the time of discontinuation ≥ 50 c/mL or who change study treatment not permitted per protocol during maintenance phase before the analysis visit are classified as 'HIV-1 RNA ≥ 50 c/mL'.</li>
- Full details of the Snapshot algorithm are provided in Section 15.9.

### **Model Specification**

- The primary efficacy endpoint will be analysed using a stratified analysis with Cochran-Mantel-Haenszel (CMH) weights, adjusting for the rederived randomization strata corresponding to prior exposure to CAB+RPV (0 weeks, 1-24 weeks, >24 weeks)
- The CMH estimate of the adjusted treatment difference will be calculated as a weighted average of strata-specific estimates of the treatment difference calculated within each stratum as follows:
  - o If  $n_k$  is the number of Q8W treated participants,  $m_k$  is the number of Q4W arm treated participants, and  $N_k = n_k + m_k$  is the total number of participants in the kth stratum, then the CMH estimate is given by

$$\hat{d}_{cmh} = \frac{\sum W_k \hat{d}_k}{\sum W_k}$$

where

$$W_k = \frac{n_k m_k}{N_k}$$

are CMH weights and  $\hat{d}_k$  are estimates of the differences in proportions between the two treatment arms, f<sub>Q8W</sub>-f<sub>Q4W</sub>, for the *kth* stratum.

• The corresponding two-sided 95% CI will be calculated as

$$\hat{d}_{omh} \pm 1.96 \times \sqrt{v a r(\hat{d}_{omh})}$$

where the variance estimator [Sato, 1989] is consistent in both sparse data and large strata and is given below:

$$\operatorname{var}(\hat{d}_{cmh}) = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{\left(\sum n_k m_k / N_k\right)^2} = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{\left(\sum W_k\right)^2}$$

where

$$P_k = \frac{n_k^2 y_k - m_k^2 x_k + n_k m_k (m_k - n_k)/2}{N_k^2}$$

$$Q_{k} = \frac{x_{k}(m_{k} - y_{k})/N_{k} + y_{k}(n_{k} - x_{k})/N_{k}}{2}$$

with  $x_k$  and  $y_k$  corresponding to the number of participants with Plasma HIV-1 RNA  $\geq$  50 c/mL at Week 48 per FDA Snapshot for Q8W and Q4W, respectively, for the *kth* stratum.

#### **Model Results Presentation**

- Adjusted CMH estimate of the difference in the proportion of subjects with Plasma HIV-1 ≥ 50 c/mL between each treatment group (Q8W Q4W) and corresponding 95% confidence interval.
- Non-inferiority will be concluded if the upper bound of the two-sided 95% confidence interval for the CMH adjusted treatment difference (Q8W Q4W) is less than 4%.
- If this analysis shows non-inferiority, then a superiority hypothesis will be tested at the two-sided 5% level of significance. Superiority favoring Q8W will be declared if the upper bound of the confidence interval is below 0% for the ITT-E population analysis. If superiority is declared, the p-value for superiority will also be calculated.

#### **Subgroup Analyses**

- 1. Treatment Heterogeneity across rederived randomization strata [prior exposure to CAB+RPV (0 weeks, 1-24 weeks, >24 weeks)]:
  - The weighted least squares chi-squared statistic [Fleiss, 1981] will be used to test for oneway homogeneity across the levels of each categorical variable, with each categorical variable considered separately.
  - Following Lui and Kelly [Lui, 2000] ½ will be added to each cell in any strata for which the stratum-specific rate estimates of either f<sub>Q8W</sub> or f<sub>Q4W</sub> are zero or one, and tests will be onesided.
  - Any heterogeneity found to be statistically significant will be explored and if necessary
    results will be reported for each level of the categorical variable. Investigation of
    heterogeneity will be confined to the primary endpoint. Tests of homogeneity will be
    assessed at the one-sided 10% level of significance.
- 2. Stratum-specific analyses for two groups of participants: (Group 1) those currently receiving Standard of Care antiretroviral therapy at Baseline (i.e. no prior exposure to CAB+RPV), (Group 2) those receiving Q4W CAB LA + RPV LA therapy in the ongoing ATLAS study (i.e. have prior exposure to CAB+RPV). For each stratum (Group 1 and Group 2), the following will be presented:
  - Proportion of subjects with plasma HIV-1 RNA ≥ 50 c/mL at Week 48 by treatment group.
  - Unadjusted difference in proportions between treatment groups and corresponding twosided 95% CI.
  - Summary of study outcomes (i.e. HIV-1 RNA < 50 c/mL, HIV-1 RNA ≥50 c/mL and reason for no data in the window)

For Group 2, a stratum-adjusted analysis will also be provided, with adjustment for prior CAB+RPV

exposure (1 to 24 weeks vs. >24 weeks) using Cochran-Mantel Haenszel (CMH) weights, as described in the model specification above for the overall primary analysis.

# 3. Exploration of Subgroups

- An analysis for subgroups listed in Section 5.4.2 will be performed. This will show the
  proportion of subjects with plasma HIV-1 RNA ≥50 c/mL at the time of analysis (Week 48)
  based on the Snapshot algorithm and will be presented by treatment group.
- Unadjusted difference in proportions between treatment groups and corresponding twosided 95% CI will also be presented by subgroups. The confidence interval will be calculated using an unconditional exact method [Chan et al, 1999] with two inverted onesided tests based on the score statistic. These results will also be presented graphically.
- Summary of study outcomes (i.e. HIV-1 RNA < 50 c/mL, HIV-1 RNA ≥50 c/mL or reason for no data in the window) by subgroup will be produced.

Note: These subgroup analyses will be exploratory and likely underpowered so that interpretation may therefore focus on point estimates as well as the upper bounds of 95% CIs for the treatment differences and response rates. Additionally, multiple comparisons are being made which inflates the risk of false positive findings. Therefore, if consistent findings across the multiple comparisons were observed then these analyses would still be suggestive of a generalizable finding of non-inferiority.

### **Sensitivity and Supportive Analyses**

- 1. Per-protocol population analysis:
  - To assess the impact of important protocol deviations, statistical analysis will be repeated using the Per-protocol population and compared for consistency with the results from the primary ITT-E population analysis.

# 7.2. Secondary Efficacy Analyses

# 7.2.1. Endpoints

The key secondary efficacy endpoint is the proportion of participants with plasma HIV-1 RNA < 50 c/mL at Week 48 using the FDA Snapshot algorithm (Intent-to-Treat Exposed [ITT-E] population).

Other secondary efficacy endpoints for the study are listed below:

- Proportion of participants with plasma HIV-1 RNA < 50 c/mL at Week 24 and Week 96 using the FDA Snapshot algorithm (ITT-E population)
- Proportion of participants with protocol-defined confirmed virologic failure (CVF) through Week 24, Week 48 and Week 96
- Proportion of participants with HIV-1 RNA ≥50 c/mL as per FDA Snapshot algorithm at Week 24 and Week 96
- Absolute values and changes from Baseline in viral load and CD4+ cell counts over time including Week 48 and Week 96

#### 7.2.2. Summary Measure

Difference in the proportion of participants with HIV-1 RNA < 50 c/mL at Week 48 and Week 96 (defined by the US FDA snapshot algorithm) between each treatment group (Q8W – Q4W).

Difference in the proportion of participants with HIV-1 RNA  $\geq$  50 c/mL at Week 24 and Week 96 (defined by the US FDA snapshot algorithm) between each treatment group (Q8W – Q4W).

#### 7.2.3. Population of Interest

The secondary efficacy analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

# 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

As defined by the snapshot algorithm, participants with last available HIV-1 RNA measurement less than 50 c/mL while the participant is on treatment within the analysis visit window of interest are classified as HIV-1 RNA < 50 c/mL.

Participants without on-treatment HIV-1 RNA data for the visit of interest and who discontinue treatment for reasons not related to adverse event while having HIV-1 RNA  $\geq 50$  c/mL at time of discontinuation or who change study treatment not permitted per protocol before the analysis window are classified as having HIV-1 RNA  $\geq 50$  c/mL.

# 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 14: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.2.5.1. Statistical Methodology Specification

#### **Key Secondary Statistical Analysis**

#### **Endpoint**

 Proportion of participants with plasma HIV-1 RNA <50 c/mL at Week 48 using the FDA Snapshot algorithm (Intent-to-Treat Exposed [ITT-E] population)

#### **Snapshot Dataset**

As Section 7.1.5.1 and Section 15.9

#### **Model Specification**

As specified in Section 7.1.5.1 but with 'HIV-1 RNA <50 c/mL' replacing HIV-1 ≥ 50 c/mL</li>

#### **Model Results Presentation**

Adjusted CMH estimate of the difference in the proportion of participants with HIV-1 RNA < 50</li>

#### **Key Secondary Statistical Analysis**

c/mL at Week 48 between each treatment group (Q8W – Q4W) and corresponding 95% confidence interval.

 Non-inferiority will be concluded if the lower bound of the two-sided 95% confidence interval for the CMH adjusted treatment difference (Q8W – Q4W) is greater than -10%.

### **Subgroup Analyses**

As specified in Section 7.1.5.1 but with HIV-1 RNA < 50 c/mL replacing 'HIV-1 RNA ≥ 50 c/mL.</li>

#### **Sensitivity and Supportive Analyses**

- 1. Per-protocol population analysis:
  - To assess the impact of important protocol deviations, statistical analysis will be repeated using the Per-protocol population and compared for consistency with the results from the primary ITT-E population analysis.

# 7.3. Exploratory Efficacy Analyses

Table 3 provides an overview of the planned exploratory efficacy analyses. Details of the planned displays are provided in Appendix 14: List of Data Displays and will be based on GSK data standards and statistical principles. The exploratory efficacy analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

Table 3 Overview of Exploratory Efficacy Analyses

| Endpoints | | | | | Absolute | | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sum | mary | Indiv | idual | Stats Analysis | | Summary | | Individua | | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Proportion of participants without efficacy-related discontinuation (ERDF) or treatment-related discontinuation (TRDF) failure at Week 24/Week 48/Week 96 | | | | | | | | | | | | | | |
| Kaplan-Meier estimate | | | | Υ | | | | | | | | | | |
| Proportion of participal<br>Snapshot | nts wi | th pla | sma | HIV-1 | RNA≥ | ≥50 c/r | nL ov | er tim | e (Ma | intena | ance F | Phase) | - | |
| by visit | | | | Υ | <b>Y</b> [1] | | | | | | | | | |
| By visit and subgroup | | | | Υ | <b>Y</b> [2] | | | | | | | | | |
| Proportion of participal Snapshot | Proportion of participants with plasma HIV-1 RNA <50 c/mL over time (Maintenance Phase) - | | | | | | | | | | | | | |
| by visit | | | | Υ | <b>Y</b> [3] | | | | | | | | | |
| By visit and subgroup | | | | Υ | <b>Y</b> [2] | | | | | | | | | |
| Proportion of participal Snapshot | Proportion of participants with plasma HIV-1 RNA ≥200 c/mL over time (Maintenance Phase) - | | | | | | | | | | | | | |
| by visit | | | | <b>Y</b> [4] | <b>Y</b> [5] | | | | | | | | | |
| Proportion of participal Snapshot | nts wi | th pla | sma | HIV-1 | RNA < | 200 c | /mL o | ver tir | ne (M | ainter | ance | Phase | <del>)</del> - | |
| by visit | | | | <b>Y</b> [4] | <b>Y</b> [5] | | | | | | | | | |
| Proportion of participal injection - Snapshot | nts wi | th pla | sma | HIV-1 | RNA≥ | ≥50 c/r | nL at | Week | 48/W | eek 90 | 6 by d | elay ir | ı IP | |
| by delay in IP injection | | | | Υ | | | | | | | | | | |
| Proportion of participa | nts wi | th pla | sma l | HIV-1 | RNA < | 2 c/m | L ove | r time | (Mair | tenar | nce Ph | nase) | | |
| by visit | | | | Υ | | | | | | | | | | |
| Plasma HIV-1 RNA ove | r time | | | | | | | | | | | | | |
| by visit | | | | Υ[7] | | <b>Y</b> [8] | <b>Y</b> [9] | | | | | | | <b>Y</b> [9] |
| Target Detected vs<br>Target Not Detected by<br>visit [10] | | | | Υ | | | <b>Y</b> [11] | | | | | | | |
| Confirmed Virologic Fa | ilure | (CVF) | | | | | | | | | | | | |
| CVF overall | | | | Υ | | | | | | | | | | |
| CVF by visit | | | | Υ | | | Υ | | | | | | | |

| Endpoints | Absolute | | | | | Change from Baseline | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats Analysis | | lysis | Summary | | Individual | | Stats Analysis | | Summary | | Individual | | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Plasma HIV-1 RNA at<br>time of suspected and<br>confirmed virologic<br>failure | | | | Υ | | | | | | | | | | |
| CD4+ & CD8+ Cell Cou | Counts Over Time | | | | | | | | | | | | | |
| CD4+ observed [12] | | | | Υ | | | | | | | Υ | | | |
| CD8+ observed [12] | | | | Υ | | | | | | | Υ | | | |
| CD4+/CD8+ ratio observed [12] | | | | Υ | | | | | | | | | | |
| HIV-1 Conditions and D | iseas | e Pro | gress | ion | | | | | | | | | | |
| HIV Conditions including/excluding Recurrences as recorded in eCRF | | | | Υ | | | Υ | | | | | | | |
| HIV Disease<br>Progressions [13] | | | | Υ | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of data.
- Individual = Represents FL related to any displays of individual participant's data.
- 1. Line plots, with 95% confidence intervals (CIs), for the proportion of participants with HIV-1 RNA ≥50 c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 0%; otherwise, they are derived using the normal approximation.
- 2. Plot of the unadjusted treatment difference and its 95% confidence intervals (Snapshot algorithm) overall and by subgroup at Week 48/Week 96.
- 3. Line plots, with 95% confidence intervals, for the proportion of participants with HIV-1 RNA<50 c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 100%; otherwise, they are derived using the normal approximation.
- 4. Study outcomes (i.e., HIV-1 RNA <200 c/mL, HIV-1 RNA ≥200 c/mL, or reason for no data in the window) based on the snapshot algorithm at Week 48 will also be produced.
- 5. Line plots, with 95% confidence intervals, for the proportion of participants with HIV-1 RNA <200 c/mL and ≥200 c/mL by treatment group at each visit. The 95% CIs will be calculated using Exact (Clopper-Pearson) confidence interval if the proportion is 0% or 100%; otherwise, they are derived using the normal approximation.</p>
- 6. Delay in IP injection (days) is defined in Section 15.6.3.
- 7. Using log10 transformed values.
- 8. Individual plasma HIV-1 RNA only for participants who are in the category of 'viral load ≥50 c/mL' at Week 48 per Snapshot algorithm or who are CVF participants. The figures will display all HIV-1 RNA values collected.
- 9. For CVF participants, participants with viral load ≥ 50 c/mL during the Maintenance Phase, and participants with viral load ≥ 50 c/mL during the Maintenance oral lead-in period.
- 10. See Section 15.6.3 for definition of "Target Detected" and "Target Not Detected", and for the specification of corresponding summary table.
- 11. Target Detected" and "Target Not Detected" are included in the listing for plasma HIV-1 RNA by visit.
- 12. Using available data without imputation for missing values.
- 13. See Section 15.6.3 for HIV disease progressions.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

### 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Section 15.14: List of Data Displays.

# 8.1.1. Analyses for Injection Site Reaction Adverse Events from Study Drug Injection

Injection Site Reaction (ISR) adverse events of interest are those from study drug injections. For the summary of study drug ISR adverse events by visit and maximum severity (overall and by common ISRs): ISRs will be assigned based on onset date to the most recent planned IM injection visit prior or equal to the AE onset date.

Maximum grade at each visit will be derived as the maximum grade among ISRs assigned to the particular visit, with consideration for whether the summary applies to a particular preferred term (vs. across preferred terms), drug-related associated to CAB and/or RPV, or stratification by subgroup (such as needle length, refer to Section 5.4.2).

Drug-related ISRs (based on investigator discretion) from study drug injections will be attributed to the causal agent (CAB vs. RPV) when this can be determined specifically based on the side of injection administration and the side of the reported ISR (as collected in the eCRF). If we are unable to determine the causal agent in those cases where both drugs are given on one side and the ISR is reported non-specifically, then the attribution to a specific causal agent will remain unknown.

Common study drug ISR adverse events are defined by MedDRA preferred terms including injection site pain, injection site induration, injection site nodules and preferred terms of any other ISR with  $\geq$ 5% participants in either treatment arm, coming from study drug injections. The same set of common terms will be applied to 'overall' (CAB and/or RPV), CAB alone, RPV alone.

Study drug ISRs will be attributed to the needle length ( $\leq 1.5$ , > 1.5 to < 2,  $\geq 2$  inches) specifically based on the side of injection administration and the side of the reported ISR (as collected in the eCRF). If we are unable to determine the needle length for events where both drugs are given on one side and their needle lengths are different, then the attribution to a needle length will remain unknown.

# 8.2. Adverse Events of Special Interest Analyses

Adverse events of special interest (AESI) are determined for CAB and/or RPV based on pre-clinical and clinical experience, along with information for the Integrase Inhibitor class of HIV medications and RPV safety profile. Table 4 shows the currently identified AESI, drug(s) of Interest and the reasons for inclusion. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting, and/or

emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of AESIs may change at the time of reporting.

A summary by system organ class and preferred term will be provided for each of AESI. The characteristics of event occurrences during the maintenance phase will be summarized for common AESI which have at least 20 participants in either treatment arm. For Depression, anxiety and suicidal ideation/behaviour AESI, a summary by system organ class, maximum DAVIDS toxicity grade and prior history of suicidal ideation will be provided. The details of the planned grouping and planned displays are provided in Section 15.11 and Appendix 14: List of Data Displays.

Table 4 Adverse Events of Special Interest

| Adverse Events of Special Interest | Drug(s) of Interest | Reason for Inclusion |
|---|---|---|
| Hepatic Safety Profile: Assessment of Risk of hepatoxicity | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in HIV<br>population |
| Hypersensitivity Reactions (HSR) | CAB | Class, Regulatory Interest,<br>Occurs in HIV population |
| Rash | RPV | Class, Regulatory Interest,<br>Occurs in HIV population |
| Prolongation of the Corrected QT Interval of the ECG in Supratherapeutic Doses | RPV | Non-clinical, Clinical,<br>Regulatory Interest |
| Suicidal Ideation/Behaviour | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in HIV<br>population |
| Depression | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in HIV<br>population |
| Bipolar Disorder | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in HIV<br>population |
| Psychosis | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in HIV<br>population |
| Mood Disorders | CAB+RPV | Clinical, Class, Regulatory<br>Interest |
| Anxiety | CAB+RPV | Clinical, Class, Regulatory<br>Interest |
| Sleep Disorders | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in HIV<br>population |
| Injection Site Reactions (ISR) from Study Drug Injections [1] | CAB+RPV | Clinical |

| Drug(s) of Interest | Reason for Inclusion |
|---|---|
| CAB | Clinical, Regulatory Interest |
| CAB | Clinical, Class |
| CAB | Clinical, Class |
| CAB | Clinical, Therapeutic Area,<br>More prevalent in HIV<br>population |
| CAB+RPV | Regulatory Interest,<br>Therapeutic Area, More<br>prevalent in HIV population |
| CAB | Regulatory Interest, Class |
| | CAB CAB CAB CAB CAB CAB |

[1] A separate analysis will be performed for ISRs from study drug injections as described in Section 8.1.1.

#### 8.3. **Clinical Laboratory Analyses**

Laboratory evaluations including the analysis of results of Chemistry laboratory tests, Haematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 14: List of Data Displays.

#### 8.4. **Other Safety Analyses**

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 14: List of Data Displays.

ECG values of potential clinical importance are defined as a QTc of > 500 msec or increase from baseline in QTc  $\geq$  60 msec.
## 9. PHARMACOKINETIC ANALYSES

The GSK Division of Clinical Pharmacology Modelling and Simulation (CPMS) will be responsible for the PK analysis of CAB. The Division of Clinical Pharmacology and Pharmacometrics at Janssen Research and Development will be responsible for conduct or oversight of the PK analysis for RPV.

## 9.1. Endpoint / Variables

## 9.1.1. Drug Concentration Measures

Refer to Appendix 5 Data Display Standards & Handling Conventions (Section 15.5.3 Reporting Standards for Pharmacokinetic)

## 9.2. Overview of Planned Analyses

Table 5 provides an overview of the planned analyses with full details being presented in Appendix 14: List of Data Displays. All PK displays will be based on the PK Population, unless otherwise specified.

Table 5 Overview of Planned Pharmacokinetic Analyses

| | Stat | s Analy | /sis | Sun | nmary | Indiv | /idual |
|---|---|---|---|---|---|---|---|
| | Т | F | L | Т | F | F | L |
| Pharmacokinetic [5] | | | | | | | |
| Plasma CAB concentration by visit | | | | <b>Y</b> [1][2] | <b>Y</b> [1][3][4] | <b>Y</b> [3] | Υ |
| Plasma RPV concentration by visit | | | | <b>Y</b> [1][2] | <b>Y</b> [1][3][4] | <b>Y</b> [3] | Y |
| Steady state concentration | Y | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- Unless otherwise specified, all displays for evaluable concentrations except for individual displays will be
  presented by both overall and the rederived randomization strata.
- 1. For both 'all' concentration and the 'evaluable' concentration. The evaluable concentration is derived from samples collected within pre-specified Time window (Section 15.6.5)
- 2. For both 'untransformed' and 'log-transformed' statistics.
- The plots will be produced for the untransformed scale (i.e., a linear plot) and the log transformed scale (i.e., log-linear plot), separately.
- 4. Separate plots will be produced for Mean (SD) and Median concentration.
- 5. Standard summary statistics for concentration data will be calculated (i.e., mean, standard deviation, coefficient of variation, median, minimum and maximum). For Logarithmically transformed data, the summary statistics (i.e. geometric mean, between subject coefficient of variation, 95% confidence interval for the geometric mean and standard deviation) will also be calculated.

## 9.3. Statistical Analyses / Methods

## Planned PK statistical analysis

## **Steady State Concentration**

## **Endpoints**

 log<sub>e</sub>-transformation of the Trough/Pre-dose evaluable plasma concentrations (CAB/RPV) on Week 16-48 (i.e. Weeks 16, 24, 32, 40 and 48) for participants receiving Q8W study treatment

#### Covariates

Study Week

#### **Data Handling**

All data remains as is (observed).

## **Model Specification**

A mixed effects ANOVA model will be fitted for each rederived randomization stratum [prior exposure to CAB+RPV (0 weeks, 1-24 weeks, >24 weeks)] with Study Week (continuous variable) as a fixed effect and subject as a random effect for each analysis separately. The Kenward & Roger (KR) degrees of freedom approach will be used. The coefficient for the slope of the week effect on the loge-scale will be used to evaluate steady state for each drug (CAB/RPV). The 90% confidence intervals for the slope for each treatment will be calculated. If it does not appear that steady-state has been demonstrated, early weeks (e.g. Week 16, 24, etc...) results will be dropped and the analysis repeated.

## **Model Checking & Diagnostics**

• The steady state will be claimed (the coefficient for the slope of the week effect on the (natural) log scale was close to 0 or the 90% CI for the slope estimate included zero. If steady-state is not demonstrated, concentrations from early weeks (e.g. Week 16, 20, 24, etc...) dropped in sequence and the analysis repeated until either steady state is shown or only two timepoints remain.

#### **Model Results Presentation**

The coefficient for the slope of the week effect on the loge-scale, its standard error and 90% interval will be presented for each rederived randomization stratum.

## 10. POPULATION PHARMACOKINETIC ANALYSES

The Population PK analyses will be described under a separate Population-PK Reporting and Analysis Plans for CAB LA and RPV LA

# 11. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

The primary goal of this analysis is to characterize the pharmacokinetic / pharmacodynamic relationship of CAB/RPV administered in participants with HIV-1-infection who are virologically suppressed. The influence of subject demographics and

baseline characteristics and additional subgroups/covariates in this population will be investigated.

## 11.1. Overview of Planned Analyses

Table 6 provides an overview of the planned analyses with full details being presented in Appendix 14: List of Data Displays. All PK displays will be based on the PK Population, unless otherwise specified.

Table 6 Overview of Planned Pharmacokinetic / Pharmacodynamic Analyses

| | Stat | s Analy | /sis | Sun | nmary | Indiv | /idual |
|---|---|---|---|---|---|---|---|
| | T | F | L | T | F | F | L |
| CAB/RPV Week 8 concentrations by snapshot 'HIV-1 RNA ≥50 c/mL' (Yes vs. No) for participants without prior exposure to CAB+RPV | | | | Y | Y | | |
| Analysis of snapshot 'HIV-1 RNA ≥50 c/mL' at Week 48 by Week 8 trough concentration, and subgroup [¹¹] – univariable analysis /multivariable analysis for participants without prior exposure to CAB+RPV | Y | | | | | | |
| Individual CAB/RPV concentration-time profiles for participants with snapshot 'HIV-1 RNA ≥50 c/mL' at Week 48 or 96 | | | | | Y | | |
| Maximum change from baseline in ALT/Total Bilirubin versus last trough CAB/RPV concentrations [2] | | | | | Y | | |
| Maximum toxicity grades of most frequently reported study drug ISR AEs <sup>[3]</sup> versus last trough CAB/RPV PK concentrations <sup>[2]</sup> | | | | | Y | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- 1. Refer to Section 11.2.
- 2. Display by rederived randomization strata, i.e. prior exposure to CAB+RPV (0, 1-24, >24 weeks) derived based on eCRF.
- 3. Most frequently reported study drug ISR AEs are those top 5 in incidence in either treatment arm (i.e. Q8W or Q4W arm).

# 11.2. Statistical Analyses / Methods

# PK/PD Efficacy Analysis for Participants without Prior Exposure to CAB+RPV Endpoints

Snapshot 'HIV-1 RNA≥50 c/mL' at Week 48 (or W96)

#### **Covariates**

 Treatment, demographic and baseline characteristics except for country and Prior Exposure to CAB+RPV (0, ≥1 weeks), and additional subgroup/covariates for PK/PD efficacy analysis see derivation details in Section 5.4.2.

#### **Data Handling**

All data remains as is (observed).

## **Model Specification**

• Logistic regression will be used to exam the correlation between the endpoint (Snapshot 'HIV-1 RNA≥50 c/mL') at Week 48 and the covariates/subgroups. This logistic regression analysis will be performed for each covariate or subgroup, separately (univariable analysis), and will also be performed with one multivariable analysis using Backward stepwise selection approach to identify the covariates/subgroups potentially affecting virologic response.

## **Model Checking & Diagnostics**

- For the multivariable analysis, a logistic regression model that best predicts the dependent variable (i.e. snapshot 'HIV-1 RNA≥50 c/mL') from the independent variables (i.e. covariates/factors with P <0.15 from univariable analysis) will be determined using the backward stepwise selecting approach. Week 8 trough PK concentration will be logarithmically transformed with base of 2 (i.e. one-unit increase of the point estimate of log2 PK concentration is equivalent to 'doubling the concentration' in the original value). The analysis will start with all covariates in the model and remove a covariate with the largest p-value (i.e. the least statistically significant) each time and continue until the stopping rule is reached when all remaining covariates have p-value <15%.
- If problems with model convergence occur due to zero event counts or complete/quasicomplete separation, then alternative methods such as exact logistic regression may be used.

#### **Model Results Presentation**

• The odds ratio, 95% confidence interval, and p-value will be presented.

## 12. HEALTH OUTCOMES ANALYSES

# 12.1. Endpoint / Variables

- Preference between injections of LA HIV treatment and daily oral HIV treatment at Week 48
- Preference between LA injection every 8 weeks and LA injection every 4 weeks at Week 48 (Q8W arm only)
- Change from baseline in total "treatment satisfaction" score, and individual item scores of the HIV Treatment Satisfaction Status Questionnaire (HIVTSQs) at Weeks 24 and 48
- Change from baseline in life satisfaction, HIV medication, and disclosure worries using HIV/AIDS Targeted Quality of Life (HAT-QoL) at Weeks 24 and 48

- Change in treatment satisfaction over time using the HIV Treatment Satisfaction Change (HIVTSQc) questionnaire at Week 48
- Change from Week 8 in Dimension Scores and individual item scores assessing pain during injection, anxiety before and after injection, willingness to be injected in the future and overall satisfaction with mode of administration over time using Perception of Injection (PIN) questionnaire at Weeks 24 and 48
- Change from baseline in treatment acceptance using ACCEPT at Weeks 24 and
   48
- Reasons for continuation of receiving injectable HIV treatment at Baseline (Day 1) visit. This is an exploratory endpoint.
- Reasons for switching to injectable HIV treatment at Baseline (Day 1) visit. This is an exploratory endpoint.

## 12.2. Summary Measure

Mean treatment difference (Q8W - Q4W) at visits of interest, except for Preference between LA injection every 8 weeks and LA injection every 4 weeks at Week 48.

## 12.3. Population of Interest

The health outcomes analyses will mainly be based on the Intent-to-Treat Exposed population, unless otherwise specified.

Analysis of Reason for continuation will be based on a subset of the Intent-to-Treat Exposed population who were randomized to Q4W arm in ATLAS (i.e. ATLAS Q4W population).

Analysis of Reason for switch will be based on a subset of Intent-to-Treat Exposed population who either were randomized to SOC arm in ATLAS or did not participate in ATLAS study (i.e. SOC population).

# 12.4. Strategy for Intercurrent (Post-Randomization) Events

If a participant discontinues treatment prior to the timepoint of interest such that there is no evaluable assessment for the timepoint of interest, the data will be computed or imputed (see Section 15.6.6).

# 12.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 14: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 12.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 12.5.1. Statistical Methodology Specification

#### Statistical Analyses

#### **Endpoints**

- Change from Baseline in
  - HIVTSQs total treatment satisfaction score at Weeks 24 and 48
  - ACCEPT general acceptance score at Weeks 24 and 48
  - o HAT-QoL (Life satisfaction, HIV medications, disclosure worries) at Weeks 24 and 48

| | | , | , | |
|---|-------------|------------------------------------------------|-----|-----|
| • | Change fror | n Week 8 in PIN Domain Scores ( <sup>CCI</sup> | , 6 | and |
| | CCI | and Individual Items Scores ( | | |
| | CCI | at Weeks 24 and 48 | | |

## **Model Specification**

- The analysis for HIVTSQs, ACCEPT and HAT-QoL will be performed for subjects with and without prior exposure to CAB+RPV separately.
  - For subjects without prior exposure to CAB+RPV, an analysis of covariance (ANCOVA) model will be used at each visit during the maintenance phase with covariates: treatment, age (<50, ≥ 50 years old), sex at birth, race (i.e. white, nonwhite) and baseline score value for other endpoints (as a continuous variable).
  - For subjects with prior exposure to CAB+RPV, an analysis of covariance (ANCOVA) model will be used at each visit during the maintenance phase with covariates: treatment, age (<50, ≥ 50 years old), prior exposure to CAB+RPV (i.e. 1 to 24 weeks, >24 weeks), sex at birth, race (i.e. white, non-white) and baseline score value (as a continuous variable).
- For PIN, an analysis of covariance (ANCOVA) model will be used at each visit during the
  maintenance phase with covariates: treatment, age (<50, ≥ 50 years old), prior exposure to
  CAB+RPV (i.e. 0 weeks, 1 to 24 weeks, >24 weeks), sex at birth, race (i.e. white, non-white),
  and Week 8 score value (as a continuous variable).
- Adjusted point estimates will be derived as LSMEANS using the observed margins (OM) option within PROC MIXED in SAS.
- The superiority testing of Q8W compared to Q4W with respect to change from baseline in HIVTSQs total score at Week 48 will be performed using the fixed sequence procedure to control for the type I error rate at the nominal level of 5%. If the superiority testing within subjects without prior exposure to CAB+RPV demonstrates Q8W is superior to Q4W in change from baseline in HIVTSQs total score at Week 48 at two-sided 5% level of significance, the superiority testing at the same level of significance (i.e. two-sided 5%) within subjects with prior exposure to CAB+RPV will be followed. No adjustment for multiplicity will be applied for other tests as they will be considered supportive.
- Interactions between treatment and each of the covariates will not be assessed unless the
  exploratory subgroup analyses on the primary endpoint highlights significant interactions. In
  this situation, the interaction(s) of interest will be assessed and, if necessary, results will be
  reported in the clinical study report. Interactions between treatment and the baseline score will
  be investigated but not included in the model. If interactions are found to be significant
  (p<0.10), results may be presented separately by subgroup.</li>

#### **Dataset**

LOCF dataset will be used.

#### **Model Results Presentation**

## **Statistical Analyses**

- Adjusted treatment difference (Q8W Q4W), its 95% CI and the associated p-value. The
  interaction between treatment and the baseline score will be included in a footnote.
- Plots of adjusted mean change from baseline (95% CI) for each treatment group, and the adjusted mean difference (95%CI) between the two treatment arms from the model will be generated across visit.

#### **Statistical Analyses**

## **HIVTSQc**

• Total Treatment Satisfaction Score (Change) at Week 48

## **Model Specification**

- An analysis of variance (ANOVA) model will be used with covariates: treatment, age (<50, ≥ 50 years old), prior exposure to CAB+RPV (i.e. 0 weeks, 1 to 24 weeks, >24 weeks), sex at birth and race (i.e. white, non-white).
- Adjusted point estimates will be derived as LSMEANS using the observed margins (OM) option within PROC MIXED in SAS.
- Interactions between treatment and each of the covariates will not be assessed unless the
  exploratory subgroup analyses on the primary endpoint highlights significant interactions. In this
  situation, the interaction(s) of interest will be assessed and, if necessary, results will be
  reported in the clinical study report. If interactions are found to be significant (p<0.10), results
  may be presented separately by subgroup.</li>
- No adjustment for multiplicity will be applied as these analyses will be considered supportive.

#### Dataset

The observed case (OC) dataset uses only the data that is available at Week 48, with no imputation for missing values.

## **Model Results Presentation**

Adjusted means, 95% CI, and associated p-value will be presented for the treatment difference (Q8W – Q4W).

## **Statistical Analyses**

#### PIN

Change from Week 8 in the PIN acceptance score at Week 24 and Week 48

#### **Statistical Test**

• The Wilcoxon Signed-Rank Test will be used to evaluate whether the change from Week 8 to Week 24 and to Week 48, respectively, is statistically different than zero based on a two-sided p<0.05. Separate tests will be performed for the change from Week 8 to Week 24 and for the change from Week 8 to Week 48.

#### **Dataset**

LOCF dataset will be used.

#### **Results Presentation**

 Summary statistics at each timepoint (Week 8, Week 24 and W48) and p-value for each comparison between scores at Week 24/48 with scores at Week 8.

## 13. VIROLOGY

The virology analyses will mainly use genotype and phenotype data based on plasma sample for CVF population, unless otherwise specified. Additional analyses for HIV-1 resistance may be carried out on peripheral blood mononuclear (PBMC) samples collected at Day 1, Week 48, Week 96, or Withdrawal if prior to Week 96.

If pre-treatment genotypic/phenotypic results are available from both the central laboratory and Monogram Biosciences, then Baseline genotype/phenotype will be determined based only upon the data provided by Monogram assays.

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 7 Overview of Planned Virology Analyses

| Endpoint | | Abs | solute | |
|---|---|---|---|---|
| | Sun | nmary | Indivi | dual |
| | T | F | F | L |
| Genotypic resistance at time of CVF <sup>[1]</sup> | 1 | | | |
| Prevalence of Resistance Mutations | <b>Y</b> [2] | | | Y |
| Prevalence of Genotypic Susceptibility | Υ | | | |
| Phenotypic resistance at time of CVF[1] | | 1 | | • |
| Prevalence of Phenotype | Y [3] | | | Y |
| Fold Change to CAB and RPV | Υ | | | Υ[4] |
| IN, PR/RT Replication Capacity | | | | Υ |
| Other | | | | |
| Viral load, Genotypic and Phenotypic data for Participants with genotype and/or phenotype data for CVF and non-CVF participants | | | | Υ[4] |
| Net Assessment | Υ | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- 1. For the CVF as indicated by two consecutive plasma HIV-1 RNA levels ≥200 c/mL after prior suppression to <200 c/mL, the first visit of these two consecutive visits is defined as 'the suspected visit', and the 2nd one is the confirmed visit. Sample used for resistance testing is taken at the suspected visit, and only tested once a participant confirms virological failure at a subsequent visit. If the test fails with the sample at the suspected visit, we will just report it as 'no data'. The sample from the confirmed visit may be used for exploratory analyses.</p>
- 2. No. and percentage of participants with IN resistance mutations or major mutations in the classes of NNRTI, NRTI, PI, respectively, as defined in Section 15.6.7.
- 3. Separate outputs by phenotypic susceptibility and by number of drugs to which participants are phenotypic resistant or partial sensitive or sensitive.
- Fold change to CAB and RPV will be included in the listing for viral load, genotypic and phenotypic data for participants with genotype and/or phenotype data for CVF and non-CVF participants.

## 14. REFERENCES

Chan, I. S. F. and Zhang, Z. (1999), "Test-Based Exact Confidence Intervals for the Difference of Two Binomial Proportions," Biometrics, 55, 1202–1209.

Chevat C, Viala-Danten M, Dias-Barbosa C, Nguyen VH. Development and psychometric validation of a self-administered questionnaire assessing the acceptance of influenza vaccination: the Vaccinees' Perception of Injection questionnaire. Health Qual Life Outcomes. 2008 mar 4; 7:21

D'Agostino RB, Vasan RS, Pencina MJ, et al. General Cardiovascular Risk Profile for Use in Primary Care (The Framingham Heart Study). Circulation 2008; 117: 743-753.

EMA/CHMP/539146/2013, Guideline on the investigation of subgroups in 4 confirmatory clinical trials, 23 January 2014

Fleiss J.L. Statistical Methods for Rates and Proportions. 2nd ed. New York: John Wiley; 1981.

Gilet H, Arnould B. Acceptance by the patients of their treatment (ACCEPT) Questionnaire, 2014.

Grundy S.M., et al. Executive summary of the third report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). JAMA. 2001; 285 (19): 2486-2497.

HIVTSQ user guidelines, Health Psychology Research Unit, Royal Holloway, University of London, 2016

Holmes WC, HIV/AIDS-Targeted Quality of Life Instrument 1999.

Kalbfleisch J.D., Prentice R.L. *The Statistical Analysis of Failure Time Data*. 1st ed. New York: John Wiley & Sons; 1980.

Levey AI, Christopher HS, Hocine T, John HE, Harold IF, Tom G, et al. Esitmating Glomerular Filtration Rate from Serum Creatinine and Cystatin C. N Engl J Med 2012, 367: 20-29.

Lui K.J., Kelly C. A Revisit on Tests for Homogeneity of the Risk Difference, Biometrics, 2000; 56:309-315.

Nilsson ME, Suryawanshi S, Gassmann-Mayer C et al, Columbia–Suicide Severity Rating Scale, Scoring and Data Analysis Guide, 2013.

Sato T. On the variance estimator for the Mantel-Haenszel risk difference. *Biometrics*. 1989; 42:311-323.

Wensing AM et al. Update of the Drug Resistance Mutations in HIV-1 Volume 24 Issue 4 December 2016/January 2017

## 15. APPENDICES

# 15.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

## 15.1.1. Exclusions from Per Protocol Population

Important protocol deviations leading to exclusion from the Per Protocol population are those deviations which may

- directly impact the efficacy endpoint of HIV-1 RNA; or
- lead to permanent discontinuation of IP/withdrawal and hence indirectly impact the efficacy endpoint by causing data to be missing.

The following criteria define the important protocol deviations which, if they occur prior to an analysis timepoint of interest (e.g. Week 48/96), will lead to exclusion of a participant from the Per-Protocol population for that analysis. Potential protocol deviations leading to exclusion from PP population will be reviewed by the study team to confirm that they meet these criteria. A final review will occur before the clinical database has been frozen for analysis.

A participant meeting any of the following criteria will be excluded from the Per Protocol population based on case-by-case clinical determination:

| Number | Exclusion Description |
|---|---|
| 01 | Participant deviates from any inclusion or exclusion criteria that may significantly affect exposure, response to therapy or participant safety or that are fundamentally inconsistent with the intended study population, as recorded in the Protocol Deviation form in the eCRF based on study team review (where indicated in the PDMP as case-by-case determination). |
| | Participant has maintenance phase non-compliance (including IM dosing errors) with investigational product up to an analysis timepoint of interest, meeting one of the following 3 conditions. For Week 48 analysis, the analysis timepoint of interest is the date of last ontreatment viral load up to Study Day 378 during maintenance phase, where Study Day 378 is the upper bound of snapshot window for Week 48 visit. For Week 96 analysis, the analysis timepoint of interest is the date of last on-treatment viral load up to Study Day 714 during the maintenance phase, where Study Day 714 is the upper bound of snapshot window for Week 96 visit. 1. Week 48 analysis only: Two or more injection intervals affected by over dosage deviations, for example |
| 02 | <ul> <li>Extra injection or excessive volume administered.</li> <li>For Q8W participants requiring oral lead-in: length of time between Week 4B injection and Week 8 injection less than 3 weeks, or between injections post Week 8 less than 7 weeks, excluding split doses.</li> <li>For Q8W participants not requiring oral lead-in: length of time between injections less than 7 weeks, excluding split doses.</li> <li>For Q4W participants: length of time between injections less than 3 weeks, excluding split doses.</li> </ul> |
| | 2. Week 96 analysis only: |
| | For participants who permanently discontinued study treatment on/before the |

| Number | Exclusion Description |
|---|---|
| | analysis timepoint of interest for Week 48 analysis (i.e. the date of last on-treatment viral load up to Study Day 378): two or more injection intervals affected by over dosage deviations. |
| | <ul> <li>For participants who received injections beyond the analysis timepoint of interest for Week 48 analysis (i.e. the date of last on-treatment viral load up to Study Day 378): three or more injection intervals affected by over dosage deviations.</li> <li>≥ 10% of total time on-treatment with under dosing deviations. The percentage of total time</li> </ul> |
| | on-treatment with under dosing deviations will be calculated by (the total number of non-compliant dosing days / the total number of intended exposure days) * 100%. |
| | Number of Intended Exposure Days = Date of Last Viral Load – Start Date of Study Treatment + 1, |
| | where the last viral load refers to the last on-treatment viral load up to Study Day 378 during maintenance phase for Week 48 analysis, and the last on-treatment viral load up to Study Day 714 during maintenance phase for Week 96 analysis. |
| | The total number of non-compliant dosing days up to the analysis timepoint visit (or date of IP discontinuation/ withdrawal, whichever is earlier), is derived as follows (summing across all instances): |
| | For Q4W arm participants requiring oral lead-in: |
| | <ul> <li>Length of time (in days) until next injection from date of dosage deviation<br/>(e.g. 2 mL administered instead of 3mL for Week 4B injection, 1ml</li> </ul> |
| | administered instead of 2 mL for post Week 4B injections). Length of time (in days) in excess beyond 35 days between injections post Week 12 and in excess beyond 28 days for Week 8 and Week 12 (e.g. missed or late injection visit). |
| | <ul> <li>Length of time (in days) in excess beyond 35 days from last injection until<br/>start of oral bridging post Week 12 and in excess beyond 28 days for<br/>Week 8 and Week 12.</li> </ul> |
| | For Q4W arm participants not requiring oral lead-in: |
| | <ul> <li>Length of time (in days) until next injection from date of dosage deviation<br/>(e.g. 1 mL administered instead of 2 mL).</li> </ul> |
| | Length of time (in days) in excess beyond 35 days between injections. Length of time (in days) in excess beyond 35 days between injections until |
| | <ul> <li>Length of time (in days) in excess beyond 35 days from last injection until<br/>start of oral bridging post Week 12.</li> </ul> |
| | For Q8W arm participants requiring oral lead-in: anoth of time (in days) until post injection from date of decays deviation. |
| | <ul> <li>Length of time (in days) until next injection from date of dosage deviation<br/>(e.g. 2 mL administered instead of 3mL).</li> </ul> |
| | <ul> <li>Length of time (in days) in excess beyond 63 days between injections post<br/>Week 16 and in excess beyond 56 days for Week 8 and Week 16 (e.g.</li> </ul> |
| | missed or late injection visit). Length of time (in days) in excess beyond 63 days from last injection until start of oral bridging post Week 16 and in excess beyond 56 days for Week 8 and Week 16. |
| | For Q8W arm participants not requiring oral lead-in: |
| | <ul> <li>Length of time (in days) until next injection from date of dosage deviation<br/>(e.g. 2 mL administered instead of 3 mL).</li> </ul> |
| | Length of time (in days) in excess beyond 63 days between injections. Length of time (in days) in excess beyond 63 days from last injection until |
| | <ul> <li>Length of time (in days) in excess beyond 63 days from last injection until</li> </ul> |

| Number | Exclusion Description |
|---|---|
| | start of oral bridging post Week 16. Interrupted days in oral study treatment (oral lead-in or oral bridging) if the oral dose has been interrupted for 3 or more consecutive days and the primary interruption reason is not adverse event or laboratory abnormality (based on the eCRF Exposure forms). 3 days will be assumed if such interrupted days are not available in the database. |
| 03 | Prohibited medications: receiving ART medication other than that prescribed/allowed by the study (excluding permanent changes in ART regimen; such cases will be retained as 'HIV1-RNA ≥50 c/mL' in the per protocol snapshot analysis) or receiving prohibited concomitant medication that would impact exposure or response to therapy with duration and route of administration taken into consideration, as recorded in the Protocol Deviation form in the eCRF based on study team review (where indicated in the PDMP as case-by-case determination). |
| 04 | Permanent discontinuation of IP/withdrawal due to a reason of "Protocol Deviation" (as recorded in the eCRF). |
| 05 | Other important protocol deviations that exclude Participant from Per protocol population as recorded in the Protocol Deviation form in the eCRF based on study team review (where indicated in the PDMP as case-by-case determination). |

## 15.2. Appendix 2: Schedule of Activities

While some assessments included in the Time and Events Table are conducted less frequently following the primary endpoint (Week 48), IM injections for participants during the Extension Phase will continue to be administered Q4W or Q8W based on original study randomization assignment.

All patients will be randomized at Day 1 to initiate either Q4 weekly or Q8 weekly administration of IM CAB LA + RPV LA. Only participants randomized from oral SOC treatment will participate in the Day 1 to Week 4 Oral CAB + Oral RPV lead-in treatment.

# 15.2.1. Protocol Defined Schedule of Events for Q4W Arm

| | æ | | | | | | | | N | Iainter | nance ] | Phase | | | | | | | | | | nsion<br>ase | 7 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | | | | | | | | | | | Wee | ek | | | | | | | | | | awal<br>ients <sup>y</sup> | erm<br>z |
| Procedure | Screening Visit a | Day 1 | Week 4A<br>(Oral Lead-in<br>ONLY) <sup>b</sup> | Week 4B | <b>&amp;</b> | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | Q4W<br>56-92 | Q8W<br>56-92 | 96 | 100 | Q4W<br>After<br>Wee<br>k 100 | Q8W<br>After<br>Week<br>96 | Withdrawal<br>Assesssments <sup>y</sup> | Long-Term<br>Follow-up <sup>Z</sup> |
| Written informed consent | X | | | | | | | | | | | | | | | | | | | | | | | |
| Eligibility Verification (Inclusion/E xclusion Criteria) | X | | Xc | | | | | | | | | | | | | | | | X | | | | | |
| Randomization | 37 | X | | | | | | | | | | | | | | | | | | | | | | |
| Demography<br>Medical<br>History <sup>d</sup> | X | | | | | | | | | | | | | | | | | | | | | | | |
| Cardiovascular<br>risk<br>assessment <sup>d</sup> | X | X | | | | | | | | | | | | | | | | | | | | | | |
| Medication<br>History/<br>Prior ART<br>history | X | | | | | | | | | | | | | | | | | | | | | | | |
| Syphilis<br>serology +<br>Reflex Rapid<br>Plasma<br>Reagin<br>(RPR) | X | X | | | | | | | | | | | | | | | | | | | | | | |

| | t a | | | | | | | | N | Iainter | nance ] | | | | | | | | | | | nsion<br>ase | y | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit a | | | | | | | | | | | Wed | ek | | | | | | | | | | awal<br>ents | erm<br>up <sup>z</sup> |
| Procedure | Screening | Day 1 | Week 4A<br>(Oral Lead-in<br>ONLY) <sup>b</sup> | Week 4B | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | Q4W<br>56-92 | Q8W<br>56-92 | 96 | 100 | Q4W<br>After<br>Wee<br>k 100 | Q8W<br>After<br>Week<br>96 | Withdrawal<br>Assesssments | Long-Term<br>Follow-up <sup>Z</sup> |
| Symptom Directed Physical Exam and Medical Assessment | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Weight,<br>Height and<br>BMI <sup>f</sup> | | X | | | | | | | | | | | | | X | | | | X | | | | X | |
| Vital Signs:<br>BP, HR,<br>Temperature) <sup>g</sup> | X | X | | | | | | | | | | | | | X | | | | X | | | | X | |
| 12-lead ECG<br>h<br>(triplicate at<br>Day 1 pre-dose) | X | X | | | | | | | | | | | | | X | | | | X | | | | X | |
| CDC HIV-1 stage | X | X | | | | | | | | | | | | | | | | | | | | | | |
| HIV<br>Associated<br>Conditions | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| AEs, SAEs,<br>Concomitant<br>Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

| | isit <sup>a</sup> | | | | | | | | N | <b>Iainte</b> i | nance ] | Phase<br>We | ek | | | | | | | | | nsion<br>ase | al<br>ts y | m z |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening Visit | Day 1 | Week 4A<br>(Oral Lead-in<br>ONLY) <sup>b</sup> | Week 4B | <b>&amp;</b> | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 84 | 52 | Q4W<br>56-92 | Q8W<br>56-92 | 96 | 100 | Q4W<br>After<br>Wee<br>k 100 | Q8W<br>After<br>Week<br>96 | Withdrawal<br>Assessments | Long-Term<br>Follow-up <sup>Z</sup> |
| ISR<br>Assessment<br>for IM<br>injections | | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Columbia<br>Suicide<br>Severity<br>Rating Scale<br>(eC-SSRS) <sup>j</sup> | X | X | | X | X | | X | | X | | X | | X | | X | | | X | X | | | | X | |
| Clinical<br>chemistry<br>and<br>Hematology | X | X | X | X | X | | X | | X | | X | | X | | X | | | X | X | X | | X | X | X |
| Pregnancy<br>Testing <sup>k</sup> | S | U | S | U | S | U | S | U | S | U | S | U | S | U | S | S | U | S | S | S | U | S | S | S |
| HIV-1 RNA<br>and sample<br>for storage<br>(S) <sup>1</sup> | X | X | X | X | X | | X | | X | | X | | X | | X | S | | X | X | S | | X | X | X |
| CD4+ cell count | X | X | | X | X | | X | | X | | X | | X | | X | | | X | X | | | X | X | X |
| CD8+ cell<br>count | | X | | | | | | | X | | | | | | X | | | | X | | | | X | |
| Urinalysis <sup>m</sup> | | X | X | | | | | | X | | | | | | X | | | | X | | | | X | |

| | isit <sup>a</sup> | | | | | | | | N | lainter | nance l | Phase<br>Wee | ek | | | | | | | | | nsion<br>ase | ral<br>ts y | m z ( |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening Visit a | Day 1 | Week 4A<br>(Oral Lead-in<br>ONLY) <sup>b</sup> | Week 4B | <b>∞</b> | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | Q4W<br>56-92 | Q8W<br>56-92 | 96 | 100 | Q4W<br>After<br>Wee<br>k 100 | Q8W<br>After<br>Week<br>96 | Withdrawal<br>Assessments | Long-Term<br>Follow-up <sup>Z</sup> |
| Fasting Lab Assessment: Glucose, Cholesterol (Total, HDL and LDL) and Triglycerides | | X | | | | | | | | | | | | | X | | | | X | | | | Xº | |
| Hepatitis B (HBsAg), Anti-HBc, and Anti- HBsAG, Hepatitis C (anti-HCV Ab) | X | | | | | | | | | | | | | | | | | | | | | | | |
| PT/PTT/INR<br>PBMCs <sup>p</sup> | X | X | | | | | | | | | | | | | X | | | | X | | | | X | |
| Genetics sample q | | X | | | | | | | | | | | | | Λ | | | | Λ | | | | Λ | |
| PK sampling <sup>r</sup> (S)=Storage only | | | | X | X | S | X | S | X | S | X | S | X | S | X | S | S | S | X | S | | | X | S |

| | 'isit <sup>a</sup> | | | | | | | | N | <b>Iaint</b> ei | nance ] | Phase<br>We | ek | | | | | | | | | nsion<br>ase | val<br>nts <sup>y</sup> | rm<br>Z d |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening Visit a | Day 1 | Week 4A<br>(Oral Lead-in<br>ONLY) <sup>b</sup> | Week 4B | <b>&amp;</b> | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | Q4W<br>56-92 | Q8W<br>56-92 | 96 | 100 | Q4W<br>After<br>Wee<br>k 100 | Q8W<br>After<br>Week<br>96 | Withdrawal<br>Assessments <sup>y</sup> | Long-Term<br>Follow-up <sup>Z</sup> |
| Oral CAB<br>and Oral<br>RPV<br>Dispensation <sup>S</sup> | | X | X | | | | | | | | | | | | | | | | | | | | | |
| IP accountability (Pill Counts) <sup>S</sup> | | | X | X | | | | | | | | | | | | | | | | | | | | |
| IM treatment administratio n when transitioning from SOC <sup>t</sup> | | | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| IM treatment<br>administration<br>when<br>transitioning<br>from CAB +<br>RPV LA<br>Q4W | | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| | | | | | | | | | I | Patient | Repo | rted O | utcom | es <sup>u</sup> | | | | | | • | | | | |
| HAT-QoL<br>(short-form) | | X | | | | | | | X | | | | | | X | | | | | | | | X | |
| HIV TSQs<br>HIV TSQc <sup>v</sup> | | X | | | | | | | X | | | | | | X | | | | | | | | X | |
| ACCEPT | | X | | | | | | | X | | | | | | X | | | | | | | | X | |

| | Visit a | | | | | | | | N | <b>Iainte</b> i | nance | Phase<br>We | ek | | | | | | | | | nsion<br>ase | awal<br>ents <sup>y</sup> | erm<br>up <sup>Z</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening | Day 1 | Week 4A<br>(Oral Lead-in<br>ONLY) <sup>b</sup> | Week 4B | <b>∞</b> | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | Q4W<br>56-92 | Q8W<br>56-92 | 96 | 100 | Q4W<br>After<br>Wee<br>k 100 | Q8W<br>After<br>Week<br>96 | Withdraw<br>Assesssmen | Long-Teri<br>Follow-up |
| Reason for<br>Switch or<br>Reason for<br>continuation w | | X | | | | | | | | | | | | | | | | | | | | | | |
| Preference x | | | | | | | | | | | | | | | X | | | | | | | | X | |
| PIN | | | | | X | | | | X | | | | | | X | | | | | | | | X | |

Safety Follow Up Visit: Conduct approximately 4 weeks after the last dose of IP. Required only if the participant has ongoing AEs or lab abnormalities at the last on-study visit. This visit may be conducted by telephone.

- a. Complete all Screening assessments within 35 days. Participants may begin the Maintenance Phase as soon as all Screening assessments are complete. Participants may be rescreened once and will be assigned a new participant number. Participants transitioning from the 201585 (ATLAS) study must reach ATLAS Week 48 (at minimum) prior to initiating Screening procedures for ATLAS-2M and must reach ATLAS Week 52 (at minimum) prior to randomization in ATLAS-2M.
- b. Visits Week 4a is part of the CAB + RPV Oral Lead-in period and is required only for participants transitioning from current SOC to CAB LA + RPV LA.
- c. Confirmation of eligibility to continue the Maintenance Phase and eligibility to enter the Extension Phase.
- d. Collect full routine medical history plus (report at Baseline visit): HIV risk factors (may be collected at a later study visit), cardiovascular risk factors (assessments include smoking status and history, family history of cardiac events), recent [≤6 months] illicit drug use, intravenous drug use, gastrointestinal disease, metabolic, psychiatric, renal, bone, and neurologic disorders.
- e. Physical exams should be conducted as part of normal routine clinical care. Medical assessments include any decisions the study staff must make for participants management and/or care of participant.
- f. Height collected at Baseline Day 1 only.
- g. Measure vital signs after about 5 minutes of rest in a semi-supine position.

- h. A 12-lead ECG will be performed after resting in a semi-supine position for at least 5 minutes. ECGs will be performed pre-dose. For participants transitioning from ATLAS, the pre-dose Week 48 ECG can also serve as the ATLAS-2M Screening ECG. ECG pre-dose will be performed in triplicate at Day 1. A 2-hour post-dose ECG will also be performed at Days 1 and Week 48 for participants receiving CAB LA + RPV LA with an allowable window of ±30 minutes.
- i. Only SAEs related to study participation or to a concomitantly administered ViiV/GSK product will be collected between obtaining informed consent and administration of study drug at Day 1.
- j. On Day 1, the eC-SSRS is to be administered prior to randomization. The eC-SSRS will preferably be completed at the beginning of the visit following administration of other PROs required prior to injections. The eC-SSRS is not required during the Withdrawal visit if withdrawal occurs during the Extension Phase.
- k. Women of childbearing potential only. SR=serum, UR=urine. Pregnancy events will be captured starting at Day 1 following initial exposure to study drug. Urine pregnancy test performed at Day 1 prior to administration of study drug, at Week 4B, and at study visits when other blood draws are not required in order to limit needle sticks. Serum pregnancy test can substitute for urine pregnancy test if locally required but must be appropriately timed to confirm pregnancy status prior to randomization and first IM administration.
- 1. Week 48 and Week 96 HIV-1 RNA retest (within 4 weeks) for results > 50 c/mL will be captured as unscheduled visit. Plasma for storage samples will be used for possible future analyses.
- m. A morning specimen is preferred. To assess biomarkers: urine albumin/creatinine ratio; urine protein/creatinine ratio; and urine phosphate. Urine phosphate results from visit 4a are not required by protocol to inform the safety review at visit 4b prior to receipt of initial CAB LA + RPV LA injections.
- n. An overnight fast is preferred; however, a minimum of a 6-hour fast is acceptable.
- o. Only collect if the Withdrawal visit occurs at Week 48 or Week 96.
- p. Whole blood/PBMC collection samples may be used for virologic analyses. PBMCs will be collected at baseline Day 1, Week 48, Week 96, or Withdrawal if prior to Week 96.
- q. Genetics sample should be collected only for patients who did not participate in the 201585(ATLAS) study (sample was previously collected and stored). Informed consent for genetic research must be obtained before sample collection. Sample may be collected at any visit after signing informed consent, but preferably at the Day 1 visit.
- r. One blood sample for CAB and RPV each to be collected at each PK timepoint. At Day 1, for participants from the ATLAS Q4W arm, PK samples are to be collected pre-dose relative to IM administration. At Week 4B, for participants randomized from SOC, Pre dose PK samples are to be collected: AFTER review of the PK diary to ensure that the samples are taken 20/28 hours after previous oral dose (diaries to be given at *Day 1 or W4a*); PRIOR to the final oral dose of CAB + RPV; PRIOR to the first IM injection.
- s. Only for Participants entering CAB + RPV Oral Treatment
- t. Participants switching to CAB LA + RPV LA will take final dose of oral lead-in regimen in the clinic at the Week 4B visit and begin injections. If possible, injections should be spaced approximately 2 cm from one another and from the site of any previous injection and or any injection site reaction. Bring RPV LA

- to approximately room temperature prior to injecting. Time and location of injection (right or left) as well as needle length used will be collected in the eCRF. The first injection can be performed as soon as central lab results become available and safety parameters are reviewed.
- u. All Patient Report Questionnaires/Surveys will be administered via paper instrument at the beginning of the visit before any other assessments are conducted and prior to administration of the eC-CSSRS. Conduct questionnaires/surveys at Withdrawal only if occurring at or prior to Week 48.
- v. The HIV-TSQc is to be administered to all participants transitioning from ATLAS and new participants transitioning from oral SOC. For participants transitioning from ATLAS, the version of the HIV-TSQc instrument to be administered will be based on the initial randomization arm at ATLAS Day 1.
- w. For patients randomized to oral SOC at Day 1 in ATLAS or new patients on SOC, the reasons for willingness to switch ART will be assessed at Day 1. For patients randomized to CAB LA + RPV LA Q4W in ATLAS, the reasons for willingness to continue long-acting ART in ATLAS-2M will be assessed at Day 1.
- x. Preference Questionnaire will be administered to all participants.
- y. Refer to Section 5.5 of the protocol for additional information on performing withdrawal assessments. HIV-1 RNA will be collected as Storage sample only if withdrawal assessments coincide with Week 52 or Week 100 (as per Section 5.5)
- z. Participants receiving one or more injections with CAB LA and/or RPV LA will be assessed with clinic visits at months 3, 6, 9 and 12 during the Long-Term Follow-Up Phase

Note: BP – Blood pressure, HR – Heart Rate, HDL – High Density Lipoprotein, LDL – Low Density Lipoprotein, PT Prothrombin Time, PTT Partial Thromboplastin Time, INR International normalized ratio

## 15.2.2. Protocol Defined Schedule of Events for Q8W Arm

| | | | | | | | | | I | Mainte | nance l | Phase | | | | | | | | Extension<br>Phase | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit <sup>a</sup> | | | | | | | | | | | Wee | k | | | | | | | riiase | awal<br>ents <sup>y</sup> | erm<br>up z |
| Procedure | Screening Visit | Day 1 | Week 4A<br>(Oral lead-in<br>ONLY) b | Week 4B<br>(Oral lead-in<br>ONLY) b | ∞ | 6 | 16 | 24 | 32 | 40 | 41 | 48 | 99 | 64 | 72 | 08 | 88 | 96 | 100 | Q8W After<br>Week 96 | Withdrawal<br>Assessments <sup>y</sup> | Long-Term<br>Follow-up z |
| Written informed consent | X | | | | | | | | | | | | | | | | | | | | | |
| Eligibility Verification (Inclusion/ Exclusion Criteria) | X | | X <sup>c</sup> | | | | | | | | | | | | | | | X <sup>c</sup> | | | | |
| Randomization | | X | | | | | | | | | | | | | | | | | | | | |
| Demography | X | | | | | | | | | | | | | | | | | | | | | |
| Medical<br>History <sup>d</sup> | X | | | | | | | | | | | | | | | | | | | | | |
| Cardiovascular<br>risk<br>assessment <sup>d</sup> | X | X | | | | | | | | | | | | | | | | | | | | |
| Medication<br>History/ Prior<br>ART history | X | | | | | | | | | | | | | | | | | | | | | |
| Syphilis<br>serology +<br>reflex Rapid<br>Plasma<br>Reagin (RPR) | X | X | | | | | | | | | | | | | | | | | | | | |

| | t a | | | | | | | | N | Mainte | nance l | Phase | | | | | | | | Extension<br>Phase | 1 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visi | | | | | | | | | | | Wee | k | | | | | | | | awal<br>nents <sup>3</sup> | Term<br>-up z |
| Procedure | Screening Visit | Day 1 | Week 4A<br>(Oral lead-in<br>ONLY) b | Week 4B<br>(Oral lead-in<br>ONLY) b | œ | 6 | 16 | 24 | 32 | 40 | 41 | 48 | 99 | 64 | 72 | 08 | 88 | 96 | 100 | Q8W After<br>Week 96 | Withdrawal<br>Assessments <sup>y</sup> | Long-Term<br>Follow-up z |
| Symptom Directed Physical Exam and Medical Assessment | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Weight, Height and BMI <sup>f</sup> | | X | | | | | | | | | | X | | | | | | X | | | X | |
| Vital Signs<br>(BP, HR,<br>Temperature) <sup>g</sup> | X | X | | | | | | | | | | X | | | | | | X | | | X | |
| 12-lead ECG h (triplicate at Day 1 pre-dose) | X | X | | | | | | | | | | X | | | | | | X | | | X | |
| CDC HIV-1 stage | X | X | | | | | | | | | | | | | | | | | | | | |
| HIV<br>Associated<br>Conditions | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| AEs, SAEs,<br>Concomitant<br>Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| ISR<br>Assessment<br>for IM<br>injection | | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

| | t a | | | | | | | | ľ | Mainte | nance l | Phase | | | | | | | | Extension<br>Phase | 1 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visi | | | | | | | | | | | Wee | k | | | | | | | | awal<br>nents <sup>3</sup> | rerm<br>-up z |
| Procedure | Screening Visit | Day 1 | Week 4A<br>(Oral lead-in<br>ONLY) b | Week 4B<br>(Oral lead-in<br>ONLY) b | <b>∞</b> | 6 | 16 | 24 | 32 | 40 | 41 | 48 | 99 | 64 | 72 | 80 | 88 | 96 | 100 | Q8W After<br>Week 96 | Withdrawal<br>Assessments <sup>y</sup> | Long-Term<br>Follow-up z |
| Columbia<br>Suicide<br>Severity<br>Rating Scale<br>(eC-SSRS) <sup>j</sup> | X | X | | X | X | | X | X | X | X | | X | X | X | X | X | X | X | | | X | |
| Clinical<br>chemistry and<br>Hematology | X | X | X | X | X | | X | X | X | X | | X | X | X | X | X | X | X | X | X | X | X |
| Pregnancy<br>Testing <sup>k</sup> | S | U | S | U | S | | S | S | S | S | | S | S | S | S | S | S | S | S | S | S | S |
| HIV-1 RNA<br>and sample<br>for storage<br>(S) <sup>1</sup> | X | X | | X | X | | X | X | X | X | | X | X | X | X | X | X | X | S | X | X | X |
| CD4+ cell<br>count | X | X | | X | X | | X | X | X | X | | X | X | X | X | X | X | X | X | X | X | X |
| CD8+ cell<br>count | | X | | | | | | X | | | | X | | | | | | X | | | X | |
| Urinalysis <sup>m</sup> | | X | X | | | | | X | | | | X | | | | | | X | | | X | |
| Fasting Labs Glucose, Cholesterol (Total, HDL and LDL) and Triglycerides | | X | | | | | | | | | | X | | | | | | X | | | Xº | |

| | a . | | | | | | | | ľ | Mainte | nance l | Phase | | | | | | | | Extension<br>Phase | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | | | | | | | | | | | Wee | k | | | | | | | | awal<br>ients <sup>y</sup> | cerm<br>cup z |
| Procedure | Screening Visit | Day 1 | Week 4A<br>(Oral lead-in<br>ONLY) b | Week 4B<br>(Oral lead-in<br>ONLY) b | <b>&amp;</b> | 6 | 16 | 24 | 32 | 40 | 41 | 48 | 99 | 64 | 72 | 80 | 88 | 96 | 100 | Q8W After<br>Week 96 | Withdrawal<br>Assessments <sup>y</sup> | Long-Term<br>Follow-up z |
| Hepatitis B<br>(HBsAg),<br>Anti-HBc, and<br>Anti-HBsAG,<br>Hepatitis C<br>(anti-HCV<br>Ab) | X | | | | | | | | | | | | | | | | | | | | | |
| PT/PTT/INR | X | X | | | | | | | | | | | | | | | | | | | | |
| PBMCs <sup>p</sup> | | X | | | | | | | | | | X | | | | | | X | | | X | |
| Genetics sample <sup>q</sup> | | X | | | | | | | | | | | | | | | | | | | | |
| PK sampling when transitioning from SOC <sup>r</sup> (S)=Storage only | | | | X | X | X | X | X | X | X | X | X | S | S | S | S | S | X | S | | X | S |
| PK sampling<br>when<br>transitioning<br>from CAB +<br>RPV Q4W <sup>r</sup><br>(S)=Storage<br>only | | X | | | X | X | X | X | X | X | X | X | S | S | S | S | S | X | S | | X | S |
| Oral CAB and<br>Oral RPV<br>Dispensation <sup>s</sup> | | X | X | | | | | | | | | | | | | | | | | | | |

| | a · | | | | | | | | Ι | Mainte | nance ] | Phase | | | | | | | | Extension<br>Phase | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | | | | | | | | | | | Wee | k | | | | | | | | awal<br>ients <sup>y</sup> | erm<br>-up z |
| Procedure | Screening Visit | Day 1 | Week 4A<br>(Oral lead-in<br>ONLY) b | Week 4B<br>(Oral lead-in<br>ONLY) b | <b>∞</b> | 6 | 16 | 24 | 32 | 40 | 41 | 48 | 99 | 64 | 72 | 80 | 88 | 96 | 100 | Q8W After<br>Week 96 | Withdrawal<br>Assessments <sup>y</sup> | Long-Term<br>Follow-up z |
| IP accountability (Pill Counts) | | | X | X | | | | | | | | | | | | | | | | | | |
| IM treatment<br>administration<br>when<br>transitioning | | | | X | X | | X | X | X | X | | X | X | X | X | X | X | X | | X | | |
| from SOC <sup>t</sup> IM treatment administration when transitioning from CAB + RPV Q4W | | X | | | X | | X | X | X | X | | X | X | X | X | X | X | X | | X | | |
| | | | | | | u . | ı | I. | | Patient | t Repo | rted Ou | tcomes | u | u. | | u . | | | | | |
| HAT-QoL<br>(short-form) | | X | | | | | | X | | | | X | | | | | | | | | X | |
| HIV TSQs | | X | | | | | | X | | | | X | | | | | | | | | X | |
| HIV TSQc V ACCEPT | | X | | | | | | X | | | | X | | | | | | | | | X | |
| Reason for<br>Switch or<br>Reason for<br>continuation<br>W | | X | | | | | | | | | | | | | | | | | | | | |
| Preference x | | | | | | | | | | | | X | | | | | | | | | X | |

| | t a | | | | | | | | N | Mainte | nance l | Phase | | | | | | | | Extension<br>Phase | 1 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | y Visi | | | | | | | | | | | Wee | k | | | | | | | | rawal<br>nents <sup>y</sup> | Ferm<br>-up z |
| Procedure | Screening | Day 1 | Week 4A<br>(Oral lead-in<br>ONLY) b | Week 4B<br>(Oral lead-in<br>ONLY) b | ∞ | 6 | 16 | 24 | 32 | 40 | 41 | 48 | 99 | 64 | 72 | 08 | 88 | 96 | 100 | Q8W After<br>Week 96 | Withdı<br>Assessn | Long-7<br>Follow |
| PIN | | | | | X | | | X | | | | X | | | | | | | | | X | |

Safety Follow Up Visit: Conduct approximately 4 weeks after the last dose of IP. Required only if the participant has ongoing AEs or lab abnormalities at the last on-study visit. This visit may be conducted by telephone.

- a. Participants may be rescreened once and will be assigned a new participant number. Participants transitioning from the 201585 (ATLAS) study must reach ATLAS Week 48 (at minimum) prior to initiating Screening procedures for ATLAS-2M and must reach ATLAS Week 52 (at minimum) prior to randomization in ATLAS-2M.
- b. Visits Weeks 4A and 4B are part of the CAB + RPV Oral Lead-in period and are required only for participants transitioning from current SOC to CAB LA + RPV LA.
- c. Confirmation of eligibility to continue the Maintenance Phase, and eligibility to enter the Extension Phase.
- d. Collect full routine medical history plus (report at Baseline visit): HIV risk factors (may be collected at a later study visit), cardiovascular risk factors (assessments include smoking status and history, family history of cardiac events), recent [≤6 months] illicit drug use, intravenous drug use, gastrointestinal disease, metabolic, psychiatric, renal, bone, and neurologic disorders.
- e. Physical exams should be conducted as part of normal routine clinical care. Medical assessments include any decisions the study staff must make for participants management and/or care of participant.
- f. Height collected at Baseline Day 1 only.
- g. Measure vital signs after about 5 minutes of rest in a semi-supine position.
- h. A 12-lead ECG will be performed after resting in a semi-supine position for at least 5 minutes. ECGs will be performed pre-dose. For participants transitioning from ATLAS, the pre-dose Week 48 ECG can also serve as the ATLAS-2M Screening ECG. ECG pre-dose will be performed in triplicate at Day 1. A 2-hour post-dose ECG will also be performed at Days 1 and Week 48 for participants receiving CAB LA + RPV LA with an allowable window of ± 30 minutes.
- i. Only SAEs related to study participation or to a concomitantly administered ViiV/GSK product will be collected between obtaining informed consent and administration of study drug at Day 1.
- j. On Day 1, the eC-SSRS is to be administered prior to randomization. The eC-SSRS will preferably be completed at the beginning of the visit following administration of other PROs required prior to injections. The eC-SSRS is not required during the Withdrawal visit if withdrawal occurs during the Extension Phase.

- k. Women of childbearing potential only. SR=serum, UR=urine. Pregnancy events will be captured starting at Day 1 following initial exposure to study drug. Serum pregnancy test can substitute for urine pregnancy test if locally required but must be appropriately timed to confirm pregnancy status prior to randomization and first IM administration.
- l. Week 48 and Week 96 HIV-1 RNA retest (within 4 weeks) for results > 50 c/mL will be captured as unscheduled visit. Plasma for storage samples will be used for possible future analyses.
- m. A morning specimen is preferred. To assess biomarkers: urine albumin/creatinine ratio; urine protein/creatinine ratio; and urine phosphate. Urine phosphate results from visit 4a are not required by protocol to inform the safety review at visit 4b prior to receipt of initial CAB LA + RPV LA injections.
- n. An overnight fast is preferred; however, a minimum of a 6-hour fast is acceptable.
- o. Only collect if the Withdrawal visit occurs at Week 48 or Week 96.
- p. Whole blood/PBMC collection samples may be used for virologic analyses. PBMCs will be collected at baseline Day 1, Week 48, Week 96, or Withdrawal if prior to Week 96.
- q. Genetics sample should be collected only for patients who did not participate in the 201585(ATLAS) study (sample was previously collected and stored). Informed consent for genetic research must be obtained before sample collection. Sample may be collected at any visit after signing informed consent, but preferably at the Day 1 visit.
- r. One blood sample for CAB and RPV each to be collected at each PK timepoint. At Day 1, for participant from the ATLAS Q4W arm, PK samples are to be collected pre-dose relative to IM administration. injection. At Week 4B, for participants randomized from SOC, Pre dose PK samples are to be collected: AFTER review of the PK diary to ensure that the samples are taken 20/28 hours after previous oral dose (diaries to be given at Day 1 or W4a); PRIOR to the final oral dose of CAB + RPV; and PRIOR to the first IM injection. At Week 9 and 41, the PK samples should be collected 3 to 10 days after the Week 8 and Week 40 visits, respectively.
- s. Only for Participants entering CAB + RPV Oral Treatment
- t. Participants switching to CAB LA + RPV LA will take final dose of oral lead-in regimen in the clinic at the Week 4B visit and begin injections. If possible, injections should be spaced approximately 2 cm from one another and from the site of any previous injection and or any injection site reaction. Bring RPV LA to approximately room temperature prior to injecting. Time and location of injection (right or left) as well as needle length used will be collected in the eCRF. The first injection can be performed as soon as central lab results become available and safety parameters are reviewed.
- u. All Patient Report Questionnaires/Surveys will be administered via paper instrument at the beginning of the visit before any other assessments are conducted and prior to administration of the eC-CSSRS. Conduct questionnaires/surveys upon Withdrawal only if occurring at or prior to Week 48
- v. The HIVTSQc is to be administered to all participants transitioning from ATLAS and new participants transitioning from oral SOC. For participants transitioning from ATLAS, the version of the HIV-TSQc instrument to be administered will be based on the initial randomization arm at ATLAS Day 1
- w. For patients randomized to oral SOC at Day 1 in ATLAS or new patients on SOC, the reasons for willingness to switch ART will be assessed at Day 1. For patients randomized to CAB LA + RPV LA Q4W in ATLAS, the reasons for willingness to continue long-acting ART in ATLAS-2M will be assessed at Day 1.
- x. Preference Questionnaire will be administered to all participants
- y. Refer to Section 5.5 of the protocol for additional information on performing withdrawal assessments. HIV-1 RNA will be collected as Storage sample only if withdrawal assessments coincide with Week 52 or Week 100 (as per Section 5.5)
- z. Participants receiving one or more injections with CAB LA and/or RPV LA will be assessed with clinic visits at months 3, 6, 9 and 12 during the Long-Term Follow-Up Phase

Note: BP – Blood pressure, HR – Heart Rate, HDL – High Density Lipoprotein, LDL – Low Density Lipoprotein, PT Prothrombin Time, PTT Partial Thromboplastin Time, INR International normalized ratio

## 15.3. Appendix 3: Assessment Windows

## 15.3.1. Definitions of Assessment Windows for Analyses

Laboratory data, vital signs, ECGs, health outcomes assessments, and genotypic/phenotypic data will be assigned to assessment windows according to actual dates rather than the nominal visit labels as recorded on the eCRF or in the laboratory database.

In most cases the window around an assessment will include all dates from the midpoints between the target day and that of the previous and the proceeding visits. In general, the nominal target study day for week w is (7\*w)+1.

For parameters which are not scheduled to be assessed at particular visits, the all-inclusive assessment windows will still be used; however, data summaries will only report scheduled visits. Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well any algorithms that make use of additional data (e.g., Snapshot).

Prior to visit slotting, assessments are first assigned to a study phase (screening, maintenance, extension, or long-term follow-up) based on the Tables in Section 15.4.1 and treatment state based on Section 15.4.2.

Maintenance phase assessments other than health outcome and PK are assigned based on the Study Day as shown in Table 8 and Table 10. Table 8 also includes visiting slotting for screening assessments. The analysis visits from Week 4 to Week 100 should be only applied to the assessments that are already assigned to Maintenance phase (on-treatment). Extension phase assessments other than health outcome and PK are assigned based on the Study Day as shown in Table 9. The analysis visits from Week 104 (except for Followup) in the Extension phase should be only applied to the assessments that are already assigned to Extension phase (on-treatment).

Long-term Follow-up phase assessments are assigned based on the LTFU study day as shown in

Table 11. The analysis visits in LTFU should be only applied to the assessments that are already assigned to LTFU phase regardless of treatment state. See Section 15.6.1, for derivation of Study Day and LTFU Study Day.

# 15.3.2. Definitions of Assessment Windows for Analyses other than Health Outcome and PK

 Table 8
 Assessment Windows for Screening and Maintenance Phase Data

| All Parameters except for where noted[c] | Target Study Day | Analysis Window | Analysis Timepoint |
|---|---|---|---|
| | The study day of first record | Study Day ≤ 1 | Screening |
| | 1 | Last available recorded value up to and including the Maintenance treatment start date, excluding 2-hour post-dose ECG taken on the Maintenance treatment start date | Baseline |
| Urinalysis <sup>[a]</sup> | 29 | 2 ≤ Study Day ≤ 70 2 ≤ Study Day ≤ 42, including 2- hour post-dose ECG taken on Maintenance treatment start date | Week 4 |
| | 57 | 43 ≤ Study Day ≤ 84 | Week 8 |
| | 113 | 85 ≤ Study Day ≤ 140 | Week 16 |
| Urinalysis <sup>[a]</sup> , CD8,<br>CD4/CD8 ratio | 169 | 141 ≤ Study Day ≤ 210 | Week 24 |
| | | 141 ≤ Study Day ≤ 196 | |
| | 225 | 197 ≤ Study Day ≤ 252 | Week 32 |
| | 281 | 253 ≤ Study Day ≤ 308 | Week 40 |
| Urinalysis <sup>[a]</sup> , fasting glucose, lipids <sup>[b]</sup> , CD8, CD4/CD8 ratio, weight, vital signs, ECG | 337 | 309 ≤ Study Day ≤ 378 | Week 48 |
| | | 309 ≤ Study Day ≤ 364 | |
| | 393 | 365 ≤ Study Day ≤ 420 | Week 56 |
| | 449 | 421 ≤ Study Day ≤ 476 | Week 64 |
| | 505 | 477 ≤ Study Day ≤ 532 | Week 72 |
| | 561 | 533 ≤ Study Day ≤ 588 | Week 80 |
| | 617 | 589 ≤ Study Day ≤ 644 | Week 88 |
| Urinalysis <sup>[a]</sup> , fasting glucose, lipids <sup>[b]</sup> , CD8, CD4/CD8 ratio, weight, vital signs, ECG | 673 | 645 ≤ Study Day ≤ 714 | Week 96 |
| | | 645 ≤ Study Day ≤ 686 | |
| | 701 | 687 ≤ Study Day ≤ (Study Day of Nominal Week 100 visit) | Week 100 |
| lf a | a participant perman | ently discontinued study treatment | <u> </u> |
| | | For Participants on Q8W Arm: Date > max (Date of Last Oral Dose of CAB+RPV + 1, Date of | Follow-up |

| All Parameters except for where noted[c] | Target Study Day | Analysis Window | Analysis Timepoint |
|---|---|---|---|
| | | Last Injection + 63) | |
| | | For Participants on Q4W Arm: | |
| | | Date > max (Date of Last Oral<br>Dose of CAB+RPV + 1, Date of<br>Last Injection + 35) | |

#### NOTES:

- The nominal Week 100 visit refers to the Week 100 visit per eCRF.
- Follow-up will be derived only for participants who permanently discontinued study treatment.

[a] **Urinalysis:** All parameters provided by the central laboratory under the category of urinalysis, including Urine Albumin/Creatinine, Urine Creatinine, Urine Protein/Creatinine, Urine Erythrocytes, Urine Specific Gravity, Urine Leukocytes, Urine Retinol Binding Protein, Urine Phosphate, Urine Creatinine.

- [b] **Lipids**: Cholesterol, HDL Cholesterol Direct, LDL Cholesterol Calculation, LDL Cholesterol Direct, Total Cholesterol/HDL Cholesterol Ratio, Triglycerides
- [c] Analysis windows for parameters with sparse collection are noted.

#### Table 9 Assessment Windows for Extension Phase Data

| Parameter (if applicable) | Target<br>Study Day | Analysis Window | Analysis Timepoint |
|---|---|---|---|
| All | 729 | (Study Day of Nominal Week 100 visit + 1) ≤ Study Day ≤ 756 | Week 104 |
| | 785 | 757≤ Study Day ≤ 812 | Week 112 |
| | 841 | 813≤ Study Day ≤868 | Week 120 |
| | 7*w + 1 | (7*w - 27)<br>$\leq$ Study Day $\leq$ $(7*w + 28)$ | Week w<br>w = 128, 136, |
| | If a partici | pant permanently discontinued study trea | atment: |
| | | For participants on Q8W Arm: Date > max (Date of Last Oral Dose of CAB+RPV + 1, Date of Last Injection + 63) | Follow-up |
| | | For participants on Q4W Arm: Date > max (Date of Last Oral Dose of CAB+RPV + 1, Date of Last Injection + 35) | r ollow-up |

#### NOTES:

- The nominal Week 100 visit refers to the Week 100 visit per eCRF.
- Follow-up will be derived only for participants who permanently discontinued study treatment.

Table 10 Assessment Windows for Summary of Snapshot Data — Data Assigned to Maintenance Phase Only

| Snapshot Anal (If no on-treatment viral load data in de | <del>-</del> | |
|---|---|---|
| Default | Expanded +6 Week Upper Window <sup>a</sup> | Analysis<br>Timepoint |
| Last available recorded value up to and including the date of first Maintenance Phase dose of IP | Last available recorded value up to and including the date of first Maintenance Phase dose of IP | Baseline |
| 2 ≤ Study Day ≤ 42 | 2 ≤ Study Day ≤ 70 | Week 4 |
| 43 ≤ Study Day ≤ 84 | 43 ≤ Study Day ≤ 98 | Week 8 |
| 85 ≤ Study Day ≤ 140 | 85 ≤ Study Day ≤ 154 | Week 16 |
| 141 ≤ Study Day ≤ 196 | 141 ≤ Study Day ≤ 210 | Week 24 |
| 197 ≤ Study Day ≤ 252 | 197 ≤ Study Day ≤ 266 | Week 32 |
| 253 ≤ Study Day ≤ 308 | 253 ≤ Study Day ≤ 322 | Week 40 |
| 295 ≤ Study Day ≤ 378 | 295 ≤ Study Day ≤ 378 | Week 48 |
| $365 \le \text{Study Day} \le 420$ | 365 ≤ Study Day ≤ 434 | Week 56 |
| 421 ≤ Study Day ≤ 476 | 421 ≤ Study Day ≤ 490 | Week 64 |
| 477 ≤ Study Day ≤ 532 | 477 ≤ Study Day ≤ 546 | Week 72 |
| 533 ≤ Study Day ≤ 588 | 533 ≤ Study Day ≤ 602 | Week 80 |
| 589 ≤ Study Day ≤ 644 | 589 ≤ Study Day ≤ 658 | Week 88 |
| 631 ≤ Study Day ≤ 714 | 631 ≤ Study Day ≤ 714 | Week 96 |

#### NOTES:

- For post-baseline visits (i.e. Week 4 and afterwards), apply Snapshot analysis windows only to viral load data that is on-treatment (per Table 16) within the Maintenance Phase (per Table 14).
- An on-treatment viral load assessment may be assigned to more than one snapshot analysis window, e.g. ontreatment assessment taken on Study Day 300 will be in both Week 40 and Week 48.
- a. ± 6 Week window is always used at key analysis timepoints (Week 48 and Week 96). For analysis timepoint of Week 24, if no viral load data in default window, expand to ± 6 Week window, i.e. (127 ≤ Study Day ≤ 210) in Week 24 IDMC and Week 24 Analyses, and expand upper bound to +6 weeks in all other analyses.

Table 11 Assessment Windows for Summaries of Long-Term Follow Up
Phase Data for Participants Who Received At Least One Injection of
CAB+RPV and Permanently Discontinued Study Treatment

| Analysis Window | Analysis Timepoint | Target Study<br>Day of Window |
|---|---|---|
| 1 ≤ LTFU Study Day ≤ 63 | LTFU Month 1/WD[a] | 30 |
| 64 ≤ LTFU Study Day ≤ 135 | LTFU Month 3 | 90 |
| 136 ≤ LTFU Study Day ≤ 225 | LTFU Month 6 | 180 |
| 226 ≤ LTFU Study Day ≤ 315 | LTFU Month 9 | 270 |
| 316 ≤ LTFU Study Day ≤ 405 | LTFU Month 12 | 360 |
| $(30*m - 44) \le LTFU \text{ Study Day} \le (30*m + 45)$ | LTFU Month m | 7*m |
| | m = 15, 18,21, | |

#### NOTES:

An assessment may be assigned to both LTFU and maintenance/extension phases.

a. For participants who receives at least one injection of CAB+RPV and permanently discontinues study treatment, they will not complete withdrawal visit, will instead move directly into the LTFU and have LTFU Month 1 visit as the first planned LTFU visit per protocol amendment 1; however, per protocol amendment 2, they will complete withdrawal visit and then have LTFU Month 3 visit as the first planned LTFU visit. Data have been collected either per protocol amendment 1 or per protocol amendment 2 and are included in the database. The analysis timepoint of LTFU Month 1/WD is intended for slotting data mainly collected from either

| Analysis Window | Analysis Timepoint | Target Study<br>Day of Window |
|---|---|---|
| LTFU Month 1 visit per protocol amendment 1 or withdrawal visit per protocol amendment 2 if the date of assessments or onset date of event falls within the specified analysis window. | | |

#### 15.3.3. Assessment Window for Phase Conclusion

The 'Phase Conclusion' records in disposition data will be slotted based on Table 8 (for Maintenance Phase conclusion records) and Table 9 (for Extension Phase conclusion records). However, if the discontinuation date is post-treatment per Table 16, the record will be slotted to the last on-treatment visit within the same phase rather than follow up.

## 15.3.4. Assessment Window for Health Outcome Data

#### 15.3.4.1. PIN / HAT-QoL / HIVTSQs / HIVTSQc / ACCEPT / Preference

PIN, HAT-QoL, HIVTSQs, HIVTSQc, ACCEPT and Preference questionnaire assessments will be assigned to analysis visits as follows:

- 1. Baseline will be defined as last available recorded value up to and including the Maintenance treatment start date (expected to be collected at Day 1). Baseline is not applicable for PIN, HIVTSQc and Preference assessments.
- 2. For post-baseline visits, if the nominal visit identifier as captured in the source dataset corresponds to a scheduled collection per the Time and Events Schedule (see Section 15.2 and Table 12) and the assessment is collected in the Maintenance Phase (per Table 14), then the nominal visit identifier will be kept as the analysis visit.
- 3. For post-baseline visits, if the nominal visit identifier is unscheduled or withdrawal, then the following procedure will be used:
  - a) Assign the assessment to a study phase according to Table 14. Proceed to step b if the assessment is assigned to the Maintenance Phase.
  - b) Identify the 'last nominal visit' with the HO assessment performed prior to the unscheduled/withdrawal visit to be slotted.
  - c) The unscheduled/withdrawal visit will be slotted to the planned nominal visit subsequent to the 'last nominal visit'. If the 'last nominal visits' does not exist (e.g. no records originate from a planned nominal visit), then the unscheduled/withdrawal visit will be slot to the first planned nominal visit after Day 1.

Example 1, for HATQoL, the planned nominal visits are Day 1, Week 24, and 48. If a participant has the 'last nominal visit' (with HATQoL assessment) at Week 24 prior to withdrawal at Week 36, the withdrawal assessment will be slotted to the subsequent planned nominal visit of Week 48.

Example 2, for HATQoL, if there is unscheduled visit between Week 24 and Week 48. This unscheduled visit will be slotted to Week 48 per the rule. In this case, there are two assessments with analysis visit equal to Week 48 (i.e. the slotted value and the value at

original nominal week 48 visit). The original nominal value will be selected for summary per the rule below for multiple records—see Section 15.3.6.

Table 12 Planned Nominal Visit of Health Outcome Data

| Questionnaire | Day 1 | Week 8 | Week 24 | Week 48 |
|---|---|---|---|---|
| PIN | | Х | Х | Х |
| HAT-QoL | Х | | Х | Х |
| HIVTSQs | Х | | Х | Х |
| HIVTSQc | | | | Х |
| ACCEPT | Х | | Х | Х |
| Preference | | | | Х |
| NOTES: | | | | |
| Day 1 visits are recorded as "Baseline" visits in the database. | | | | |

#### 15.3.4.2. Reasons for Continuation/Switch

Reasons for Continuation/Switch assessments are planned to be taken at nominal Baseline (Day 1) visit only. The assessments taken within  $\pm$  2 weeks window from maintenance phase treatment start date will be regarded as evaluable. The assessments taken outside this window will be excluded from the summary.

#### 15.3.5. Assessment Window for PK Concentration Data

For PK concentration data at the withdrawal/unscheduled/LTFU Month 1visits during maintenance phase (after assignment to study phase per Table 14), the visit will be slotting to the analysis visit per the following steps:

- Identify the 'last nominal visit' with the PK pre-dose assessment performed prior to the visit to be slotted during the same study phase
- Identify the nominal visit corresponding to the next planned pre-dose PK assessment visit (excluding visits with storage PK collection), that is subsequent to the 'last nominal visit' with PK pre-dose assessment during the same study phase.
- If the nominal visit corresponding to next planned pre-dose PK assessment visit is prior to/at Week 48 visit, the PK assessment at the unscheduled/withdrawal/LTFU Month1 visit will be slotted to this nominal visit corresponding to next planned pre-dose PK assessment visit.
- Otherwise, the PK assessment at the unscheduled/withdrawal/LTFU Month1 visit will be slotted to the earliest nominal visit from the following:
  - Nominal visit corresponding to the next planned pre-dose PK assessment visit
  - The nominal visit of the next planned injection occurring on or after the date of the PK assessment during the same study phase

During maintenance phase, the planned nominal visits for PK Pre-dose are Week 4B, 8, 16, 24, 32, 40, 48, 96 for Q4W arm; and are Day 1, Week 4B, 8, 16, 24, 32, 40, 48, 96 for

Q8W arm while Day 1 is required only for those transitioning from ATLAS on Q4W injections and Week 4B is required only for participants transitioning from oral SOC and requiring oral CAB+RPV lead-in. In addition, the participants on Q8W arm have planned nominal visits at Week 9 and 41 for 1-week post-dose.

For participants requiring oral CAB+RPV lead-in, the planned injection visits are Week 4B, Week 8, continuing every 4 weeks for Q4W arm and continuing every 8 weeks for Q8W arm. For participants not requiring oral CAB+RPV lead-in, the planned injection visits are every 4 weeks starting from Day 1 for Q4W arm and every 8 weeks starting from Day 1 for Q8W arm.

Example 1: If a participant on Q8W arm has the 'last nominal visit' (with PK pre-dose assessment) at Week 24 and then withdraws around Week 28, with the last injection at Week 24 and a Maintenance Phase PK assessment labelled at 'LTFU Month 1'., This PK assessment labelled as 'LTFU Month 1' will be slotted to the subsequent planned nominal visit of Week 32.

Example 2: If a participant on Q4W arm has the 'last nominal visit' (with PK pre-dose assessment) at Week 48 and then have an unscheduled Maintenance Phase PK assessment around Week 74. This assessment will be slotted to the next planned injection visit, Week 76.

There will be no slotting for planned nominal visits (i.e. analysis visit =visit).

## 15.3.6. Multiple Assessments within an Assessment Window

If after window assignment there are multiple valid assessments of a parameter within the same window, then the following hierarchy will be used to determine the value to be used for summary statistics of observed values:

For data other than health outcome/PK concentration:

- 1. the assessment closest to the window target Study Day;
- 2. if there are multiple assessments equidistant from the target Study Day, then the mean of these values will be used. For HIV-1 RNA, the geometric mean of the number of copies will be used as opposed to the arithmetic mean.

For Health outcome and PK concentration data, the following hierarchy will be used to determine the value to be used for summary statistics of observed values:

- 1. If there are multiple on-treatment assessments assigned to the same analysis visit, the assessment from the planned nominal visit will be used for summary statistics.
- 2. If there are multiple on-treatment assessments assigned to the same analysis visit and none originates from a planned nominal visit (e.g. two unscheduled/withdrawal nominal visits), then
  - a. the assessment closest to the window target Study Day will be used;
  - b. if there are multiple assessments equidistant from the target Study Day, then the earliest assessment will be used.
Assessments not chosen for use in summary statistics by this algorithm will still appear in the associated listings. Also, all applicable valid assessments, irrespective of proximity to the target study day, will be used when categorizing values across visits, such as 'maximum grade' or 'at any time', and for any algorithm that has specific rules for which observation to use (e.g. snapshot algorithm, LOCF or CVF identification).

# 15.4. Appendix 4: Study Phases and Treatment State

# 15.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to the Treatment Start Date defined in Section 15.6.1.

AEs will be assigned to study phases as defined in Table 13. For example, adverse events on/after start of maintenance phase IP and prior to start of Extension phase IP/LTFU ART will be assigned to the Maintenance Phase.

Laboratory data (efficacy, safety, PK and virology), HIV associated Conditions, health outcomes assessments, vital signs, and ECGs will be assigned to study phases as defined as in Table 14. For example, assessments/events occurring after start of maintenance phase IP and up to and including start of extension phase IP/LTFU ART will be assigned to the Maintenance Phase.

Assessments/events are assigned to study phases sequentially, starting from the top of each table. No study phases will be assigned to medications.

Table 13 Assignment of Study Phases for AEs

| Study Phase | Definition |
|---|---|
| Screening | Date < Maintenance Treatment Start Date |
| Maintenance | For participants continuing into Extension Phase: |
| | Maintenance Treatment Start Date ≤ Date < Date of Nominal Week 100 Visit |
| | For participants <u>not</u> continuing into Extension Phase <sup>[a]</sup> : |
| | Maintenance Treatment Start Date ≤ Date < LTFU ART Start Date |
| | For AEs leading to withdrawal and started on the same date as LTFU ART |
| | Start Date, Maintenance Phase, instead of Long-term Follow-up phase, will |
| | be assigned. |
| Extension | Participants continuing into Extension Phase <sup>[a]</sup> : |
| | Date of Nominal Week 100 Visit ≤ Date < LTFU ART Start Date |
| | For AEs leading to withdrawal and started on the same date as LTFU ART |
| | Start Date, Extension Phase, instead of Long-term Follow-up phase, will be |
| | assigned. |

### NOTES:

- Date = AE Start date
- [a] If participants have missing LFTU ART start date, only the lower bound will be considered in the derivation.

Table 14 Assignment of Study Phases for Lab Assessments (including PK and Virology), ECG, Protocol Deviations, Vital Sign, Health Outcomes, HIV Associated Conditions

| Study Phase | Definition |
|---|---|
| Screening | Date ≤ Maintenance Treatment Start Date Note: 2-hour post-dose ECG taken on the Maintenance Treatment Start Date will be excluded. |
| Maintenance | For participants continuing into Extension Phase: Maintenance Treatment Start Date < Date ≤Date of Nominal Week 100 Visit Note: 2-hour post-dose ECG taken on the Maintenance Treatment Start Date will be included. For participants not continuing into Extension Phase <sup>[a]</sup> : Maintenance Treatment Start Date < Date ≤ LTFU ART Start Date Note: 2-hour post-dose ECG taken on the Maintenance Treatment Start Date will be included. |
| Extension | Participants continuing into Extension Phase <sup>[a]</sup> : Date of Nominal Week 100 Visit < Date ≤ LTFU ART Start Date |

- Date = start or assessment date
- [a] If participants have missing LFTU ART start date (i.e. the participants have not started ART in LFTU yet), only the lower bound of the window will be considered in the derivation.

Table 15 Assignment to Long-term Follow-up Phase

| Study Phase | Definition |
|---|---|
| Long-term<br>Follow-up | Date > max (Last IM Injection Date, Last Oral Bridging End Date) |

- Date = Assessment/Start Date
- For AEs leading to withdrawal and started on the same date as LTFU ART Start Date, maintenance phase or extension phase depending on participant's continuation status to extension phase, instead of long-term follow-up phase, will be assigned. Refer to Table 13 for details.

Only participants who received at least one CAB and/or RPV injection will enter the long-term follow-up. Note that the long-term follow-up phase and maintenance/extension phases are not necessarily mutually exclusive and are to be defined with separate phase variables in the datasets. For example, an Q4W IM participant who has Week 44 injection and withdrawal at Week 48 without receiving Week 48 injection, the "Week 48 withdrawal visit" belongs to both the maintenance phase and long-term follow-up phase.

### 15.4.2. Treatment State

Within each treatment study phase (i.e. Maintenance and Extension—based on assignment of study phase described in Section 15.4.1), only those assessments which occur within the ranges shown in Table 16 will be considered 'on-treatment' for the given phase. No treatment states will be assigned to medications.

Table 16 Treatment State within Study Phases<sup>b</sup>

| Study Phase <sup>a</sup> | Treatment State | Date Range |
|---|---|---|
| Screening | Pre-treatment | All assessments/events within the phase |
| Maintenance | On-treatment | Q8W arm: |
| | | Date ≤ max (Date of Last Injection + 63, Date of Last Dose |
| | | of Oral CAB+RPV + 1) |
| | | Q4W arm: |
| | | Date ≤ max (Date of Last Injection + 35, Date of Last Dose |
| | | of Oral CAB+RPV + 1) |
| | Post-treatment | Q8W arm: |
| | | Date > max (Date of Last Injection + 63, Date of Last Dose |
| | | of Oral CAB+RPV + 1) |
| | | Q4W arm: |
| | | Date > max (Date of Last Injection + 35, Date of Last Dose |
| | | of Oral CAB+RPV + 1) |
| Extension | On-treatment | Q8W arm: |
| | | Date ≤ max (Date of Last Injection + 63, Date of Last Dose |
| | | of Oral CAB+RPV + 1) |
| | | 0.000 |
| | | Q4W arm: |
| | | Date ≤ max (Date of Last Injection + 35, Date of Last Dose |
| | D 11 1 | of Oral CAB+RPV + 1) |
| | Post-treatment | Q8W arm: |
| | | Date > max (Date of Last Injection + 63, Date of Last Dose |
| | | of Oral CAB+RPV + 1) |
| | | Q4W arm: |
| | | Date > max (Date of Last Injection + 35, Date of Last Dose |
| | | of Oral CAB+RPV + 1) |
| Long-term Follow- | On-treatment | Q8W arm: |
| up | | Date ≤ min (LTFU ART start date, max (Date of Last |
| • | | Injection + 63, Date of Last Dose of Oral CAB+RPV + 1)) |
| | | , |
| | | Q4W arm: |
| | | Date ≤ min (LTFU ART start date, max (Date of Last |
| | | Injection + 35, Date of Last Dose of Oral CAB+RPV + 1)) |
| | Post-treatment | Q8W arm: |
| | | Date > min (LTFU ART start date, max (Date of Last |
| | | Injection + 63, Date of Last Dose of Oral CAB+RPV + 1)) |
| | | 04144 |
| | | Q4W: |
| | | Date > min (LTFU ART start date, max (Date of Last |
| | | Injection + 35, Date of Last Dose of Oral CAB+RPV + 1)) |

### NOTE:

- Date = Assessment/Start Date.
- a. Treatment State is determined after data has been assigned to the study phases as defined in Section 15.4.1.
- b. Last injection and/or last dose of oral CAB+RPV are only applied to participants who permanently discontinued the study treatment. The assessments for participants who did not permanently discontinue the study treatment will be considered 'On-treatment'. For participants continuing into extension phase, all data assigned to maintenance phase per Section 15.4.1 will be considered 'On-treatment'.

### 15.4.2.1. Treatment States for AE Data

For adverse events, partial AE start date will use imputation as described in Section 15.7.2.1. In the case of a completely missing start date, the event will be considered to have started On-treatment in the Maintenance phase unless an end date for the AE is provided which is before start of study treatment at Maintenance phase; in such a case the AE is assigned as Pre-treatment.

Additional variables will be derived as shown in Table 17.

Table 17 Days since First Dose of Each Study Phase, Days since Phase Start, AE Duration and Relation to Study Treatment

| | Definition |
|---|---|
| Days since<br>First Dose<br>(Days) <sup>a</sup> | AE Start Date – Maintenance Treatment Start Date + 1 |
| Days since<br>Last Dose<br>(Days) <sup>a</sup> | AE Start Date – Date of Last Dose of Study Treatment prior to/on the Start Date of AE + 1 |
| Days since<br>Phase Start | For AEs in Maintenance Phase: AE Start Date - Maintenance Treatment Start Date + 1 For AEs in Extension Phase: AE Start Date - Date of Nominal Week 100 Visit + 1 For AEs in Long-term Follow-up Phase: AE Start Date - Date of Last Dose of Study Treatment <sup>b</sup> |
| Duration<br>(Days) | AE Resolution Date – AE Start Date + 1 |
| Drug-related | If relationship is marked 'YES' on Inform/eCRF or value is missing. |

### NOTES

- a. Days since First/Last Dose will only be derived for AEs assigned to maintenance phase, extension phase and long-term follow-up phase.
- b. Date of Last Dose of Study Treatment = max (Last IM Injection Date, Last Oral Bridging End Date), only applicable to participants who permanently discontinued study treatment.

# 15.4.3. Study Period

Certain displays will be produced for data collected during the oral lead-in. The study period variable is defined in Table 18 and Table 19. Study period is assigned after the study phase is assigned (screening, maintenance, extension, or long-term follow-up) based on the Tables in Section 15.4.1.

Table 18 Assignment of Study Period for AE Data

| Study Period | Date range |
|---|---|
| Oral Lead-in | For participants receiving at least one Injection: |
| | Maintenance Treatment Start Date ≤ Date < Date of First IM Injection |
| | For participants withdrawing prior to first Injection: |
| | Date ≥ Maintenance Treatment Start Date |
| | Note that the oral lead-in period is only applicable to the participants who received at least one dose of study treatment during the oral lead-in period in the study. Oral lead-in period is within the maintenance phase. |

### NOTES:

• Date = AE Start date.

 Table 19
 Assignment of Study Period for Lab Assessments:

| Period | Date range |
|---|---|
| Oral Lead-in | For participants receiving at least one Injection: Maintenance Treatment Start Date < Date ≤ Date of First IM Injection |
| | For participants withdrawing prior to first Injection: Date > Maintenance Treatment Start Date |
| | Note that the oral lead-in period is only applicable to the participants who received at least one dose of study treatment during the oral lead-in period in the study. Oral lead-in period is within the maintenance phase. |

# NOTES:

• Date = Date of assessment.

# 15.5. Appendix 5: Data Display Standards & Handling Conventions

# 15.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : us1salx00259 |
| HARP Compound | : \ARPROD\GSK1265744\mid207966 |

### **Analysis Datasets**

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.0).
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

### **Generation of RTF Files**

RTF files will be generated for every reporting effort described in the RAP.

# 15.5.2. Reporting Standards

### General

 The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics

### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Actual time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - If space allows, planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

- When data falls within both maintenance / extension and long-term follow-up phases, it will be presented in maintenance / extension phase, unless otherwise specified.
- Unless otherwise specified, when data falls within both screening and baseline visits per analysis visit windows, it will be presented at baseline visit.

### **Unscheduled Visits**

- Unscheduled visits will be assigned to a study visit using the all-inclusive windows defined in Section 15.3.
- However, data summaries will only report visits that are planned assessment time points for each parameter (according to the Time and Events table).
- Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well any algorithms that make use of additional data (e.g., Snapshot).

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 | |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 15.5.3. Reporting Standards for Pharmacokinetic

| Reporting of Pharmacokinetic Concentration Data | |
|---|---|
| Descriptive<br>Summary Statistics,<br>Graphical Displays<br>and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1 Assign the low limit of quantification (CAB 0.025 ug/mL, RPV 1 ng/mL) to NQ values. |
| Reporting of Pharmacokinetic Parameters | |
| Descriptive Summary Statistics (Loge Transformed) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of log <sub>e</sub> transformed data and between participant coefficient of variation (CV <sub>b</sub> (%)) will be reported. |
| | $ CV_b(\%) = \sqrt{\exp(SD^2) - 1} \times 100 $ (SD = SD of log <sub>e</sub> transformed data) |

# 15.6. Appendix 6: Derived and Transformed Data

### 15.6.1. General

# **Multiple Measurements at One Time Point**

• If after window assignment there are multiple valid assessments of a parameter within the same window, refer to Section 15.3.6 for determination of the value to be used for summary statistics of observed values. Assessments not chosen for use in summary statistics will still appear in the associated listings. Assessments not chosen for use in summary statistics by this algorithm will still appear in the associated listings. Also, all applicable valid assessments, irrespective of proximity to the target study day, will be used when categorizing values across visits, such as 'maximum grade' or 'at any time', and for any algorithm that has specific rules for which observation to use (e.g. snapshot algorithm, LOCF or CVF identification).

### **Treatment Start Date**

Treatment start date is defined as follows:

Maintenance Phase

 Date of first ATLAS-2M dose of CAB+RPV (oral or injection) entered onto the IP exposure eCRF form.

### **Extension Phase**

- For participants not continuing into extension phase, treatment start date is missing.
- For participants continuing into extension phase, treatment start date is the date of first dose of CAB+ RPV (oral or injection) at or after nominal Week 100 visit.

### Long-term Follow-up Phase

- If a participant is still on study treatment, or permanently discontinued the study treatment and did not have any previous injections, treatment start date is missing.
- If a participant permanently discontinued the study treatment and had at least one injection, treatment start date is the date of first ART treatment after the last dose of study treatment (oral or injection).

# Study Day

The Study Day of an event (e.g., lab assessment, vital sign, ECG, start date of AE or HIV associated condition) will be derived as the number of days between the date of the event and the start date of study treatment during the Maintenance Phase as follows:

if date of event  $\geq$  start date of study treatment, then

Study Day=date of event - start date of Maintenance Phase treatment +1

if date of event < start date of study treatment, then

Study Day=date of event - start date of Maintenance Phase treatment

Note that the start date of study treatment during maintenance phase is considered to be on Study Day 1 and the day before this is Study Day -1; i.e., there is no Study Day 0.

### **Extension Phase Study Day**

The Study Day of an event (e.g., lab assessment, vital sign, ECG, start date of AE or HIV associated condition) will be derived as the number of days between the date of the event and the date of nominal Week 100 visit as follows:

if date of event ≥ date of nominal Week 100 visit, then

Study Day=date of event - date of nominal Week 100 visit + 1

if date of event < date of nominal Week 100 visit, then

Study Day = date of event - date of nominal Week 100 visit

Note that the date of nominal Week 100 visit is considered to be on Extension Phase Study Day 1 and the day before this is Extension Phase Study Day -1; i.e., there is no Extension Phase Study Day 0.

# Long-term Follow-up Study Day

The Long-Term Follow Up (LTFU) Study Day of an event (e.g., lab assessment, start date of AE or HIV associated condition) will be derived as the number of days between the date of the event and the end of IP treatment [i.e. max(Last IM Injection Date, Last Oral Bridging End Date)] as follows:

If the date of event falls in Long-term Follow up phase, then

LTFU Study Day = Date of Event - End Date of IP

### **Change from Baseline**

- Post-Dose Visit Value Baseline
  - Unless otherwise specified, the baseline definitions specified in Section 5.2 will be used for derivations for endpoints / parameters.

# 15.6.2. Study Population

### **Demographics and Baseline Characteristics**

### Age

- Age, in whole years, will be calculated with respect to the participant's Screening visit.
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any participant with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Completely missing dates of birth will remain as missing, with no imputation applied. Consequently, the age of the participant will not be calculated and will remain missing.

### **Body Mass Index (BMI)**

Calculated as Weight (kg) / Height (m)<sup>2</sup>

### **Hepatitis Status**

- Hepatitis C status will be determined using antibody and/or hepatitis C virus (HCV) RNA assessments performed during screening or during the conduct of the study.
- If both antibody and virus RNA assessments are available, then the latter will take precedence
  and positive/negative status will be based on whether HCV RNA is detectable (i.e., ≥ limit of
  quantification) or not.
- A participant will be considered positive for hepatitis B virus (HBV) if they have a positive

# **Demographics and Baseline Characteristics**

surface antigen or detectable HBV DNA result. "HBV DNA DETECTED" in the lab comment takes precedence over HBV DNA test result for positive hepatitis B status, for example, if a participant has HBV test result below level of detection, however, the lab comment shows that HBV DNA detected, this participant will be considered positive for hepatitis B. If HBV DNA result is available, it will be used to qualify hepatitis B status as positive or negative (positive if ≥ limit of quantification); otherwise Hepatitis B status will be determined using the surface antigen result.

 Hepatitis status at entry will be based on the assessments prior to/on the start of the study treatment.

# Framingham Risk Equation

• The predicted probability,  $\hat{p}$ , of having a cardiovascular disease (CVD) within the next 10-years according to the Framingham formula [D'Agostino et al. 2008] is

### For females:

$$\widehat{p}_F = 1 - S_0(t)^{\exp\left\{2.32888 \times \log(age) + 1.20904 \times \log(TC) - 0.70833 \times \log(HDL) + 2.76157 \times \log(SBP_u) + \frac{1}{2.82263 \times \log(SBP_t) + 0.52873 \times I_s + 0.69154 \times I_d - 26.1981}\right\}}$$

For males:

$$\hat{p}_{M} = 1 - S_{0}(t)^{\exp\left\{3.06117 \times \log(ag\cdot e) + 1.12870 \times \log(TC) - 0.93263 \times \log(HDL) + 1.93908 \times \log(SBP_{u}) + 1.99881 \times \log(SBP_{t}) + 0.65451 \times I_{S} + 0.57367 \times I_{d} - 23.9802 \right\}}$$

where

$$S_0(t) = \begin{cases} 0.95012, \text{ females} \\ 0.88936, males \end{cases}$$

$$I_s = \begin{cases} 1, \text{ current smoker} \\ 0, & \text{otherwise} \end{cases}$$

$$I_d = \begin{cases} 1, & \text{diabetic} \\ 0, & \text{otherwise} \end{cases}$$

TC = total serum cholesterol (mg/dL),

HDL = serum HDL cholesterol (mg/dL).

SBPu = systolic blood pressure (mmHg) if participant is not treated for high blood pressure (note that if a participant is treated for high blood pressure then log(SBPu) = 0)
SBPt = systolic blood pressure (mmHg) if participant is treated for high blood pressure (note that if a participant is not treated for high blood pressure then log(SBPt) = 0)

- A participant will be considered as treated for high blood pressure if during screening it has specified that is suffering from hypertension.
- A participant is classified as diabetic if current or past is indicated in the medical conditions eCRF for Type 1 or Type 2 diabetes mellitus, or if baseline fasting glucose ≥7.00 mmol/L (126 mg/dL).
- Smoking status is collected in the eCRF at Day 1. A current smoker is defined as currently smoking/using tobacco or has smoked/used tobacco within the previous 6 months; a former smoker is defined as previously smoked/used tobacco products and has not smoked/used

# **Demographics and Baseline Characteristics**

tobacco products within the previous 6 months.

This calculation will not be performed for participants who have indicated current or past
myocardial infarction conditions on the eCRF. These participants will not be included in
summary statistics of risk, but they will be counted in the highest category of risk in the
summary by category.

# **Prior Exposure to CAB+RPV**

- For participants transitioning from ATLAS study and having prior exposure to CAB+RPV in ATLAS study: Duration of Prior Exposure to CAB+RPV = Randomization Date – Prior Oral CAB Start Date in ATLAS Study + 1.
- For participants transitioning from ATLAS study and not having prior exposure to CAB+RPV in ATLAS study, or for participants randomized from current SOC, Duration of Prior Exposure to CAB+RPV = 0.
- Duration of Prior Exposure to CAB+RPV will be categorized to 0 weeks, 1-24 weeks and >24 weeks.

# **Lipid-modifying Agents**

- The following ATC codes correspond to lipid-modifying agents:
  - o ATC Level 2: C10
  - o ATC Level 3: C10A, C10B (if Level 2 is not available)
  - ATC Level 4: C10AA, C10AB, C10AC, C10AD, C10AX, C10BA, C10BX (if level 2, 3 are not available)
- Participants are considered to have used a lipid-modifying agent at baseline if they are taking the medication at the time of their baseline lipid testing date.
- Participants are also considered to have used a lipid-modifying agent at baseline if they stopped their lipid modifying medication within 12 weeks prior to their baseline lipid testing date.

# 15.6.3. **Efficacy**

### **Snapshot**

- The Snapshot algorithm is intended to be primarily a virologic assessment of the endpoint, and as such follows a "virology first" hierarchy.
- 'HIV-1 RNA < 50 c/mL' or 'HIV-1 RNA ≥ 50 c/mL' within an analysis window (see Table 10) is typically determined by the last available HIV-1 RNA measurement in that window while the participant is On-treatment in the Maintenance Phase (as assigned based on Section 15.4).
- When no HIV-1 RNA data is available within a window, a participant cannot be assigned to the category of 'HIV-1 RNA < 50 c/mL'. Depending on the reason for lack of data, the participant will be classified as 'HIV-1 RNA < 50 c/mL' or reported as 'No Virologic Data at Week X'; in the latter case, the algorithm further classifies the nature of the missing data. Typically, a participant withdrawn (i) due to AE or, (ii) for another reason yet was suppressed at the time, will be counted as 'No Virologic Data at Week X'. Should a participant withdraw for reasons other than AE and was not suppressed at the time, they will be categorized as 'HIV-1 RNA ≥ 50 c/mL'.</p>
- Full details of the algorithm, including the handling of special cases, are included in Section 15.9

### Plasma HIV-1 RNA

- For summaries and analyses which use HIV-1 RNA level as a continuous measure, the logarithm to base 10 of the value will be used.
- HIV-1 RNA results may be provided as censored values, such as <40 or >9,999,999 c/mL. For
  the purposes of summary statistics, such values will be replaced by the next value beyond the
  limit of detection, e.g., 39 or 10,000,000 c/mL, respectively, for the given examples. Data
  listings will show the censored values as provided.

# Target Detected / Target Not Detected / Super Low Viral Load Testing

- When a measurement of plasma HIV-1 RNA is below the limit of quantification (i.e. 40 c/mL) and is qualitatively observable that will be denoted as a "Target Detected" measure, while HIV-1 RNA below the limit of quantification that is not qualitatively observable that will be denoted as "Target Not Detected". Any measurements <40 c/mL characterised as "Target Not Detected" or "Target Detected" will be captured in the database.</li>
- Super low viral load will also be tested by BioMNTR lab for viral loads below the limit of quantification at some visits (e.g. Week 48).

# **Confirmed Virologic Failure (CVF)**

- The definition of CVF is provided in the Protocol, Section 5.5.4 Definition of Confirmed Virologic Failure.
- In case there are multiple plasma HIV-1 RNA results on the same day, the worst result (i.e. the largest value) will be used in determination of CVF.

# Treatment (TRDF) and Efficacy Related (ERDF) Discontinuation = Failure

- The analysis of time to confirmed virologic failure (CVF) or discontinuation due to treatment related reasons (i.e., drug-related AE, intolerability of injections, protocol defined safety stopping criteria, or lack of efficacy) will censor participants who have not met CVF criteria and are ongoing in the study, or who have discontinued for reasons other than those related to treatment. This will be the Treatment Related Discontinuation = Failure (TRDF) data.
- Participants who have not met CVF criteria and are ongoing in the study, or who have discontinued for reasons other than lack of efficacy, will be censored in the analysis of the Efficacy Related Discontinuation = Failure (ERDF) data.
- Proportion of Participants without virologic (ERDF) or tolerability (TRDF) failure will be
  estimated using the Kaplan-Meier nonparametric method based on the time to ERDF or TRDF.
  The estimated proportion at time point of interest will be presented by treatment group, along
  with estimated difference in proportions between treatment groups and its associated two-sided
  95% CI. The estimate of the standard error used to derive confidence intervals will be based on
  Greenwood's formula [Kalbfleisch.1980].
- See Appendix 10: Variables Defined for Time to Event Analysis for additional details.

# Summary for Participants per Viral Load Category by Visit

- Summary will be based on observed available data, with no imputation for missing values. The
  proportion of participants in each viral load category will be calculated using the denominator
  and numerator specified below:
  - Denominator: Number of participants with on-treatment viral load within the snapshot visit window.
  - Numerator: Number of participants with plasma HIV-1 RNA in the specified category based on the last on-treatment viral load assessment collected within the snapshot visit window.

# **HIV-1 Disease progression Stage**

- Categories:
  - CDC Stage I at Baseline to CDC Stage III;
  - CDC Stage II at Baseline to CDC Stage III;
  - CDC Stage III at Baseline to new CDC Stage III event;
  - o CDC Stage I, II, III at Baseline to Death.

Please refer to Protocol (Appendix 4: CDC Classification for HIV-1 Infection) for defining Stage.

- For the purpose of analysis, the CDC at Baseline and at post-baseline during Maintenance Phase will be derived as below:
  - At Baseline, the 'Baseline CDC stage' for each participant was assessed by investigator and recorded in the eCRF. However, for the analysis, Baseline CDC stage will be rederived based Baseline CD4+ values as well as whether any HIV-associated/AIDS-defining conditions present at baseline per the Criteria's thresholds (Appendix 4 in Protocol).
  - To analyse disease progression, the most advanced post-baseline CDC stage within the period of interest (e.g. Maintenance Phase) will be derived based on the occurrences of new AIDs-defining conditions (please refer to Appendix 4 in Protocol for the list of AIDsdefining Conditions) as well as the nadir value of post-baseline CD4+.
    - ➤ For example, if a participant with CDC 'Stage I' at Baseline had the lowest Maintenance Phase CD4+ =120 cell/mm³ without new AIDs-defining conditions, then HIV disease progression for this participant during the Maintenance Phase would be considered as 'CDC stage I at Baseline to CDC stage III'.
    - ➤ If a participant with CDC 'Stage II' at Baseline had the lowest Maintenance Phase CD4+ =220 cell/mm3 AND had at least one new AIDs-defining condition, then HIV disease progression for this participant during the Maintenance Phase would be considered as 'CDC stage II at Baseline to CDC stage III'.

### **Delay in IP Injection**

- For participants on the Q4W arm, IM dosing is expected to occur every 4 weeks from Week 4B onwards for those transitioning from SOC (i.e. those requiring oral lead-in) and from Day 1 onwards for those transitioning from CAB+RPV Q4W in ATLAS (i.e. those not requiring oral lead-in). The Delay in IP injection (days) will be calculated as:
  - Delay in IP Injection (days) = Injection date date of preceding injection 28 days
- For participants on the Q8W arm, IM dosing is expected to occur at Week 4B and then every 8
  weeks from Week 8 onwards for those transitioning from SOC (i.e. those requiring oral lead-in)
  and every 8 weeks from Day 1 for those transitioning from CAB+RPV Q4W (i.e. those not
  requiring oral lead-in) in ATLAS.
  - For participants transitioning from SOC on the Q8W arm, if the preceding injection occurs at Week 4B, the Delay in IP injection (days) will be calculated as:
     Delay in IP Injection (days) = Date of Week 8 injection - date of Week 4B injection - 28 days
  - For participants transitioning from SOC on the Q8W arm, if the preceding injection occurs at a visit later than Week 4B, the Delay in IP injection (days) will be calculated as:
     Delay in IP Injection (days) = Injection date - date of preceding injection - 56 days
  - o For participants transitioning from CAB+RPV Q4W in ATLAS on the Q8W arm, the Delay in

IP injection (days) will be calculated as: Delay in IP Injection (days) = Injection date - date of preceding injection - 56 days

- Delay in IP injection will be grouped into: ≤1, 2-3, 4-7, >7 days.
- The proportion of participants with HIV-1 RNA ≥50 c/mL at Week 48 (Snapshot) will be summarized by last delay in IP Injection. The last delay in IP injection will be the delay in IP injection at Week 48, or the delay in last IP injection prior to Week 48 if a participant did not receive Week 48 injection (i.e. missing visit or withdrawal).

# 15.6.4. Safety

# **Adverse Events**

# **DAIDS Grading**

 Clinical adverse events will be graded based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.1, March 2017, as specified in the protocol Appendix 11.2.

# Potential QTc Interval Prolonging Events of Interest

Potential QTc Interval Prolonging Events of Interest will be identified based on Standardised MedDRA Query (SMQ) for Torsade de pointes/QT prolongation, broad (MedDRA). The terms per this reference are listed below.

| AE preferred term |
|----------------------------------------------|
| Electrocardiogram QT interval abnormal |
| Electrocardiogram QT prolonged |
| Long QT syndrome |
| Long QT syndrome congenital |
| Torsade de pointes |
| Ventricular tachycardia |
| Cardiac arrest |
| Cardiac death |
| Cardiac fibrillation |
| Cardio-respiratory arrest |
| Electrocardiogram repolarisation abnormality |
| Electrocardiogram U wave inversion |
| Electrocardiogram U wave present |
| Electrocardiogram U-wave abnormality |
| Loss of consciousness |
| Sudden cardiac death |
| Sudden death |
| Syncope |
| Ventricular arrhythmia |
| Ventricular fibrillation |

| Adverse Events |
|-----------------------------|
| Ventricular flutter |
| Ventricular tachyarrhythmia |

# **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value. If a character value starting with "<=x", then the numeric value will be x.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' or '>=x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

# Estimate of Glomerular Filtration Rate (GFR) (Levey AI et al, 2012)

Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation [Levey et al, 2012] will be used by the central laboratory to provide an estimate of GFR, in mL/min per 1.73 m², as follows:

$$\begin{aligned} \text{GFR} &= 141 \times \text{min} \left( \frac{\text{CRT}_{\text{mg/dL}}}{\kappa}, 1 \right)^{\alpha} \times \text{max} \left( \frac{\text{CRT}_{\text{mg/dL}}}{\kappa}, 1 \right)^{-1.209} \times 0.993^{\text{Age}} \times \\ & [1.018 \text{ if Female}] \times [1.159 \text{ if Black}] \end{aligned}$$

where age (in years) is at time of assessment,  $\kappa$  = 0.7 if female or 0.9 if male,  $\alpha$  = -0.329 if female and -0.411 if male, min() indicates the minimum of CRT/ $\kappa$  or 1, max() indicates the maximum of CRT/ $\kappa$  or 1, and CRTmg/dL is serum creatinine concentration in mg/dL. The serum creatinine concentration in mg/dL is obtained from GSK standard units of  $\mu$ mol/L as CRTmg/dL =0.0113x CRT $\mu$ mol/L.

• The CKD-EPI GFR will also be calculated using Cystatin C, as follows

133 X min(Scys/0.8, 1) -0.499 X max (Scys/0.8, 1)-1.328 X 0.996 Age X[0.932 if female]

Where Scys is serum cystatin C mg/Liter, min indicates the minimum of Scr/0.8 or 1, and max indicates the maximum of Scys/0.8 or 1.

**Lab Toxicities – DAIDS Grading based on** Version 2.1, March 2017, as specified in the protocol of Appendix 11.2.

- Toxicities will be based on the Division of AIDS (DAIDS) grading system, Version 2.1, March 2.17, as specified in the protocol of Appendix 11.2
- Toxicity grades provided by the central laboratory do not distinguish between abnormally high or low criteria, when both are relevant for a parameter.
- When summarising toxicity grades for such parameters, they will be categorised as to whether they are above or below the midpoint of normal range.

| Laboratory Parameters | | | |
|---|---|---|---|
| | Parameter | Below Midpoint for | Above Midpoint for |
| | | those ≥Grade 1 | those ≥Grade 1 |
| | Fasted glucose | Hypoglycemia | Hyperglycemia |
| | Sodium | Hyponatremia | Hypernatremia |
| | Potassium | Hypokalemia | Hyperkalemia |

# National Cholesterol Education Program (NCEP) Lipid Categories

• In addition to DAIDS toxicity grades (see protocol), lipid values will be categorized according to the 2001 NCEP Adult Lipid Guidelines [Grundy, 2001]

| Parameter | Value Range (mmol/L) | Value Range (mg/dL) | Category |
|---|---|---|---|
| Triglycerides | <1.70 | <150 | Normal |
| | 1.70 to <2.26 | 150 to <200 | Borderline High |
| | 2.26 to <5.65 | 200 to <500 | High |
| | ≥5.65 | ≥500 | Very High |
| Total Cholesterol | <5.18 | <200 | Desirable |
| | 5.18 to <6.21 | 200 to <240 | Borderline High |
| | ≥6.21 | ≥240 | High |
| HDL Cholesterol | <1.04 | <40 | Low |
| | 1.04 to <1.56 | 40 to <60 | Normal |
| | ≥1.56 | ≥60 | High |
| LDL Cholesterol | <2.59 | <100 | Optimal |
| | 2.59 to <3.37 | 100 to <130 | Near/Above Optimal |
| | 3.37 to <4.14 | 130 to <160 | Borderline High |
| | 4.14 to <4.92 | 160 to <190 | High |
| | ≥4.92 | ≥190 | Very High |

# Percentage change for lipids

The percentage change from baseline is calculated as:

% change from baseline =  $\frac{\text{value at Week 48 or 96-baseline value}}{\text{baseline value}} \times 100\%$ 

### Total Cholesterol / HDL Cholesterol Ratio

When both total cholesterol and HDL cholesterol results are available from the same date for a
participant, then the ratio will be calculated by dividing the total cholesterol result by the HDL
cholesterol result. The ratio can be classified as follows:

| Parameter | Value Range |
|-------------------|--------------|
| Total Cholesterol | < 3.5 |
| / HDL Ratio | 3.5 to < 4.4 |
| | 4.4 to < 5 |
| | ≥ 5 |

# **Other Safety Endpoints**

# Corrected QT (QTc)

When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fridericia's

# **Other Safety Endpoints**

(QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.

If RR interval (in msec) is provided then missing QTcB and/or QTcF will be derived as

$$QTcB = \frac{QT}{\sqrt{RR/1000}} \qquad \qquad QTcF = \frac{QT}{\sqrt[3]{RR/1000}}$$

where uncorrected QT interval is also measured in msec.

If RR interval is not provided directly and one of QTcB or QTcF has been entered, then RR interval can be obtained from the above formulas and used to calculate the other correction method value; i.e.,

$$QTcB = \sqrt{\frac{QTcF^{3}}{QT}} \qquad \qquad QTcF = \sqrt[3]{QT \cdot QTcB^{2}}$$

# **Extent of Exposure**

- Exposure to CAB+RPV (oral lead-in or oral bridging) and CAB LA+RPV LA will be calculated from the IP eCRF pages.
- For Maintenance Phase:
  - Exposure to oral CAB+RPV (oral lead-in) = IP (oral lead-in) stop date IP (oral lead-in) start date +1
  - Exposure to CAB LA + RPV LA = Number of IP injections received during maintenance phase (up to but not including injections administered at Week 100)
  - Overall exposure to IP:

For participants on Q4W arm: min [Date of Latest Maintenance Phase Visit up to and including Week 100, max (Date of Last Injection + 35, Date of Last Dose of Oral CAB+RPV)] – min (Start Date for Oral lead-in CAB+RPV, Date of First Study Injection) + 1

For participants on Q8W arm: min [Date of Latest Maintenance Phase Visit up to and including Week 100, max (Date of Last Injection + 63, Date of Last Dose of Oral CAB+RPV)] – min (Start Date for Oral lead-in CAB+RPV, Date of First Study Injection) + 1

- For Maintenance + Extension Phase
  - Exposure to CAB LA + RPV LA = Number of IP injections received during Maintenance Phase + Extension Phase
  - Overall Exposure to IP:

For participants on Q4W arm: min [Date of Latest Visit, max (Date of Last Injection + 35, Date of Last Dose of Oral CAB+RPV)] – min (Start Date for Oral lead-in CAB+RPV, Date of First Study Injection) + 1

For participants on Q8W arm: min [Date of Latest Visit, max (Date of Last Injection + 63, Date of Last Dose of Oral CAB+RPV)] – min (Start Date for Oral lead-in CAB+RPV, Date of First Study Injection) + 1

Last Injection and/or Last Dose of Oral CAB+RPV are only applicable to those who
permanently discontinued study treatment.

### **Other Safety Endpoints**

- Duration of dosing in participant years will be calculated as the sum of participant duration of dosing in days (across all participants)/365.25
- Participants who were randomized but did not report a IP start date will be categorised as having zero days of exposure.

# Adherence to CAB/RPV Injection Schedule

Timeliness of Injections relative to Date of Projected Dosing Visits are assessed by using "actual injection visit date - projected visit date from first injection". The injections of interest in adherence analysis are those after first injection. For participants requiring the oral CAB+RPV lead-in, the first injection is planned to be taken at Week 4B. For participants not requiring the oral CAB+RPV lead-in, the first injection is planned to be taken at Baseline/Day 1. Each injection visit is counted only once. Individual CAB and RPV injections administered at the same visit are not counted twice. "Extra" unscheduled injections are excluded from all derivations. For example, if during a scheduled visit a participant receives 1 ml of injection instead of 2 ml due to a dosing error, but this participant returns one week later for the remaining 1 ml injection, then the additional visit is excluded. If a participant receives an extra injection at an unscheduled visit by mistake, this visit will also be excluded.

The categories of Timeliness of Injections relative to Date of Projected Dosing Visits for summary are listed below:

```
< -14 days
-14 to -8 days
-7 to -4 days
-3 to -2 days -1
0 day
1
2 to 3 days
4 to 7 days
8 to 14 days
>14 days
Missed Injection without Oral Bridging
Missed Injection with Oral Bridging
```

### Columbia Suicide Severity Rating Scale (C-SSRS)

Missing data will not have any imputation performed (Nilsson et al, 2013).

### 15.6.5. Pharmacokinetic

This document is intended for planning analysis of PK concentration data only. Population pharmacokinetics and identification of important determinants of variability will be described in a separate document.

### **Pharmacokinetic Analyses**

# Plasma CAB and RPV Concentration-time Data

Plasma samples for determination of CAB and RPV concentration will be collected throughout the Maintenance Phase and at the withdrawal visit. Additional samples will be collected for storage during the Long-Term Follow-Up Phase.

### **Evaluable Concentration**

PK concentration will be summarized in two ways: 'all data' without regard to timing relative to scheduled time and 'evaluable data'.

The 'evaluable data' are from the samples that met sample collection window criteria. Sampling windows are set relative to the previous dose as follows:

- 20-28 hrs after last oral dose taken and properly administered last 3 oral doses for pre-dose sample at Week 4B for participants requiring oral lead-in
- ± 4 days for pre-dose sample at visits other than Week 4B, and for pre-dose samples at Week 4B for participants not requiring oral lead-in (e.g. participants transitioning from ATLAS Q4W and remain on Q4W arm in this study)
- 3-10 days post last injection for 1-week post injection visits;
- Samples impacted by dosing errors (wrong dose) or oral bridging will also be excluded

| Timepoint | Evaluable<br>Window | For Programming: |
|---|---|---|
| Pre-dose: WK4B for participants requiring oral lead-in | 20-28 hrs after last oral dose taken and the last 3 oral doses administered properly | 20 hrs ≤ Time since Last Oral Dose ≤ 28 hrs and the last 3 oral doses administered on the three consecutive days prior to WK4B. |
| Pre-dose at other visits, Pre-dose WK4B for participants not requiring oral lead-in | ± 4 days | For Q4W arm, Day 1 pre-dose, and Week 8 for those transitioning from SOC (i.e. requiring oral lead-in) on Q8W arm: 24 days ≤ Days Since Last Injection ≤ 32 days For visits other than above on Q8W arm: 52 days ≤ Days Since Last Injection ≤ 60 days |
| 1-WK-Post: | 3-10 days post last injection | 3 days ≤ Days Since Last Injection ≤ 10 days |

Relative Time is calculated relative to the date and time of last previous dose. For example, if the time of the last previous dose (e.g. oral lead-in/oral-bridging) is missing, then the relative time for

# **Pharmacokinetic Analyses**

pre-dose PK sample will be set to missing and the sample will not be considered 'evaluable'.

If a pre-dose sample is collected on the same day as the first dose of oral bridging, the time of the first dose (not recorded in eCRF) is assumed to be 'after' the collection of pre-dose sample, unless medical monitor or Data querying informs otherwise.

The time-deviation (hours) from the targeted timepoint will be calculated for the samples '1-Week-POST' only using the following formula:

Time\_deviation (hrs) for '1-Week-POST' = Sample date.time - last previous injection date.time - 7\*24 hours

The following windows are for defining 'evaluable' Long-term Follow-up phase PK concentrations.

| Timepoint | Evaluable Window | For Programming: |
|---|---|---|
| LTFU MONTH<br>1/WD | ± 4 days | 24 days ≤ Days Since Last Injection ≤ 32 days |
| LTFU MONTH 3 | ± 1 Weeks | 77 days ≤ Days Since Last Injection ≤ 91 days |
| LTFU MONTH 6 | ± 2 Weeks | 154 days ≤ Days Since Last Injection ≤ 182 days |
| LTFU MONTH 9 | ± 2 Weeks | 238 days ≤ Days Since Last Injection ≤ 266 days |
| LTFU MONTH 12 | ± 2 Weeks | 322 days ≤ Days Since Last Injection ≤ 350 days |

### 15.6.6. Health Outcomes

# Questionnaire (Questions 1-12 are scored Collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.



### **Total Treatment Satisfaction Score**

- Total Treatment Satisfaction Score is computed with items 1-11. Items 1-11 are summed to produce a score with a possible range of to ...
- Item 12 will not be included in Total Treatment Satisfaction Score. Instead, it will be treated as a stand-alone item only.
- Higher scores represent greater treatment satisfaction as compared to the past few weeks.
- A maximum of 5 items can be missing, which can be imputed to reflect the mean of the completed item scores. If 6 or more items are missing, then the treatment satisfaction scale score should not be computed and instead be imputed using LOCF.

### **Individual Item Scores**

- Items are rated as (CC), etc.).
- Higher scores represent greater satisfaction with each aspect of treatment
  - For individual item scores outputs, missing scores will not be computed (according to Page 7 of the [HIVTSQ User Guidelines, 2016]) and instead be imputed using LOCF.

### **HIVTSQc**

# Questionnaire (Questions 1-12 are scored to



# **Total Treatment Satisfaction Score (change)**

- Total Treatment Satisfaction Score is computed with items 1-11. Items 1-11 are summed to produce a score with a possible range of column to column to column.
- Item 12 will be computed as an individual item only.
- The higher the score, the greater the improvement in satisfaction with treatment; the lower the score, the greater the deterioration in satisfaction with treatment. A score of represents
- A maximum of 5 items can be missing, the missing scores will be imputed with the mean of the
  completed item scores. If 6 or more items are missing, then the overall treatment satisfaction
  scale score should not be computed and will remain missing.

# **Individual Treatment Satisfaction Change Item Scores**

- Items are rated as CCI (CCI etc.) to CI (CCI etc.).
- The higher the score, the greater the improvement in satisfaction with each aspect of treatment and the lower the score, the greater the deterioration in satisfaction with each aspect of treatment.

### **Questionnaire Version**

- Three versions of the HIVTSQc questionnaire are available with the questions the same and only the overhead text is different.
  - Q4W ATLAS to Q4W ATLAS-2M: for participants who randomized to Q4W arm in ATLAS and then randomized to Q4W arm in ATLAS-2M
  - Q4W ATLAS to Q8W ATLAS-2M: for participants who randomized to Q4W arm in ATLAS and then randomized to Q8W arm in ATLAS-2M
  - SOC to Q4W or Q8W ATLAS-2M: for participants who either were randomized to SOC arm in ATLAS or did not participate in ATLAS
- If a participant takes a wrong version of the questionnaire, the data collected from the wrong version will be considered invalid and will not be included in the summary.

### PIN

# Questionnaire (Each question is scored







# Life satisfaction, HIV medications, disclosure worries

The ratings for Items (a, b, c, d, e) will be recoded as below for analysis:
 Response option
 Life Satisfaction
 Medication/disclosure worries

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or ndices, which are protected by third party copyright laws and therefore have been excluded.

- A maximum of 50% question items can be missing within a domain, which can be computed and replaced with the mean of the completed item scores within the domain. Thus, if there are more than 1 item missing for Life Satisfaction, and more than 2 items missing for Medication/disclosure worries, then the total score for the domain should not be computed and instead be imputed using LOCF (Section 15.7.2.2). A computed score for missing value will be added to calculate a total score for the domain. Total score for each of the three domains will be calculated and will be denoted as 'LISAT' for life satisfaction, 'MEDWO' for medication worries, and 'DISWO' for disclosure worries.
- Transform each dimension's total imputed value score to the 0-100 scale using the following formulae:

Life satisfaction: CCI
Medication worries: CCI

Disclosure worries:

The higher the score, the greater satisfaction to life and the less worry. The transformed dimension score for each domain will be summarized and analysed.

### **Individual Item Scores**

• For individual item scores outputs, missing scores will not be computed and instead be imputed using LOCF (Section 15.7.2.2).

### ACCEPT (Acceptance/General Dimension) (Gilet H et al, 2014)

Questionnaire (Questions 1-3 constitute to Acceptance/General Dimension)

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protecte by third party copyright laws and therefore have been excluded.



- □ Other, please specify
- 3. What is the main benefit related to this HIV therapy supporting your preference?
- □ More convenient, easier to integrate into one's daily life
- □ Less stressful
- □ Less stigma
- □ Easier to take the drug exactly as prescribed
- □ More efficacious
- □ Other, please specify

### **Questionnaire Version**

- Two versions of questionnaire are available. The questions in each version of the questionnaire are the same and only the overhead text is different.
  - ATLAS (from Q4W ATLAS): for participants randomized to Q4W arm in ATLAS.
  - ATLAS-2M (from SOC ATLAS or out): for participants who either were randomized to SOC arm in ATLAS or did not participate in ATLAS.

# **Data Handling**

Any missing values will remain missing (i.e. no imputation).

### Reasons for Continuation/Switch

# Questionnaires

- Reasons for Continuation questionnaire is collected for participants who were randomized to Q4W arm in ATLAS.
- Reason for Switch questionnaire is collected for participants who either were randomized to SOC arm in ATLAS or did not participate in ATLAS.

### **Data Handling**

- If a participant takes a wrong questionnaire, for example, the participant randomized to SOC arm in ATLAS took Reasons for Continuation questionnaire, the data collected from this wrong version will be considered invalid and will not be included in the summary.
- If the questionnaire is taken beyond ± 2 weeks window from maintenance phase treatment start date (i.e. Study Day < -14 or Study Day > 14) will be consider not evaluable and will not be included in the summary.
- Any missing values will remain missing (i.e. no imputation).

### 15.6.7. Virology

### Genotype

### **Amino Acid Changes**

- A mutation is considered present whenever the encoded amino acid residue differs from the amino acid that would have been encoded by the wild-type (e.g., HXB2, NL43) comparator gene; e.g., Q148K.
- If the encoded amino acid is seen as a mixture of wild-type and mutant amino acid, e.g., Q148Q/K, the mutated amino acid is considered present at the codon of interest.
- If the encoded amino acid is seen as a mixture of two or more amino acids, which may or may
  not include wild type, e.g., Q184K/H or Q184K/H/Q, etc., for the purposes of calculating the
  number of mutated amino acids, only one mutation is considered to be present at the codon of
  interest.

# **Representation of Amino Acid Changes**

| Mutations | Amino acid change |
|---|---|
| T69S | Single mutation from amino acid 'T' (vendor reference) to 'S' (sample) at codon '69' |
| Q148H/K/R | Mixture of amino acid mutations 'H', 'K' and 'R' (sample) from amino acid 'Q' (vendor reference) at codon '148' |
| _69_1T | First insertion of amino acid 'T' (sample) at codon '69' |
| _69_2S | Second insertion of amino acid 'S' (sample) at codon '69' |
| _69_3S/A | Third insertion of a mixture of amino acids 'S' and 'A' (sample) at codon '69' |
| L74L/- | Mixture of amino acid 'L' (sample) and a deletion at codon '74' |
| V75- | Single deletion of amino acid (sample) at codon '75' |

### **Resistance Associated Mutations**

Known INI mutations associated with the development of resistance to BIC, RAL, EVG or DTG:

| HIV Integrase for | H51Y, <b>T66A/I/K</b> , <b>E92Q/V</b> /G, Q95K, T97A, G118R, <b>F121Y</b> , E138A/K/T, G140A/C/R/S**, <b>Y143C/H/R/K/S/G/A</b> , <b>P145S</b> , <b>Q146P</b> , <b>S147G</b> , <b>Q148H/K/R/N</b> , <b>V151</b> I/L/A, S153F/Y, <b>N155H</b> /S/T, E157Q, G163R/K, S230R, R263K, L68V/I*, L74I/M*, E138D*, V151I*, G193E* |
|---|---|
|---|---|

### NOTES:

- Draft listing; may be modified in case of additional substantive data availability.
- INI mutations listed taken from Stanford HIV Resistance Database (<a href="http://hivdb.stanford.edu/DR/cgi-bin/rules">http://hivdb.stanford.edu/DR/cgi-bin/rules</a> scores hivdb.cgi?class=INI cited 18Jul2018) and accessed on 06Oct2018.
- Each INI mutation listed had a score of ≥15. INI substitutions listed above in bold had a score of =60.
- \* Denotes additional INI mutations added as they were identified during in vitro passage of DTG or seen in a previous DTG study in INI-experienced participants (ING112574).
- \*\*G140R is potentially associated with CAB based on in-stream data monitoring of CVF participants.
- Major resistance mutations to other classes (i.e., NRTI, NNRTI, PI) as defined by the International Antiviral Society-USA (IAS-USA). The most up to date IAS-USA guidelines available at the time of DBF will be used in the analysis [Wensing AM et al 2017].

| Class | Mutations |
|---|---|
| NRTIs | M41L, A62V, K65R/E/N, D67N, 69 insert, K70E/R, L74V, V75I, F77L, Y115F, F116Y, |
| | Q151M, M184V/I, L210W, T215Y/F, K219Q/E |
| NNRTIs | L100I, K101E/P, K103N/S, V106A/M, V108I, E138/A/G/K/Q/R, V179L, |
| | Y181C/I/V, Y188C/L/H, G190S/A, H221Y, P225H, F227C, M230I/L, |
| Pls | D30N, V32I, M46I/L, I47A/V, G48V, I50V/L, I54M/L, Q58E, T74P, L76V, |
| | V82A/T/F/L/S, N83D, I84V, N88S, L90M |
| Note: List generated from IAS_USA Guideline, [Wensing et al. 2017] | |

# Phenotype

# Phenotypic Susceptibility

Phenotypic susceptibility to all licensed antiretroviral drugs and CAB will be determined using PhenoSense HIV assays from Monogram Inc. and will be reported as fold change (FC) in IC50 relative to wild-type control virus NL4-3, i.e., FC of sample virus = IC50 of sample virus/IC50 of control virus.

Phenotypic susceptibilities will be categorised according to FC as shown in tables below (based on Monogram PhenoSense assay). Clinical cutoffs (where available) or biological cutoffs by PhenoSense will be used to define the phenotypic susceptibility of background treatment by Monogram.

Replication capacity is generated as part of standard phenotypic assays.

# **PhenoSense Algorithm**

| Drug | Abbreviation | Class | PhenoSense cutoff |
|-----------------|--------------|-------|-------------------|
| Abacavir | ABC | NRTI | (4.5 – 6.5)a |
| Lamivudine | 3TC | NRTI | 3.5 a |
| Didanosine | ddl | NRTI | (1.3 – 2.2) a |
| Stavudine | d4T | NRTI | 1.7 a |
| Zidovudine | AZT (ZDV) | NRTI | 1.9 |
| Emtricitabine | FTC | NRTI | 3.5 |
| Tenofovir | TDF (TAF) | NRTI | (1.4 – 4) a |
| Delavirdine | DLV | NNRTI | 6.2 |
| Efavirenz | EFV | NNRTI | 3 |
| Nevirapine | NVP | NNRTI | 4.5 |
| Etravirine | ETR | NNRTI | (2.9-10) a |
| Rilpivirine | RPV | NNRTI | 2.0 |
| Fosamprenavir/r | FPV/r | PI | (4-11) a |
| Atazanavir | ATV | PI | 2.2a |
| Atazanavir/r | ATV/r | PI | 5.2 a |
| Indinavir/r | IDV/r | PI | 10 a |
| Lopinavir/r | LPV/r | PI | (9 – 55) a |
| Nelfinavir | NFV | PI | 3.6 |
| Saquinavir/r | SQV/r | PI | (2.3 – 12) a |
| Tipranavir/r | TPV/r | PI | (2 – 8) a |
| Darunavir/r | DRV/r | PI | (10 – 90) a |
| Ritonavir | RTV | PI | 2.5 |
| Enfuvirtide | T20 | FI | 6.48 |
| Cabotegravir | CAB | INI | 2.5 |
| Raltegravir | RAL | INI | 1.5 |
| Elvitegravir | EVG | INI | 2.5 |
| Dolutegravir | DTG | INI | (4-13) a |
| Bictegravir | BIC | INI | (2.5- 10) |

a. clinical cutoff (lower cutoff – higher cutoff).

### Phenotypic Susceptibility

Phenotypic susceptibility to each drug in a participant's background regimen is determined by applying drug-associated cutoffs as defined by the PhenoSense algorithm to the phenotypic fold resistance as below:

# **Full Sensitivity**

| Fold Change | Interpretation |
|----------------------------------------------|----------------|
| > clinical lower cutoff or biological cutoff | resistant |
| ≤ clinical lower cutoff or biological cutoff | sensitive |

# **Partial Sensitivity**

| Fold Change | Interpretation |
|------------------------------------------------------|---------------------|
| > clinical higher cutoff | resistant |
| ≤ clinical higher cutoff and > clinical lower cutoff | partially sensitive |
| ≤ clinical lower cutoff | sensitive |

PHENOTYP dataset from Monogram contains the phenotypic susceptibility for each drug derived from the cutoff listed above. Thus, phenotypic susceptibility (i.e. full sensitivity and partial sensitivity) will not be re-derived for our analysis.

# **Genotypic and Net Assessment Susceptibility**

Genotypic and Net assessment susceptibility to all licensed antiretroviral drugs and CAB will be determined from Monogram Inc. Net assessment susceptibility will be reported with the categories of 'resistant', 'partially sensitive', and 'sensitive' as what will be performed for phenotypic susceptibility. Genotypic susceptibility will be reported with the categories of 'resistant', 'resistance possible' and 'sensitive'. Genotypic and Net assessment susceptibility will be assessed at time of CVF using plasma sample, Genotypic susceptibility may be assessed at baseline using PBMC.

# 15.7. Appendix 7: Reporting Standards for Missing Data

# 15.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (i.e. as specified in the protocol) was defined as <ul> <li>Randomly assigned to either treatment group, completed the randomized Maintenance Phase including Week 100 and did not enter the Extension Phase;</li> <li>Randomly assigned to either treatment group, completed the randomized Maintenance Phase including Week 100, and entered and completed the Extension Phase (defined as remaining on study until commercial supplies of CAB LA + RPV LA Q4W or Q8W regimen become locally available or development of CAB LA + RPV LA is terminated).</li> </ul> </li> </ul> |
| | Participants who withdraw from CAB LA + RPV LA and go into the LTFU Phase, and participants who withdraw from oral lead-in will be considered to have prematurely withdrawn from the study treatment. |
| | In addition to the 52-week Follow-Up phase required for participants who receive one or more injections with CAB LA or RPV LA, an in-clinic Follow-Up visit will be conducted approximately 4 weeks after the last dose of study medication for participants who withdraw during the oral lead-in period with ongoing AEs, and serious adverse events (SAEs) and also any laboratory abnormalities that are considered to be AEs or potentially harmful to the participant, at the last on-study visit. Assessments at the Follow-up visit should reflect any ongoing complaints (e.g., blood draws to follow a laboratory abnormality). Follow-Up visits are not required for successful completion of the study. |
| | Withdrawn participants were not replaced in the study. |
| | <ul> <li>All available data from participants who were withdrawn from the study will be listed<br/>and all available planned data will be included in summary tables and figures, unless<br/>otherwise specified.</li> </ul> |
| | Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits. |

# 15.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 15.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | eneral • Partial dates will be displayed as captured in participant listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment State.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> </ul> |
| | <ul> <li>Completely missing start or end dates will remain missing, with no imputation<br/>applied. Consequently, time to onset and duration of such events will be<br/>missing.</li> </ul> |
| ART/Non-<br>ART<br>Medications<br>or Medical<br>History | <ul> <li>Partial dates recorded in the eCRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month. If medications recorded in the eCRF as prior (e.g. recorded in prior ART or prior ATLAS ART forms, taken prior to study), the earlier date of the imputed and the day prior to the maintenance phase treatment start date will be used, i.e. min (imputed stop date, maintenance phase treatment start date - 1).</li> </ul> </li> <li>For medications with completely missing start date, they will be considered started prior to the maintenance phase treatment start date.</li> <li>For medications with completely missing stop date, they will be considered ongoing unless recorded in eCRF as prior (e.g. recorded in prior ART or prior ATLAS ART forms, taken prior to study).</li> <li>For ART booster medications, the start and stop dates are not recorded in the database (i.e. missing), the dates will be imputed to be the same as the dates of their parent medications.</li> <li>The recorded partial or missing date will be displayed in listings.</li> </ul> |
| Health outcomes | <ul> <li>For the health outcomes questionnaire data, please refer to Section12.</li> <li>For the summary of individual item scores outputs, missing scores will not be computed.</li> </ul> |

# 15.7.2.2. Handling of Missing data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| Snapshot | <ul> <li>In the Snapshot dataset, participants without HIV-1 RNA data in the assessment window for the visit of interest (due to missing data or discontinuation of IP prior to the visit window) do not belong to 'HIV-1 RNA &lt; 50 c/mL (or &lt;200 c/mL)'. The nature of this missing data will be further classified in Snapshot summaries as either 'HIV-1 RNA ≥ 50 c/mL' (or "HIV-1 RNA ≥ 200 c/mL') or 'No Virologic Data at Week X'; Appendix 9: Snapshot Algorithm Details for full details</li> </ul> |
| LOCF | • In the LOCF dataset, missing values will be carried forward from the previous, non-missing available on-treatment assessment. If the baseline value is missing any missing values until the first non-missing value will remain missing. |
| Lipid LOCF | <ul> <li>Baseline for Lipids LOCF Analyses:</li> <li>Last evaluable lipids assessment up to and including the start of IP, where 'evaluable' is defined as: Lipid modifying agents not taken within 12 weeks of the date of assessment and Lipids are collected in a fasting state. Participants with unevaluable Baseline for Lipids (as defined above) will be excluded from this dataset.</li> <li>During the Maintenance:</li> <li>If participants initiate serum lipid-lowering agents during the maintenance, then the last available fasted on-treatment lipid values prior to the initiation will be used in place of future, observed on-treatment values.</li> <li>Imputation at visits with observed on-treatment values will continue even if the participant discontinues the lipid-lowering agent. Missing assessments will not be imputed</li> </ul> |
| Analyses Evaluated with Lipid LOCF Dataset: | |
| | This dataset will be used to summarize fasting lipids parameters in the following displays: Summary of Fasting TC/HDL ratio Change from Baseline Summary of Fasting Lipids Percentage Changes from Baseline |
| | All other displays of lipids (e.g. toxicity tables and NCEP tables) will use observed fasting data, without LOCF imputation. |

# 15.8. Appendix 8: Values of Potential Clinical Importance

ECG values of potential clinical importance are defined as QTc > 500 msec or increase from baseline in QTc  $\geq$  60 msec.

# 15.9. Appendix 9: Snapshot Algorithm Details

# **Detailed Algorithm Steps**

- Consider an analysis visit window for Week X as defined in Table 10.
- The HIV-1 RNA threshold of 50, 200 c/mL will be analysed, respectively, in this study
- The analysis window 'Week 48' and HIV-1 RNA threshold of '50 c/mL' are used for the purpose of illustration. A participant's Snapshot response and reason at Week 48 are categorized as below.
  - o HIV-1 RNA < **50** c/mL o HIV-1 RNA ≥ **50** c/mL Data in window not below 50 Discontinued for lack of efficacy Discontinued for other reason while not below 50 Change in background therapy\*
  - o No Virologic Data at Week 48 Window
    Discontinued study due to AE or death
    Discontinued study for other reasons
    On study but missing data in window
  - \* Note: since permanent change in ART are not permitted in this protocol, all such participants who permanently change ART will be considered 'HIV-1 RNA ≥ 50 c/mL' if the permanent change in ART is made prior to an analysis timepoint. Participants with protocol permitted oral bridging treatment or a temporary change in ART prior to an analysis timepoint (e.g. participant took the ART different from study treatment during oral lead-in by mistake for a short period and then went back to the study treatment) will not be considered 'HIV-1 RNA ≥ 50 c/mL' due to 'change in ART'.
- The steps in determining response and reasons are indicated in the table below, in the order stated:

### **Detailed steps**

Please note that the following scenarios will NOT be penalized Per Snapshot algorithm (i.e. please exclude these scenarios from **Condition** 1-4).

• Dose reduction, dropping a component, or change in formulation (e.g. 'Tivicay + Kivexa' to 'Triumeg' with the identical ingredients)

| Condition ('Week 48' indicates Week 48 window) | | Response | Reasons |
|---|---|---|---|
| 1 | . If non-permitted change in background therapy prior to Week 48 | HIV-1 RNA ≥ 50 | Change in background therapy |
| 2 | If permitted change <sup>[a]</sup> in background therapy prior to Week 48<br>AND the latest on-treatment VL prior to/on the date of change<br>is ≥ 50 c/mL (NA to this study) | HIV-1 RNA ≥ 50 | Change in background therapy |

| | 1 | |
|---|---|---|
| <ol> <li>If non-permitted change in background therapy during Week</li> <li>48</li> </ol> | | |
| <ul> <li>Last on-treatment VL during Week 48 prior to/on the date<br/>of change ≥ 50 c/mL</li> </ul> | HIV-1 RNA ≥<br>50 | Data in<br>window not<br>below 50 |
| <ul> <li>Last on-treatment VL during Week 48 prior to/on the date<br/>of change &lt; 50 c/mL</li> </ul> | HIV-1 RNA <<br>50 | |
| No VL during Week 48 prior to/on the date of change | HIV-1 RNA ≥<br>50 | Change in background therapy |
| <ol> <li>If permitted change<sup>[a]</sup> in background therapy during Week 48 AND the last on-treatment VL prior to/on the date of change is ≥ 50 c/mL (NA to this study)</li> </ol> | | |
| 4.1 this last on-treatment VL occurs prior to Week 48 | HIV-1 RNA ≥ 50 | Change in background therapy |
| 4. 2 this last on-treatment VL occurs during Week 48 but prior to/on the date of change | HIV-1 RNA ≥ 50 | Data in<br>window not<br>below 50 |
| 5. If none of the above conditions met | | |
| 5.1 On-treatment VL available during Week 48 | | |
| Last on-treatment VL during Week 48 ≥ 50 c/mL | HIV-1 RNA ≥ 50 | Data in<br>window not<br>below 50 |
| Last on-treatment VL during Week 48 < 50 c/mL | HIV-1 RNA < 50 | |
| 5.2 No on-treatment VL during Week 48 | | |
| 5.2.1 If participants still on study, i.e. a participant has not permanently discontinued the study treatment yet, or if a participant permanently discontinued the study treatment and the upper bound of analysis snapshot window is prior to the following date: Q8W arm: Min[max(Date of last injection + 63, Date of Last Dose of Carl OAR DRY (1) With Javant Date 1 | No virologic<br>data at Week<br>48 Window | On study<br>but missing<br>data in<br>window |
| Oral CAB+RPV + 1), Withdrawal Date] Q4W arm: Min[max(Date of last injection + 35, Date of Last Dose of | | |
| T | 1 | 1 |
|---|---|---|
| Oral CAB+RPV + 1), Withdrawal Date] , where 'Withdrawal Date' refers to the date the failed to complete per corresponding conclusion | | |
| 5.2.2 If participants withdraw before/during Week | | |
| 5.2.2.1 Safety reasons (e.g. AE/death, liver che stopping criteria, renal toxicity withdrawal criteria etc, as recorded in eCRF (form) | eria, QTc data at Week | Disc due to<br>AE/death |
| 5.2.2.2 Non-safety related reasons (e.g. Lack efficacy, protocol deviation, withdrew consent follow-up, study closed/terminated, investigat discretion etc, as recorded in eCRF Conclusion | t, loss to<br>or | |
| <ul> <li>Last on-treatment VL &lt;50 c/mL OR no on-treatment vl &lt;50 c/mL or on-treatm</li></ul> | atment VL No virologic<br>Data at<br>Week 48<br>Window | Disc for other reasons |
| <ul> <li>Last on-treatment VL ≥ 50 c/mL AND withdra<br/>Lack of efficacy</li> </ul> | wal due to HIV-1 RNA ≥ 50 | Disc. for lack of efficacy |
| <ul> <li>Last on-treatment VL ≥ 50 c/mL AND withdra<br/>all other non-safety related reasons</li> </ul> | wal due to HIV-1 RNA ≥ 50 | Disc. for<br>other<br>reason<br>while not<br>below 50 |

a. Excluding permitted change in background therapy where change or decision to change is made prior to/on the first on-treatment viral result

## **Examples from FDA guidance**

#### Data in Window

Virologic outcome should be determined by the last available measurement while the patient is on treatment and continued on trial within the time window:

 HIV-1 RNA = 580 c/mL at Day 336, HIV-1 RNA below 50 c/mL on Day 350. This should be categorized as HIV-1 RNA below 50 c/mL.

#### No Data in Window

Discontinued study due to Adverse Event or Death:

- Any patient who discontinues because of an AE or death before the window should be classified as *Discontinued due to AE or Death* (as appropriate), regardless of the HIV-1 RNA result, even if the HIV-1 RNA is below 50 c/mL at the time of discontinuation.
- However, if a patient has an HIV-1 RNA value in the time window and also discontinues in the time window, the viral load data should be used to classify the patient's response. This is the Virology First hierarchy:

- a. HIV-1 RNA below 50 c/mL at Day 336 and discontinues because of AE or even dies on Day 360 — this person is categorized as having HIV-1 RNA below 50 c/mL.
- b. HIV-1 RNA is 552 c/mL on Day 336 and the patient discontinues on Day 360, the patient is categorized as having HIV-1 RNA ≥ 50 c/mL.

#### Discontinued for Other Reasons:

- Only patients who have achieved virologic suppression can be counted as Discontinued for Other Reasons.
- If a patient discontinues the study before the time window because of *lack of efficacy* then
  the patient should be included in the HIV-1 RNA ≥ 50 row and not in the Discontinued for
  Other Reasons row.
- If a patient discontinues because *participant withdrew consent* and his or her HIV-1 RNA result at the time of discontinuation was equal to or above 50 c/mL, then he or she should be categorized as HIV-1 RNA ≥ 50 and NOT as Discontinued for Other Reasons.
- If a patient discontinued because of *Lost to Follow-Up* and the last HIV-1 RNA result was 49 c/mL, then the patient can be categorized as Discontinued for Other Reasons.
- If patients changed background treatment not permitted by protocol— they should be considered an efficacy failure and captured in the HIV-1 RNA ≥ 50 c/mL row.

#### On study but missing data in window:

- If there are no data during Days 294 to 377, but there is an HIV-1 RNA below 50 c/mL on Day 380, this patient should be considered *On Study but Missing Data in Window.*
- If there are no data during Days 294 to 377, but there is an HIV-1 RNA equal to or above 50 c/mL on Day 280, this patient also should be classified as *On Study but Missing Data in Window*.

# 15.10. Appendix 10: Variables Defined for Time to Event Analysis

| Programming Instructions for the Kaplan-Meier analysis of treatment-related discontinuation equals failure (TRDF) | | |
|---|---|---|
| Condition | Censor<br>Status | Event Description/AVAL |
| Participant met CVF event criteria during the Maintenance Phase (based on derived CVF) | CNSR=0 | EVNTDESC=CVF AVAL=Study Day of SVF* *immediately preceding CVF |
| 2. Participant with Maintenance Phase withdrawal due to 'Lack of Efficacy', 'Treatment Related AE', 'Intolerability due to Injection', or 'Protocol Defined Safety Stopping Criteria' during Maintenance Phase Note: primary reason and/or standardized subreason for discontinuation based on Maintenance Conclusion form in the eCRF. 'Protocol Defined Safety Stopping Criteria' includes GSK defined liver chemistry stopping criteria, renal toxicity criteria and QTc withdrawal criteria. Treatment Related AE' is defined as participants who have primary reason for withdrawal =AE and who have at least one AE considered drug related and leading to withdrawal/permanent discontinuation of investigational product. | CNSR=0 | EVNTDESC= terms in italic, respectively. For Q4W arm: AVAL= min [Study Day of Maintenance Phase Discontinuation, max(Study Day of Last Injection + 35, Study Day of Last Dose of Oral CAB+RPV + 1)] For Q8W arm: AVAL= min [Study Day of Maintenance Phase Discontinuation, max(Study Day of Last Injection + 63, Study Day of Last Dose of Oral CAB/RPV + 1)] Note: Date of Maintenance Phase discontinuation is from the Maintenance Phase Conclusion form in the eCRF. |
| If none of the above conditions met | CNSR=1 | EVNTDESC-'Consored due to Study Discontinuation |
| Participant with Maintenance Phase withdrawal due to other | CNOK=1 | EVNTDESC='Censored due to Study Discontinuation for Other Reasons' |
| reasons | ONOD 4 | AVAL will be defined as the same as above 2 |
| 4. Participant who did not have premature withdrawal from | CNSR=1 | EVNTDESC='Censored due to data cutoff for analysis' |

| Programming Instructions for the Kaplan-Meier analysis of treatment-related discontinuation equals failure (TRDF) | | |
|---|---|---|
| Condition | Censor<br>Status | Event Description/AVAL |
| the Maintenance Phase | | AVAL = Study Day of last on-treatment date during the maintenance phase, which is defined as follows: For Q4W arm: min [Study Day of Nominal Week 100 Visit, Study Day of LTFU ART Start Date, Study Day of Last Contact Date at time of analysis, max(Study Day of Last Injection + 35, Study Day of Last Dose of Oral CAB+RPV + 1)] |
| | | For Q8W arm min [Study Day of Nominal Week 100 Visit, Study Day of LTFU ART Start Date, Study Day of Last Contact Date at time of analysis, max(Study Day of Last Q8W IM Dose + 63, Study Day of Last Dose of Oral CAB+RPV + 1)] |

Note that last injection and last dose of oral CAB+RPV mentioned in table above are only applied to participants who permanently discontinued from the study treatment. The similar approach will be used to derive for Kaplan-Meier analysis of efficacy-related discontinuation equals failure (ERDF), except that the reason of withdrawal in Condition 2 will be restricted to 'Lack of Efficacy'.

# 15.11. Appendix 11: Identification of Adverse Events of Special Interest

The adverse events of special interest are identified based on MedDRA coded values and/or AE data available in the study database. The system organ classes (SOCs), preferred terms (PTs) or codes, Standardised MedDRA Queries (SMQs), High Level Group Terms (HLGTs), and High Level Terms (HLTs) below are from MedDRA 21.1. SMQs use narrow terms unless otherwise specified. In case there is a change to the version of MedDRA at time of reporting, the coded values based on the MedDRA version at the time of reporting will be used. The additional events may also be added based on the blinded review of AE data collected on study prior to the database freeze.

## 1. Hepatic Safety Profile: Assessment of risk of hepatoxicity

## Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions (SMQ)

| РТ | PT Code |
|--------------------------------------|----------|
| Acquired hepatocerebral degeneration | 10080860 |
| Acute hepatic failure | 10000804 |
| Acute on chronic liver failure | 10077305 |
| Acute yellow liver atrophy | 10070815 |
| Ascites | 10003445 |
| Asterixis | 10003547 |
| Bacterascites | 10068547 |
| Biliary cirrhosis | 10004659 |
| Biliary fibrosis | 10004664 |
| Cholestatic liver injury | 10067969 |
| Chronic hepatic failure | 10057573 |
| Coma hepatic | 10010075 |
| Cryptogenic cirrhosis | 10063075 |
| Diabetic hepatopathy | 10071265 |
| Drug-induced liver injury | 10072268 |
| Duodenal varices | 10051010 |
| Gallbladder varices | 10072319 |
| Gastric variceal injection | 10076237 |
| Gastric variceal ligation | 10076238 |
| Gastric varices | 10051012 |
| Gastric varices haemorrhage | 10057572 |
| Hepatectomy | 10061997 |
| Hepatic atrophy | 10019637 |
| Hepatic calcification | 10065274 |
| Hepatic cirrhosis | 10019641 |
| Hepatic encephalopathy | 10019660 |
| Hepatic encephalopathy prophylaxis | 10066599 |

| PT | PT Code |
|--------------------------------------|----------|
| Hepatic failure | 10019663 |
| Hepatic fibrosis | 10019668 |
| Hepatic hydrothorax | 10067365 |
| Hepatic infiltration eosinophilic | 10064668 |
| Hepatic lesion | 10061998 |
| Hepatic necrosis | 10019692 |
| Hepatic steato-fibrosis | 10077215 |
| Hepatic steatosis | 10019708 |
| Hepatitis fulminant | 10019772 |
| Hepatobiliary disease | 10062000 |
| Hepatocellular foamy cell syndrome | 10053244 |
| Hepatocellular injury | 10019837 |
| Hepatopulmonary syndrome | 10052274 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Hepatotoxicity | 10019851 |
| Intestinal varices | 10071502 |
| Intestinal varices haemorrhage | 10078058 |
| Liver and small intestine transplant | 10052280 |
| Liver dialysis | 10076640 |
| Liver disorder | 10024670 |
| Liver injury | 10067125 |
| Liver operation | 10062040 |
| Liver transplant | 10024714 |
| Lupoid hepatic cirrhosis | 10025129 |
| Minimal hepatic encephalopathy | 10076204 |
| Mixed liver injury | 10066758 |
| Nodular regenerative hyperplasia | 10051081 |
| Non-alcoholic fatty liver | 10029530 |
| Non-alcoholic steatohepatitis | 10053219 |
| Non-cirrhotic portal hypertension | 10077259 |
| Oedema due to hepatic disease | 10049631 |
| Oesophageal varices haemorrhage | 10030210 |
| Peripancreatic varices | 10073215 |
| Portal fibrosis | 10074726 |
| Portal hypertension | 10036200 |
| Portal hypertensive colopathy | 10079446 |
| Portal hypertensive enteropathy | 10068923 |
| Portal hypertensive gastropathy | 10050897 |

| PT | PT Code |
|---------------------------------------|----------|
| Portal vein cavernous transformation | 10073979 |
| Portal vein dilatation | 10073209 |
| Portopulmonary hypertension | 10067281 |
| Primary biliary cholangitis | 10080429 |
| Regenerative siderotic hepatic nodule | 10080679 |
| Renal and liver transplant | 10052279 |
| Retrograde portal vein flow | 10067338 |
| Reye's syndrome | 10039012 |
| Reynold's syndrome | 10070953 |
| Splenic varices | 10067823 |
| Splenic varices haemorrhage | 10068662 |
| Steatohepatitis | 10076331 |
| Subacute hepatic failure | 10056956 |
| Varices oesophageal | 10056091 |
| Varicose veins of abdominal wall | 10072284 |
| White nipple sign | 10078438 |

# Hepatitis, non-infectious (SMQ)

| PT | PT Code |
|--------------------------------------------|----------|
| Acute graft versus host disease in liver | 10066263 |
| Allergic hepatitis | 10071198 |
| Alloimmune hepatitis | 10080576 |
| Autoimmune hepatitis | 10003827 |
| Chronic graft versus host disease in liver | 10072160 |
| Chronic hepatitis | 10008909 |
| Graft versus host disease in liver | 10064676 |
| Hepatitis | 10019717 |
| Hepatitis acute | 10019727 |
| Hepatitis cholestatic | 10019754 |
| Hepatitis chronic active | 10019755 |
| Hepatitis chronic persistent | 10019759 |
| Hepatitis fulminant | 10019772 |
| Hepatitis toxic | 10019795 |
| Immune-mediated hepatitis | 10078962 |
| Ischaemic hepatitis | 10023025 |
| Lupus hepatitis | 10067737 |
| Non-alcoholic steatohepatitis | 10053219 |
| Radiation hepatitis | 10051015 |
| Steatohepatitis | 10076331 |

# 2. Hypersensitivity Reactions (HSR)

# Drug reaction with eosinophilia and systemic symptoms syndrome (SMQ)

| PT | PT Code |
|-------------------------------------------------------|----------|
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |
| Pseudolymphoma | 10037127 |

# PTs (Selective)

| PT | PT Code |
|-----------------------------------|----------|
| Drug hypersensitivity | 10013700 |
| Hypersensitivity | 10020751 |
| Type IV Hypersensitivity reaction | 10053613 |
| Eosinophillia | 10014950 |
| Eye swelling | 10015967 |
| Eyelid oedema | 10015993 |
| Lip swelling | 10024570 |
| Angioedema | 10002424 |
| Circumoral oedema | 10052250 |
| Face oedema | 10016029 |
| Idiopathic angioedema | 10073257 |
| Lip oedema | 10024558 |
| Mouth swelling | 10075203 |
| Oedema mouth | 10030110 |
| Periorbital oedema | 10034545 |
| Swelling face | 10042682 |
| Periorbital swelling | 10056647 |
| Swelling of eyelid | 10042690 |

# 3. Rash

## Severe cutaneous adverse reactions (SMQ)

| PT | PT Code |
|-------------------------------------------------------|----------|
| Acute generalised exanthematous pustulosis | 10048799 |
| Cutaneous vasculitis | 10011686 |
| Dermatitis bullous | 10012441 |
| Dermatitis exfoliative | 10012455 |
| Dermatitis exfoliative generalised | 10012456 |
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |

| PT | PT Code |
|-----------------------------|----------|
| Epidermal necrosis | 10059284 |
| Erythema multiforme | 10015218 |
| Exfoliative rash | 10064579 |
| Oculomucocutaneous syndrome | 10030081 |
| Skin necrosis | 10040893 |
| Stevens-Johnson syndrome | 10042033 |
| Toxic epidermal necrolysis | 10044223 |
| Toxic skin eruption | 10057970 |

# PTs (Selective), Grade 3 and higher

| PT | PT Code |
|----------------------|----------|
| Eyelid rash | 10074620 |
| Genital rash | 10018175 |
| Mucocutaneous rash | 10056671 |
| Nodular rash | 10075807 |
| Perineal rash | 10075364 |
| Rash | 10037844 |
| Rash erythematous | 10037855 |
| Rash generalised | 10037858 |
| Rash macular | 10037867 |
| Rash maculo-papular | 10037868 |
| Rash maculovesicular | 10050004 |
| Rash morbilliform | 10037870 |
| Rash papular | 10037876 |
| Rash rubelliform | 10057984 |
| Rash scarlatiniform | 10037890 |
| Rash vesicular | 10037898 |
| Rash pruritic | 10037884 |
| Rash follicular | 10037857 |
| Rash pustular | 10037888 |
| Drug eruption | 10013687 |

# 4. Prolongation of the Corrected QT Interval of the ECG in Supratherapeutic Doses Torsade de pointes/QT prolongation (SMQ)

| PT | PT Code |
|----------------------------------------|----------|
| Electrocardiogram QT interval abnormal | 10063748 |

| PT | PT Code |
|--------------------------------|----------|
| Electrocardiogram QT prolonged | 10014387 |
| Long QT syndrome | 10024803 |
| Long QT syndrome congenital | 10057926 |
| Torsade de pointes | 10044066 |
| Ventricular tachycardia | 10047302 |

# PTs (Selective)

| PT | PT Code |
|----------------------------------------------|----------|
| Electrocardiogram repolarisation abnormality | 10052464 |

## 5. Suicidal Ideation/Behaviour

# Suicide/self-injury (SMQ)

| PT | PT Code |
|-------------------------------------------------|----------|
| Assisted suicide | 10079105 |
| Columbia suicide severity rating scale abnormal | 10075616 |
| Completed suicide | 10010144 |
| Depression suicidal | 10012397 |
| Intentional overdose | 10022523 |
| Intentional self-injury | 10022524 |
| Poisoning deliberate | 10036000 |
| Self-injurious ideation | 10051154 |
| Suicidal behaviour | 10065604 |
| Suicidal ideation | 10042458 |
| Suicide attempt | 10042464 |
| Suicide threat | 10077417 |
| Suspected suicide attempt | 10081704 |

# 6. Depression

# Depression (excl suicide and self injury) (SMQ)

| PT | PT Code |
|-----------------------------------------------------------|----------|
| Activation syndrome | 10066817 |
| Adjustment disorder with depressed mood | 10001297 |
| Adjustment disorder with mixed anxiety and depressed mood | 10001299 |
| Agitated depression | 10001496 |
| Anhedonia | 10002511 |

| PT | PT Code |
|---------------------------------------|----------|
| Antidepressant therapy | 10054976 |
| Childhood depression | 10068631 |
| Decreased interest | 10011971 |
| Depressed mood | 10012374 |
| Depression | 10012378 |
| Depression postoperative | 10012390 |
| Depressive symptom | 10054089 |
| Dysphoria | 10013954 |
| Electroconvulsive therapy | 10014404 |
| Feeling guilty | 10049708 |
| Feeling of despair | 10016344 |
| Feelings of worthlessness | 10016374 |
| Helplessness | 10077169 |
| Major depression | 10057840 |
| Menopausal depression | 10067371 |
| Mixed anxiety and depressive disorder | 10080836 |
| Perinatal depression | 10078366 |
| Persistent depressive disorder | 10077804 |
| Post stroke depression | 10070606 |
| Postictal depression | 10071324 |

# 7. Bipolar Disorder

# **HLGT Manic and Bipolar mood disorders and disturbances**

| PT | PT Code |
|----------------------|----------|
| Bipolar I disorder | 10004939 |
| Bipolar II disorder | 10004940 |
| Bipolar disorder | 10057667 |
| Cyclothymic disorder | 10011724 |
| Hypomania | 10021030 |
| Mania | 10026749 |

# 8. Psychosis

# Psychosis and psychotic disorders (SMQ)

| PT | PT Code |
|---------------------|----------|
| Acute psychosis | 10001022 |
| Alcoholic psychosis | 10001632 |

| PT | PT Code |
|---------------------------------------------------|----------|
| Alice in wonderland syndrome | 10001666 |
| Brief psychotic disorder with marked stressors | 10048549 |
| Brief psychotic disorder without marked stressors | 10056395 |
| Brief psychotic disorder, with postpartum onset | 10006362 |
| Charles Bonnet syndrome | 10063354 |
| Childhood psychosis | 10061040 |
| Clang associations | 10009232 |
| Cotard's syndrome | 10059591 |
| Delusion | 10012239 |
| Delusion of grandeur | 10012241 |
| Delusion of reference | 10012244 |
| Delusion of replacement | 10012245 |
| Delusional disorder, erotomanic type | 10012249 |
| Delusional disorder, grandiose type | 10012250 |
| Delusional disorder, jealous type | 10012251 |
| Delusional disorder, mixed type | 10012252 |
| Delusional disorder, persecutory type | 10053195 |
| Delusional disorder, somatic type | 10012254 |
| Delusional disorder, unspecified type | 10012255 |
| Delusional perception | 10012258 |
| Dementia of the Alzheimer's type, with delusions | 10012295 |
| Depressive delusion | 10063033 |
| Derailment | 10012411 |
| Epileptic psychosis | 10059232 |
| Erotomanic delusion | 10015134 |
| Flight of ideas | 10016777 |
| Hallucination | 10019063 |
| Hallucination, auditory | 10019070 |
| Hallucination, gustatory | 10019071 |
| Hallucination, olfactory | 10019072 |
| Hallucination, synaesthetic | 10062824 |
| Hallucination, tactile | 10019074 |
| Hallucination, visual | 10019075 |
| Hallucinations, mixed | 10019079 |
| Hypnagogic hallucination | 10020927 |
| Hypnopompic hallucination | 10020928 |
| Hysterical psychosis | 10062645 |
| Ideas of reference | 10021212 |
| Illusion | 10021403 |

| PT | PT Code |
|-------------------------------------------------------|----------|
| Jealous delusion | 10023164 |
| Loose associations | 10024825 |
| Mixed delusion | 10076429 |
| Neologism | 10028916 |
| Neuroleptic-induced deficit syndrome | 10075295 |
| Paranoia | 10033864 |
| Paranoid personality disorder | 10033869 |
| Parkinson's disease psychosis | 10074835 |
| Paroxysmal perceptual alteration | 10063117 |
| Persecutory delusion | 10034702 |
| Postictal psychosis | 10070669 |
| Post-injection delirium sedation syndrome | 10072851 |
| Posturing | 10036437 |
| Psychosis postoperative | 10065617 |
| Psychotic behaviour | 10037249 |
| Psychotic disorder | 10061920 |
| Psychotic disorder due to a general medical condition | 10061921 |
| Reactive psychosis | 10053632 |
| Rebound psychosis | 10074833 |
| Schizoaffective disorder | 10039621 |
| Schizoaffective disorder bipolar type | 10068889 |
| Schizoaffective disorder depressive type | 10068890 |
| Schizophrenia | 10039626 |
| Schizophreniform disorder | 10039647 |
| Schizotypal personality disorder | 10039651 |
| Senile psychosis | 10039987 |
| Shared psychotic disorder | 10040535 |
| Somatic delusion | 10041317 |
| Somatic hallucination | 10062684 |
| Substance-induced psychotic disorder | 10072388 |
| Tangentiality | 10043114 |
| Thought blocking | 10043495 |
| Thought broadcasting | 10052214 |
| Thought insertion | 10043496 |
| Thought withdrawal | 10043497 |
| Transient psychosis | 10056326 |
| Waxy flexibility | 10047853 |

# 9. Mood Disorders

# **HLGT Mood disorders and disturbances NEC, Psychiatric disorders SOC**

| PT | PT Code |
|----------------------------------------|----------|
| Crying | 10011469 |
| Mood swings | 10027951 |
| Boredom | 10048909 |
| Mood altered | 10027940 |
| Apathy | 10002942 |
| Affective ambivalence | 10077173 |
| Emotional poverty | 10014557 |
| Euphoric mood | 10015535 |
| Premenstrual dysphoric disorder | 10051537 |
| Alexithymia | 10077719 |
| Laziness | 10051602 |
| Blunted affect | 10005885 |
| Constricted affect | 10010778 |
| Affect lability | 10054196 |
| Anger | 10002368 |
| Affective disorder | 10001443 |
| Lethargy | 10024264 |
| Listless | 10024642 |
| Inappropriate affect | 10021588 |
| Dysphoria | 10013954 |
| Mood disorder due to a general medical | |
| condition | 10027944 |
| Morose | 10027977 |
| Screaming | 10039740 |
| Steroid withdrawal syndrome | 10042028 |
| Emotional disorder | 10014551 |
| Irritability | 10022998 |
| Moaning | 10027783 |
| Premenstrual syndrome | 10036618 |
| Neuroleptic-induced deficit syndrome | 10075295 |
| Substance-induced mood disorder | 10072387 |
| Flat affect | 10016759 |
| Diencephalic syndrome of infancy | 10012774 |
| Emotional distress | 10049119 |
| Frustration tolerance decreased | 10077753 |
| Seasonal affective disorder | 10039775 |

# 10. Anxiety

# **HLGT Anxiety disorders and symptoms**

| РТ | PT Code |
|-----------------------------------------------------|----------|
| Acrophobia | 10000605 |
| Activation syndrome | 10066817 |
| Acute stress disorder | 10001084 |
| Aerophobia | 10080300 |
| Agitation | 10001497 |
| Agitation neonatal | 10001500 |
| Agitation postoperative | 10049989 |
| Agoraphobia | 10001502 |
| Akathisia | 10001540 |
| Algophobia | 10078056 |
| Animal phobia | 10002518 |
| Anniversary reaction | 10074066 |
| Anticipatory anxiety | 10002758 |
| Anxiety | 10002855 |
| Anxiety disorder | 10057666 |
| Anxiety disorder due to a general medical condition | 10002859 |
| Arachnophobia | 10051408 |
| Astraphobia | 10078372 |
| Autophobia | 10071070 |
| Body dysmorphic disorder | 10052793 |
| Burnout syndrome | 10065369 |
| Claustrophobia | 10009244 |
| Compulsions | 10010219 |
| Compulsive cheek biting | 10076510 |
| Compulsive handwashing | 10071263 |
| Compulsive hoarding | 10068007 |
| Compulsive lip biting | 10066241 |
| Compulsive shopping | 10067948 |
| Dermatillomania | 10065701 |
| Dysmorphophobia | 10049096 |
| Emetophobia | 10070637 |
| Fear | 10016275 |
| Fear of animals | 10016276 |
| Fear of closed spaces | 10016277 |
| Fear of crowded places | 10050365 |
| Fear of death | 10066392 |

| PT | PT Code |
|-------------------------------------------------------------|----------|
| Fear of disease | 10016278 |
| Fear of eating | 10050366 |
| Fear of falling | 10048744 |
| Fear of injection | 10073753 |
| Fear of open spaces | 10016279 |
| Fear of pregnancy | 10067035 |
| Fear of weight gain | 10016280 |
| Fear-related avoidance of activities | 10080136 |
| Generalised anxiety disorder | 10018075 |
| Glossophobia | 10080077 |
| Haemophobia | 10073458 |
| Haphephobia | 10067580 |
| Hydrophobia | 10053317 |
| Hyperarousal | 10080831 |
| Immunisation anxiety related reaction | 10075205 |
| Kinesiophobia | 10078430 |
| Limited symptom panic attack | 10024511 |
| Mysophobia | 10078769 |
| Nail picking | 10066779 |
| Nervousness | 10029216 |
| Neurosis | 10029333 |
| Noctiphobia | 10057946 |
| Nocturnal fear | 10057948 |
| Nosophobia | 10063546 |
| Obsessive need for symmetry | 10077179 |
| Obsessive rumination | 10056264 |
| Obsessive thoughts | 10029897 |
| Obsessive-compulsive disorder | 10029898 |
| Obsessive-compulsive symptom | 10077894 |
| Ochlophobia | 10050095 |
| Osmophobia | 10060765 |
| Paediatric autoimmune neuropsychiatric disorders associated | 40070447 |
| with streptococcal infection | 10072147 |
| Panic attack | 10033664 |
| Panic disorder | 10033666 |
| Panic reaction | 10033670 |
| Paruresis | 10069024 |
| Performance fear | 10034432 |
| Phagophobia | 10050096 |
| Pharmacophobia | 10069423 |

| PT | PT Code |
|--------------------------------|----------|
| Phobia | 10034912 |
| Phobia of driving | 10056676 |
| Phobia of exams | 10034913 |
| Phobic avoidance | 10034918 |
| Phonophobia | 10054956 |
| Photaugiaphobia | 10064420 |
| Post-traumatic stress disorder | 10036316 |
| Postpartum neurosis | 10036419 |
| Postpartum stress disorder | 10056394 |
| Procedural anxiety | 10075204 |
| Pseudoangina | 10056610 |
| Selective mutism | 10039917 |
| Separation anxiety disorder | 10040045 |
| Sitophobia | 10080170 |
| Social anxiety disorder | 10041242 |
| Social fear | 10041247 |
| Stress | 10042209 |
| Tension | 10043268 |
| Terminal agitation | 10077416 |
| Thanatophobia | 10064723 |
| Thermophobia | 10075147 |
| Trichotemnomania | 10072752 |
| Trichotillomania | 10044629 |

# 11. Sleep Disorders

# **HLGT Sleep Disorders and Disturbances**

| PT | PT Code |
|-----------------------------------|----------|
| Behavioural insomnia of childhood | 10072072 |
| Hyposomnia | 10067530 |
| Initial insomnia | 10022035 |
| Insomnia | 10022437 |
| Middle insomnia | 10027590 |
| Terminal insomnia | 10068932 |
| Breathing-related sleep disorder | 10006344 |
| Dyssomnia | 10061827 |
| Hypersomnia | 10020765 |
| Periodic limb movement disorder | 10064600 |
| Pickwickian syndrome | 10035004 |

| PT | PT Code |
|-------------------------------------------------------------|----------|
| Poor quality sleep | 10062519 |
| Sleep apnoea syndrome | 10040979 |
| Somnolence | 10041349 |
| Somnolence neonatal | 10041350 |
| Stupor | 10042264 |
| Upper airway resistance syndrome | 10063968 |
| Cataplexy | 10007737 |
| Hypnagogic hallucination | 10020927 |
| Hypnopompic hallucination | 10020928 |
| Narcolepsy | 10028713 |
| Sleep attacks | 10040981 |
| Sleep paralysis | 10041002 |
| Abnormal dreams | 10000125 |
| Abnormal sleep-related event | 10061613 |
| Confusional arousal | 10067494 |
| Exploding head syndrome | 10080684 |
| Loss of dreaming | 10065085 |
| Nightmare | 10029412 |
| Parasomnia | 10061910 |
| Rapid eye movement sleep behaviour disorder | 10077299 |
| Rapid eye movements sleep abnormal | 10037841 |
| Sleep inertia | 10067493 |
| Sleep sex | 10067492 |
| Sleep talking | 10041009 |
| Sleep terror | 10041010 |
| Sleep-related eating disorder | 10067315 |
| Somnambulism | 10041347 |
| Hypersomnia related to another mental condition | 10020767 |
| Hypersomnia-bulimia syndrome | 10053712 |
| Insomnia related to another mental condition | 10022443 |
| Sleep disorder | 10040984 |
| Sleep disorder due to a general medical condition | 10063910 |
| Sleep disorder due to general medical condition, | |
| hypersomnia type | 10040985 |
| Sleep disorder due to general medical condition, | |
| insomnia type | 10040986 |
| Sleep disorder due to general medical condition, mixed type | 10040987 |
| Sleep disorder due to general medical condition, | 10040301 |
| parasomnia type | 10040988 |
| Sopor | 10058709 |

| PT | PT Code |
|--------------------------------------|----------|
| Advanced sleep phase | 10001423 |
| Circadian rhythm sleep disorder | 10009191 |
| Delayed sleep phase | 10012209 |
| Irregular sleep phase | 10022995 |
| Irregular sleep wake rhythm disorder | 10080301 |
| Non-24-hour sleep-wake disorder | 10078086 |
| Shift work disorder | 10078088 |

# **HLGT Sleep disturbances (incl subtypes)**

| PT | PT Code |
|--------------------------------------|----------|
| Abnormal dreams | 10000125 |
| Abnormal sleep-related event | 10061613 |
| Confusional arousal | 10067494 |
| Loss of dreaming | 10065085 |
| Sleep inertia | 10067493 |
| Sleep paralysis | 10041002 |
| Sleep sex | 10067492 |
| Sleep talking | 10041009 |
| Sleep terror | 10041010 |
| Sleep-related eating disorder | 10067315 |
| Somnambulism | 10041347 |
| Behavioural insomnia of childhood | 10072072 |
| Hyposomnia | 10067530 |
| Initial insomnia | 10022035 |
| Insomnia | 10022437 |
| Middle insomnia | 10027590 |
| Terminal insomnia | 10068932 |
| Advanced sleep phase | 10001423 |
| Circadian rhythm sleep disorder | 10009191 |
| Delayed sleep phase | 10012209 |
| Irregular sleep phase | 10022995 |
| Irregular sleep wake rhythm disorder | 10080301 |
| Non-24-hour sleep-wake disorder | 10078086 |
| Shift work disorder | 10078088 |
| Cataplexy | 10007737 |
| Hypersomnia | 10020765 |
| Narcolepsy | 10028713 |
| Central-alveolar hypoventilation | 10007982 |
| Sleep apnoea syndrome | 10040979 |

| PT | PT Code |
|---------------------------------------------|----------|
| Breathing-related sleep disorder | 10006344 |
| Dyssomnia | 10061827 |
| Fatal familial insomnia | 10072077 |
| Microsleep | 10076954 |
| Periodic limb movement disorder | 10064600 |
| Pickwickian syndrome | 10035004 |
| Poor quality sleep | 10062519 |
| Rapid eye movement sleep behaviour disorder | 10077299 |
| Rapid eye movements sleep abnormal | 10037841 |
| Sleep deficit | 10080881 |
| Sudden onset of sleep | 10050014 |
| Upper airway resistance syndrome | 10063968 |

## 12. Injection Site Reactions (ISR) from Study Drug Injections

Study drug ISR data available in the database, i.e. data collected from non-serious ISR AE eCRF form and collected serious adverse events with 'STUDY DRUG INJECTION SITE' included in the AE term.

#### 13. Seizures and Seizure-like Events

# Convulsions (SMQ)

| PT | PT Code |
|--------------------------------------------------------|----------|
| 2-Hydroxyglutaric aciduria | 10078971 |
| Acquired epileptic aphasia | 10052075 |
| Acute encephalitis with refractory, repetitive partial | |
| seizures | 10076948 |
| Alcoholic seizure | 10056347 |
| Aspartate-glutamate-transporter deficiency | 10079140 |
| Atonic seizures | 10003628 |
| Atypical benign partial epilepsy | 10056699 |
| Automatism epileptic | 10003831 |
| Autonomic seizure | 10049612 |
| Baltic myoclonic epilepsy | 10054895 |
| Benign familial neonatal convulsions | 10067866 |
| Benign rolandic epilepsy | 10070530 |
| Biotinidase deficiency | 10071434 |
| Change in seizure presentation | 10075606 |
| Clonic convulsion | 10053398 |
| Convulsion in childhood | 10052391 |

| PT | PT Code |
|------------------------------------------------------|----------|
| Convulsion neonatal | 10010911 |
| Convulsions local | 10010920 |
| Convulsive threshold lowered | 10010927 |
| CSWS syndrome | 10078827 |
| Deja vu | 10012177 |
| Double cortex syndrome | 10073490 |
| Dreamy state | 10013634 |
| Drug withdrawal convulsions | 10013752 |
| Early infantile epileptic encephalopathy with burst- | |
| suppression | 10071545 |
| Eclampsia | 10014129 |
| Epilepsy | 10015037 |
| Epilepsy surgery | 10079824 |
| Epilepsy with myoclonic-atonic seizures | 10081179 |
| Epileptic aura | 10015049 |
| Epileptic psychosis | 10059232 |
| Febrile convulsion | 10016284 |
| Febrile infection-related epilepsy syndrome | 10079438 |
| Focal dyscognitive seizures | 10079424 |
| Frontal lobe epilepsy | 10049424 |
| Generalised non-convulsive epilepsy | 10018090 |
| Generalised tonic-clonic seizure | 10018100 |
| Glucose transporter type 1 deficiency syndrome | 10078727 |
| Gray matter heterotopia | 10080533 |
| Hemimegalencephaly | 10078100 |
| Hyperglycaemic seizure | 10071394 |
| Hypocalcaemic seizure | 10072456 |
| Hypoglycaemic seizure | 10048803 |
| Hyponatraemic seizure | 10073183 |
| Idiopathic generalised epilepsy | 10071081 |
| Infantile spasms | 10021750 |
| Juvenile myoclonic epilepsy | 10071082 |
| Lafora's myoclonic epilepsy | 10054030 |
| Lennox-Gastaut syndrome | 10048816 |
| Migraine-triggered seizure | 10076676 |
| Molybdenum cofactor deficiency | 10069687 |
| Multiple subpial transection | 10079825 |
| Myoclonic epilepsy | 10054859 |
| Myoclonic epilepsy and ragged-red fibres | 10069825 |
| Partial seizures | 10061334 |

| PT | PT Code |
|------------------------------------------------|----------|
| Partial seizures with secondary generalisation | 10056209 |
| Petit mal epilepsy | 10034759 |
| Polymicrogyria | 10073489 |
| Post stroke epilepsy | 10076982 |
| Post stroke seizure | 10076981 |
| Postictal headache | 10052470 |
| Postictal paralysis | 10052469 |
| Postictal psychosis | 10070669 |
| Postictal state | 10048727 |
| Post-traumatic epilepsy | 10036312 |
| Schizencephaly | 10073487 |
| Seizure | 10039906 |
| Seizure anoxic | 10039907 |
| Seizure cluster | 10071350 |
| Seizure like phenomena | 10071048 |
| Severe myoclonic epilepsy of infancy | 10073677 |
| Simple partial seizures | 10040703 |
| Status epilepticus | 10041962 |
| Sudden unexplained death in epilepsy | 10063894 |
| Temporal lobe epilepsy | 10043209 |
| Tonic clonic movements | 10051171 |
| Tonic convulsion | 10043994 |
| Tonic posturing | 10075125 |
| Topectomy | 10073488 |
| Transient epileptic amnesia | 10081728 |
| Tuberous sclerosis complex | 10080584 |
| Uncinate fits | 10045476 |

# PTs (Selective)

| PT | PT Code |
|----------------------------------|----------|
| Confusional state | 10010305 |
| Loss of consciousness | 10024855 |
| Syncope | 10042772 |
| Sopor | 10058709 |
| Stupor | 10042264 |
| Altered state of consciousness | 10050093 |
| Depressed level of consciousness | 10012373 |
| Consciousness fluctuating | 10050093 |

# 14. Weight Gain

# **HLT General nutritional disorders NEC (Selective)**

| PT | PT Code |
|----------------------|----------|
| Abdominal fat apron | 10077983 |
| Overweight | 10033307 |
| Abnormal weight gain | 10000188 |
| Central obesity | 10065941 |
| Obesity | 10029883 |

# HLT Physical examination procedures and organ system status (Selective)

| PT | PT Code |
|----------------------------------------|----------|
| Weight abnormal | 10056814 |
| Weight increased 10047899 | |
| Waist circumference increased 10064863 | |
| Body mass index abnormal 10074506 | |
| Body mass index increased 10005897 | |

# **General signs and symptoms NEC (Selective)**

| PT PT Code | |
|----------------------|----------|
| Fat tissue increased | 10016251 |

## 15. Rhabdomyolysis

# Rhabdomyolysis/myopathy (SMQ)

| PT | PT Code |
|----------------------------------|----------|
| Muscle necrosis | 10028320 |
| Myoglobin blood increased | 10028625 |
| Myoglobin blood present | 10059888 |
| Myoglobin urine present 10028631 | |
| Myoglobinaemia 10058735 | |
| Myoglobinuria | 10028629 |
| Myopathy | 10028641 |
| Myopathy toxic | 10028648 |
| Necrotising myositis | 10074769 |

| PT | PT Code |
|---------------------|----------|
| Rhabdomyolysis | 10039020 |
| Thyrotoxic myopathy | 10081524 |

# PTs (Selective)

| PT | PT Code |
|----------|----------|
| Myalgia | 10028411 |
| Myositis | 10028653 |

# 16. Pancreatitis

# Acute pancreatitis (SMQ)

| PT | PT Code |
|------------------------------------|----------|
| Cullen's sign | 10059029 |
| Grey Turner's sign | 10075426 |
| Haemorrhagic necrotic pancreatitis | 10076058 |
| Hereditary pancreatitis | 10056976 |
| Ischaemic pancreatitis | 10066127 |
| Oedematous pancreatitis | 10052400 |
| Pancreatic abscess | 10048984 |
| Pancreatic haemorrhage | 10033625 |
| Pancreatic necrosis | 10058096 |
| Pancreatic phlegmon 10056975 | |
| Pancreatic pseudoaneurysm 10081762 | |
| Pancreatic pseudocyst 10033635 | |
| Pancreatic pseudocyst drainage | 10033636 |
| Pancreatitis | 10033645 |
| Pancreatitis acute 10033647 | |
| Pancreatitis haemorrhagic 10033650 | |
| Pancreatitis necrotising 10033654 | |
| Pancreatitis relapsing 10033657 | |
| Pancreatorenal syndrome | 10056277 |

# 17. Impact on Creatinine

# Acute renal failure (SMQ)

| PT | PT Code |
|-----------------------------|----------|
| Acute kidney injury | 10069339 |
| Acute phosphate nephropathy | 10069688 |

| PT | PT Code |
|---------------------------------|----------|
| Anuria | 10002847 |
| Azotaemia | 10003885 |
| Continuous haemodiafiltration | 10066338 |
| Dialysis | 10061105 |
| Foetal renal impairment | 10078987 |
| Haemodialysis | 10018875 |
| Haemofiltration | 10053090 |
| Hyponatriuria | 10077515 |
| Neonatal anuria 10049778 | |
| Nephropathy toxic 10029155 | |
| Oliguria | 10030302 |
| Peritoneal dialysis | 10034660 |
| Prerenal failure 10072370 | |
| Renal failure 10038435 | |
| Renal failure neonatal 10038447 | |
| Renal impairment 10062237 | |
| Renal impairment neonatal | 10049776 |

# Renal Failure and Impairment HLT

| PT | PT Code |
|-------------------------------------------|----------|
| Acute Kidney injury | 10069339 |
| Anuria | 10002847 |
| Atypical haemolytic uraemic syndrome | 10079840 |
| Cardiorenal syndrome | 10068230 |
| Chronic kidney disease | 10064848 |
| Crush syndrome | 10050702 |
| Diabetic end stage renal disease 10012660 | |
| End stage renal disease 10077512 | |
| Foetal renal impairment 10078987 | |
| Haemolytic uraemic syndrome 10018932 | |
| Hepatorenal failure 10019845 | |
| Hepatorenal syndrome 10019846 | |
| Nail-patella syndrome 10063431 | |
| Neonatal anuria 10049778 | |
| Oliguria 10030302 | |
| Pancreatorenal syndrome 10056277 | |
| Postoperative renal failure 10056675 | |
| Postrenal failure 10059345 | |
| Prerenal failure 10072370 | |

| PT | PT Code |
|------------------------------------|----------|
| Propofol infusion syndrome | 10063181 |
| Renal failure | 10038435 |
| Renal failure neonatal 10038447 | |
| Renal impairment 10062237 | |
| Renal impairment neonatal 10049776 | |
| Renal injury 10061481 | |
| Scleroderma renal crisis 10062553 | |
| Traumatic anuria | 10044501 |

# 18. Safety in Pregnancy

Use AE terms co-reported in pregnancy exposures to CAB and/or RPV.

## 15.12. Appendix 12: IDMC

Independent review will be provided by an IDMC to ensure external objective medical and/or statistical review of efficacy and safety in order to protect the ethical interests and well-being of participants and to protect the scientific validity of this study. An ad-hoc review of data by the IDMC will be triggered whenever the number of confirmed virologic failures in the Q8W arm exceeds thresholds pre-specified in the IDMC charter. Further, analyses including futility checking will be performed for the IDMC to evaluate the efficacy and safety when approximately 50% of participants have completed their visit at Week 24.

The list of required outputs is provided in the IDMC Charter, Section 12.3, Appendix C.

Data handing methods and derived data definitions will be the same as detailed in this RAP, unless otherwise stated.

## 15.12.1. Adhoc CVF IDMC Analyses

The number of participants meeting Confirmed Virologic Failure (CVF) Criterion per the protocol will be monitored and may result in ad-hoc IDMC data reviews.

The Statistics Data Analysis Centre (SDAC) will be notified by the study virologist in writing every time a CVF occurs in the study. The SDAC will track the number of participants on Q8W arm past Week 4. The rate of CVF will be monitored against the thresholds specified in IDMC Charter Table 1 (See IDMC Charter, Section 3.5.2).

## 15.12.2. Week 24 IDMC Analyses

Analyses including futility checking will be performed when approximately 50% of participants have completed their Week 24 visit.

A futility rule will assess the evidence that the CAB LA + RPV LA Q8W arm is non-inferior to the Q4W control arm. This rule will use the interim data (~ 50% participants completing Week 24) to calculate the Bayesian predictive probabilities that the CAB LA + RPV LA Q8W arm is non-inferior to the Q4W arm at Week 24. A 4% non-inferiority margin will be used. The details of statistical methods can be found in IDMC Charter, Section 12.6.1. The list of outputs is also provided in Section 15.14.4.

# 15.13. Appendix 13: Abbreviations & Trademarks

# 15.13.1. Abbreviations

| Abbreviation | Description |
|--------------|------------------------------------------------------------|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AESI | Adverse Events of Special Interest |
| BMI | Body Mass Index |
| CAB | Cabotegravir |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| СМН | Cochran-Mantel-Haenszel |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| eC-SSRS | Electronic Columbia Suicide Severity Rating Scale |
| CVb | Coefficient of Variation (Between) |
| CVD | Cardiovascular Disease |
| CVF | Confirmed Virologic Failure |
| DAIDS | Division of AIDS |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Place |
| DTG | Dolutegravir |
| eCRF | Electronic Case Record Form |
| eGFR | Estimated Glomerular Filtration Rate |
| EMA | European Medicines Agency |
| ERDF | Efficacy Related Discontinuation Failure |
| FDA | Food and Drug Administration |
| FSFV | First Subject First Visit |
| GSK | GlaxoSmithKline |
| GUI | Guidance |
| HAT-QoL | Health-related Quality of Life |
| HBV | Hepatitis B Virus |
| HCV | Hepatitis C Virus |
| HIV | Human Immunodeficiency Virus |
| HIVTSQc | Change Version of HIV Treatment Satisfaction Questionnaire |
| HIVTSQs | Status Version of HIV Treatment Satisfaction Questionnaire |
| HLGT | High Level Group Term |
| HLT | High Level Term |
| HSR | Hypersensitivity Reaction |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |

| IMMS | International Modules Management System |
|-------|--------------------------------------------------|
| INI | Integrase Inhibitors |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| ITT-E | Intent-To-Treat Exposed |
| LOCF | Last Observation Carries Forward |
| MMRM | Mixed Model Repeated Measures |
| NA | Not Applicable |
| NCEP | National Cholesterol Education Program |
| NNRTI | Non-Nucleoside Reverse Transcriptase Inhibitors |
| NQ | Non Quantifiable |
| NRTI | Nucleoside Reverse Transcriptase Inhibitors |
| OC | Observed Case |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PI | Protease Inhibitors |
| PIN | Perception of Injection |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PT | Preferred Term |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAMOS | Randomization & Medication Ordering System |
| RAP | Reporting & Analysis Plan |
| RPV | Rilpivirine |
| SAE | Serious Adverse Event |
| SAC | Statistical Analysis Complete |
| SD | Standard Deviation |
| SDAC | Statistics Data Analysis Centre |
| SDRP | Study Results Dissemination Plan |
| SDTM | Study Data Tabulation Model |
| SMQ | Standardised MedDRA Query |
| SOC | System Organ Class |
| SOP | Standard Operation Procedure |
| TFL | Tables, Figures & Listings |
| TRDF | Treatment Related Discontinuation Failure |

# 15.13.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| Tivicay |
| Triumeq |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| Edurant |
| NONMEM |
| SAS |
| WinNonlin |

## 15.14. Appendix 14: List of Data Displays

## 15.14.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|-----------------------------------|------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Pharmacokinetic / Pharmacodynamic | 5.1 to 5.n | 5.1 to 5.n |
| Health Outcomes | 6.1 to 6.n | 6.1 to 6.n |
| Virology | 7.1 to 7.n | 7.1 to 7.n |
| Section | Listi | ngs |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

## 15.14.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays will be provided in a separate document.

The example mock-up displays from other reporting efforts will be named in the format: Study Number/HARP Reporting Effort/Output Type (T/ F/L)/Display Number, where T stands for Table, F stands for Figure and L stands for Listing. For example, the Table 1.1 from primary\_02 reporting effort for Study 201585 will be named by 201585/primary 02/T1.1.

Other example mock-up displays will be named using the following format.

| Section | Figure | Table | Listing |
|-----------------------------------|---------|---------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |
| Health Outcomes | HO_Fn | HO_Tn | HO_Ln |
| Virology | VIR_Fn | VIR_Tn | VIR_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column.

#### 15.14.3. Deliverables

| Delivery [1] | Description |
|---|---|
| IW24 | IDMC analyses when approximately 50% participants have completed |

| Delivery [1] | Description |
|---|---|
| | their Week 24 visits |
| W24 | Week 24 when 100% participants have completed their Week 24 visits |
| HL | Headline at Week 48 |
| W48 | Week 48 |
| W96 | Week 96 |
| EOS | End of study |

#### NOTES:

# 15.14.4. List of Data Displays for Week 24 IDMC and Week 24 Planned Analyses

For Week 24 planned analyses, the Week 24 Futility population will be replaced by the Intent-to-Treat Exposed population. In addition, unless otherwise specified, present the listings by prior exposure to CAB+RPV (i.e. rederived randomization strata, 0, 1-24, >24 weeks, refer to Section 15.6.2 for calculation details) except for study population listings.

<sup>1.</sup> Indicates order in which displays will be generated for the reporting effort

# 15.14.4.1. Study Population Tables

| Study P | Study Population Tables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Subject | Disposition | on | | | | |
| 1.1 | NA | Week 24<br>Futility | ES1 | Summary of Subject Accountability: Maintenance Phase Conclusion Record - Week 24 Futility | ICH E3, GSKCTR, FDAAA,<br>EudraCT, see also in<br>201585/primary_02/T1.7. | IW24 |
| 1.2 | 1.1 | Intent-to-<br>Treat<br>Exposed | ES1 | Summary of Subject Accountability: Maintenance<br>Phase Conclusion Record - ITT-E | ICH E3, GSKCTR, FDAAA,<br>EudraCT, see also in<br>201585/primary_02/T1.7. | IW24, W24 |
| Demogr | aphic and | Baseline Cha | racteristics | | | |
| 1.3 | NA | Week 24<br>Futility | 201585/primary_02/T1.16 | Summary of Demographic Characteristics - Week 24 Futility | ICH E3, FDAAA, EudraCT | IW24 |
| 1.4 | 1.2 | Intent-to-<br>Treat<br>Exposed | 201585/primary_02/T1.16 | Summary of Demographic Characteristics - ITT-E | ICH E3, FDAAA, EudraCT | IW24, W24 |
| 1.5 | NA | Week 24<br>Futility | 201584/idmc_03/T1.3 | Summary of Prior Exposure to CAB+RPV - Week 24 Futility | Adjust footnote and row labels as appropriate. | IW24 |
| 1.6 | 1.3 | Intent-to-<br>Treat<br>Exposed | 201584/idmc_03/T1.3 | Summary of Prior Exposure to CAB+RPV - ITT-E | Adjust footnote and row labels as appropriate. | IW24, W24 |
| 1.7 | 1.4 | Intent-to-<br>Treat<br>Exposed | 201584/idmc_03/T1.7 | Summary of Prior Exposure to CAB+RPV by Country | Adjust footnote and row labels as appropriate. | IW24, W24 |
| 1.8 | 1.5 | Intent-to-<br>Treat<br>Exposed | 201585/primary_02/T1.19 | Summary of Hepatitis Status at Entry | Add footnote as appropriate for subjects classified as Hepatitis B positive in analysis. | IW24, W24 |

# 15.14.4.2. Efficacy Tables

| Efficacy | Efficacy Tables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.1 | 2.1 | Week 24<br>Futility | 201585/primary_02/T2.1 | Summary of Analysis for<br>Proportion of Subjects with<br>Plasma HIV-1 RNA ≥50 c/mL at<br>Week 24 and Posterior Predictive<br>Probability of Success for the<br>Q8W Arm - Snapshot Analysis | For Week 24 IDMC, add a column on right with 'Posterior Predictive Probability of Success" and adjust the footnotes as appropriate, also add a footnote "Target threshold for posterior predictive probability is 15%.". For planned Week 24, remove 'and Posterior Predictive Probability of Success for the Q8W Arm' from the title, adjust the footnote as appropriate. For proportions, keep one decimal place. The adjustment is based on rederived randomization strata. | IW24, W24 |
| 2.2 | 2.2 | Week 24<br>Futility | 201585/primary_02/T2.4 | Summary of Study Outcomes (50 c/mL Threshold) at Week 24 (Maintenance Phase) - Snapshot Analysis | For proportions, keep one decimal place. | IW24, W24 |
| 2.3 | 2.3 | Week 24<br>Futility | 201585/primary_02/T2.6 | Summary of Analysis for<br>Proportion of Subjects with<br>Plasma HIV-1 RNA ≥50 c/mL at<br>Week 24 by Randomization<br>Strata (Maintenance Phase) -<br>Snapshot Analysis | Note that only by randomization strata summary is provided. Change the footnote to "[1] Difference: Proportion on Q8W - Proportion on Q4W. 95% Cls were calculated using an unconditional exact method with two inverted one-sided tests based on the score statistic." Add Footnote "Note: Randomization strata are rederived using the prior exposure to CAB+RPV in Study 201585, collected from eCRF." For proportions, keep one decimal place. | IW24, W24 |

| Efficac | Efficacy Tables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.4 | 2.4 | Week 24<br>Futility | 201585/primary_02/T2.21 | Cumulative Proportion of<br>Subjects Meeting Confirmed<br>Virologic Failure by Visit (Up to<br>Week 24) | For proportions, keep one decimal place. Non-snapshot visit window will be used. | IW24, W24 |
| 2.5 | 2.5 | Week 24<br>Futility | 201585/primary_02/T2.21 | Cumulative Proportion of<br>Subjects Meeting Confirmed<br>Virologic Failure by Visit and<br>Randomization Strata (Up to<br>Week 24) | Add column for 'Analysis Strata', add footnote for randomization strata similar to T2.3. For proportions, keep one decimal place. Non-snapshot visit window will be used. | IW24, W24 |
| 2.6 | 2.6 | Intent-to-<br>Treat<br>Exposed | 201585/primary_02/T2.21 | Cumulative Proportion of<br>Subjects Meeting Confirmed<br>Virologic Failure during the<br>Maintenance Phase | Note that this is overall summary, not by visit. Replace the column 'Timepoint' with 'CVF Category'. For proportions, keep one decimal place. | IW24, W24 |
| 2.7 | 2.7 | Intent-to-<br>Treat<br>Exposed | 201584/idmc_03/T2.7 | Cumulative Proportion of<br>Subjects Meeting Confirmed<br>Virologic Failure by<br>Randomization Strata during the<br>Maintenance Phase | Adjust footnote and row labels as appropriate. For proportions, keep one decimal place. Use rederived Randomization strata. | IW24, W24 |
| 2.8 | 2.8 | Week 24<br>Futility | EFF_T1 | Summary of Kaplan-Meier Estimates of Proportion of Subjects without CVF at Week 24 - Treatment Related Discontinuation = Failure | The non-snapshot visit window for Week 24 will be used. | IW24, W24 |

| Efficacy | Efficacy Tables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 2.9 | 2.9 | Week 24<br>Futility | EFF_T2 | Summary of Kaplan-Meier Estimates of Proportion of Subjects without CVF at Week 24 - Efficacy Related Discontinuation=Failure | The non-snapshot visit window for Week 24 will be used. | IW24, W24 |
| 2.10 | 2.10 | Intent-to-<br>Treat<br>Exposed | 201584/idmc_03/T2.10 | Proportion of Subjects with Plasma HIV-1 RNA < 50 c/mL by Visit - Observed Case Analysis | Adjust the footnote as appropriate. The non-<br>snapshot visit window will be used. For W24, add<br>'(Up to Week 24)' to the title, only display visits up to<br>Week 24. | IW24, W24 |
| 2.11 | 2.11 | Intent-to-<br>Treat<br>Exposed | 201584/idmc_03/T2.11 | Proportion of Subjects with<br>Plasma HIV-1 RNA <50 c/mL by<br>Visit and Randomization Strata -<br>Observed Case Analysis | Adjust footnote and row labels as appropriate. The non-snapshot visit window and rederived randomization strata will be used. For W24, add '(Up to Week 24)' to the title, only display visits up to Week 24. | IW24, W24 |
# 15.14.4.3. Efficacy Figures

| Efficacy | Efficacy Figures | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 2.1 | 2.1 | Week 24<br>Futility | 201584/idmc_03/F2.1 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit for Subjects Who are in the Category of 'Viral Load ≥50 c/mL' at Week 24 per Snapshot Algorithm | Adjust the x-axis label and footnote as appropriate. The x-values are based on study day of the assessment. | IW24, W24 |
| 2.2 | 2.2 | Intent-to-Treat<br>Exposed | 201584/idmc_03/F2.2 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit for Subjects with a Viral Load ≥50 c/mL during the Maintenance Phase | Adjust the x-axis label and footnote as appropriate. The x-values are based on study day of the assessment. | IW24, W24 |

# 15.14.4.4. Safety Tables

| Safety T | Tables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| Adverse | Adverse Events | | | | | |
| 3.1 | 3.1 | Safety | AE3 | Summary of All Adverse Events by Overall Frequency - Maintenance Phase | See also in 201585/primary_02/T3.20. | IW24, W24 |
| 3.2 | 3.2 | Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class - Maintenance Phase | See also in 201585/primary_02/T3.16. | IW24, W24 |
| 3.3 | 3.3 | Safety | AE3 | Summary of Grade 3-5 Adverse Events by Overall Frequency - Maintenance Phase | See also in 201585/primary_02/T3.20. | IW24, W24 |
| Serious | and Othe | er Significant A | Adverse Events | | | |
| 3.4 | 3.4 | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class - Maintenance Phase | See also in 201585/primary_02/T3.21. | IW24, W24 |
| 3.5 | 3.5 | Safety | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by System Organ Class - Maintenance Phase | See also in 201585/primary_02/T3.31. | IW24, W24 |
| Injection | n Site Rea | action Advers | e Events | | | |
| 3.6 | 3.6 | Safety | 201585/primary_02/T3.<br>40 | Summary of Injection Site Reaction Adverse Events (Event-Level Summary) - Maintenance Phase | For W24, add 'Study Drug' before 'Injection' in the title and only summarize ISR from study drug injections. | IW24, W24 |

| Safety T | Safety Tables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 3.7 | 3.7 | Safety | 201585/primary_02/T3.<br>43 | Summary of Subject-Level Characteristics of Injection<br>Site Reaction Adverse Events - Overall and Common<br>(Maintenance Phase) | Common ISR adverse events includes injection site pain, injection site induration, injection site nodules and any other ISR with ≥5% subjects in either treatment arm. For W24, add 'Study Drug' before 'Injection' in the title and only summarize ISR from study drug injections. | IW24, W24 |
| Laborat | ory: Che | mistry and He | matology | | | |
| 3.8 | 3.8 | Safety | 201584/idmc_03/T3.8 | Summary of Maximum Post-Baseline Emergent<br>Clinical Chemistry Toxicities Parameters of Special<br>Interest - Maintenance Phase | Replace "Day 1" with "Study Day 1" in the first footnote. Use the same parameter list as the one in 201584/idmc_03/T3.8. | IW24, W24 |
| 3.9 | 3.9 | Safety | 201584/idmc_03/T3.9 | Summary of Maximum Post-Baseline Emergent<br>Hematology Toxicities Parameters of Special Interest -<br>Maintenance Phase | Replace "Day 1" with "Study Day 1" in the first footnote. Adjust the second footnote to be: "Note: Parameters of Special Interest include Hemogoblin, Leukocytes, Neutrophils, and Platelets." In output, change the parameter label 'White Blood Cell count' to 'Leukocytes'. | IW24, W24 |

# 15.14.4.5. Safety Figures

| Safety F | Safety Figures | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Laborat | Laboratory: Hepatobiliary (Liver) | | | | | |
| 3.1 | 3.1 | Safety | 201584/idmc_<br>03/F3.2 | Scatter Plot of Maximum Maintenance Phase vs. Baseline for ALT | Adjust the legend as needed. Change the first footnote to "Axes are on a log10 scale". Remove the second footnote. Adjust the treatment label from empty triangle to solid triangle. | IW24, W24 |
| 3.2 | 3.2 | Safety | 201584/idmc_<br>03/F3.1 | Matrix Plot of Maximum Liver Chemistries - Maintenance<br>Phase | Replace ">5.1" with ">5.0" in the second footnote. Make treatment labels in the plot consistent across figures. | IW24, W24 |

# 15.14.4.6. Pharmacokinetic Tables

| Pharma | Pharmacokinetic Tables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example Shell | Title | Programming Notes | Deliverable |
| 4.1 | 4.1 | Pharmacokinetic | 201585/primary_02/T4.1 | Summary of Plasma CAB PK Concentrations (ug/mL) - Time Data by Treatment and Visit - Including Log-Transformed Statistics | Remove the first footnote "Note:". | IW24, W24 |
| 4.2 | 4.2 | Pharmacokinetic | 201585/primary_02/T4.2 | Summary of Plasma RPV PK Concentrations (ng/mL) - Time Data by Treatment and Visit - Including Log-Transformed Statistics | Remove the first footnote "Note:" | IW24, W24 |
| 4.3 | NA | Pharmacokinetic | 201584/idmc_03/T4.3 | Proportion of Subjects with Evaluable PK<br>Concentration below Expected Values | | IW24 |

# 15.14.4.7. Pharmacokinetic Figures

| Pharmacokinetic Figures | | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 4.1 | NA | Pharmacokinetic | 201584/idmc_03/<br>F4.1 | Scatter Plot of Evaluable PK Concentrations in Relation to Occurrence of CVF up to Week 16 for Subjects on Q8W Arm by Visit and Randomization Strata | Note that this plot is by visit and rederived randomization strata. Add footnote for strata as appropriate. | IW24 |

# 15.14.4.8. Virology Tables

| Virology | Virology Tables | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 7.1 | 7.1 | Confirmed<br>Virologic Failure | 201585/primary<br>_02/T8.1 | Summary of the Prevalence of Known INI Resistance<br>Mutations at Time of CVF (Maintenance Phase) -<br>Plasma Sample | | IW24, W24 |
| 7.2 | 7.2 | Confirmed<br>Virologic Failure | 201585/primary<br>_02/T8.2 | Summary of the Prevalence of Major Resistance<br>Mutations of NNRTI, NRTI, and PI Class at Time of CVF<br>(Maintenance Phase) - Plasma Sample | | IW24, W24 |
| 7.3 | 7.3 | Confirmed<br>Virologic Failure | 201585/primary<br>_02/T8.3 | Summary of Phenotypic Susceptibility at Time of CVF (Maintenance Phase) - Plasma Sample | | IW24, W24 |
| 7.4 | 7.4 | Confirmed<br>Virologic Failure | 201585/primary<br>_02/T8.7 | Summary of Fold Change to CAB and RPV at Time of CVF (Maintenance Phase) - Plasma Sample | | IW24, W24 |
| 7.5 | 7.5 | Confirmed<br>Virologic Failure | 201585/primary<br>_02/T8.8 | Summary of Viral Load, Genotypic and Phenotypic Data for Subjects Who Met Confirmed Virologic Failure Criteria during the Maintenance Phase | Remove the Columns 'ARTs' and 'FC for ARTs'. Remove the footnotes [1] and [2]. Adjust the footnote as appropriate. | IW24, W24 |

# 15.14.4.9. ICH Listings

Note: Both unique subject ID and latest subject ID for a subject will be included in the listings, unless otherwise specified.

| ICH List | ings | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Study P | Study Population | | | | | |
| 1 | 1 | Randomized | 201584/idmc_03/L1.<br>3 | Listing of Randomized and Actual Strata and Treatment Assignment | Randomized and Actual Treatments will include oral lead-in information (e.g. Oral followed by Q4W). For W24 analyses, remove column for Futility Population. | IW24, W24 |
| Efficacy | | | | | | |
| 2 | 2 | Week 24 Futility | 201585/primary_02/L<br>11 | Listing of Study Outcomes (50 c/mL<br>Threshold) at Week 24 - Snapshot Analysis | | IW24, W24 |
| Adverse | Events | | | | | |
| 3 | 3 | Safety | 201585/primary_02/L<br>17 | Listing of Adverse Events Leading to<br>Withdrawal/Permanent Discontinuation of<br>Investigational Product - Maintenance Phase | Remove "Time Since Last Dose" from the column header. | IW24, W24 |
| 4 | 4 | Safety | 201585/primary_02/L<br>17 | Listing of All Serious Adverse Events -<br>Maintenance Phase | Remove "Time Since Last Dose" from the column header. | IW24, W24 |
| Laborate | ory | | | | | |
| 5 | NA | Safety | 201584/idmc_03/L3.<br>5 | Listing of All Parameters of Special Interest<br>Laboratory Data for Subjects with Grade 3 or<br>4 Maintenance Phase Emergent Toxicities<br>for Parameters of Special Interest | Replace 'Day 1' with 'Study Day 1' in the second footnote. | IW24 |

| ICH List | ICH Listings | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| PK | PK | | | | | |
| 6 | 5 | Pharmacokinetic | 201584/idmc_03/L4.<br>1 | Listing of Plasma CAB PK Concentration-<br>Time Data | Change the first footnote to "Relative Time is calculated relative to the date and time of last previous dose. If the time of the last previous dose (e.g. oral lead-in/oral-bridging) is missing, then the relative time will be set to missing and the sample will not be considered 'evaluable'." Remove the second footnote. Change column header 'Visit' to 'Analysis Visit/Nominal Visit' to include both visits. | IW24, W24 |
| 7 | 6 | Pharmacokinetic | 201584/idmc_03/L4.<br>2 | Listing of Plasma RPV PK Concentration-<br>Time Data | Change the first footnote to "Relative Time is calculated relative to the date and time of last previous dose. If the time of the last previous dose (e.g. oral lead-in/oral-bridging) is missing, then the relative time will be set to missing and the sample will not be considered 'evaluable'." Remove the second footnote. Change column header 'Visit' to 'Analysis Visit/Nominal Visit' to include both visits. | IW24, W24 |

# 15.14.4.10. Non-ICH Listings

**Note:** Both unique subject ID and latest subject ID for a subject will be included in the listings, unless otherwise specified.

| Non-ICH | Non-ICH Listings | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Study P | Study Population | | | | | |
| 8 | 7 | Intent-to-Treat<br>Exposed | ES2 | Listing of Reasons for Maintenance Phase Withdrawal | See also in 201585/primary_02/L30. | IW24, W24 |
| 9 | 8 | Screened | Shell POP_L2 | Listing of Subjects Who Were Rescreened | | IW24, W24 |
| 10 | 9 | Intent-to-Treat<br>Exposed | 201584/idmc_0<br>3/L1.1 | Listing of Prior Antiretroviral Therapy | Remove the column 'Treatment Phase/Treatment State'. Add a column for Route. | IW24, W24 |
| 11 | 10 | Intent-to-Treat<br>Exposed | 201584/idmc_0<br>3/L1.2 | Listing of Concomitant Antiretroviral Therapy | Change column 'Treatment Phase/Actual Treatment State' to 'Phase during Which Concomitant', remove 'Induction Study Day' from column headers, and remove 'Maintenance' from 'Maintenance Study Day' in column headers. | IW24, W24 |
| Efficacy | ' | | | | | |
| 12 | 11 | Confirmed Virologic<br>Failure | 201585/primary<br>_02/L40 | Listing of All Plasma HIV-1 RNA Viral Load<br>Data for Subjects with Confirmed Virologic<br>Failure during the Maintenance Phase | Non-snapshot visit window will be used for deriving the visits in Column 'Actual Relative Time'. Replace 'Period' in column header with 'Phase'. | IW24, W24 |

| Non-ICH | Non-ICH Listings | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 13 | 12 | Week 24 Futility | 201585/primary<br>_02/L40 | Listing of All Plasma HIV-1 RNA Viral Load Data for Subjects Who are in the Category of 'Viral load ≥50 c/mL' at Week 24 per Snapshot Algorithm | Non-snapshot visit window will be used for deriving the visits in Column 'Actual Relative Time'. Replace 'Period' in column header with 'Phase'. | IW24, W24 |
| Adverse | Events | | | | | |
| 14 | 13 | Safety | 201585/primary<br>_02/L17 | Listing of All Drug-Related Adverse Events -<br>Maintenance Phase | Remove "Time Since Last Dose" from the column header. | IW24, W24 |
| 15 | 14 | Safety | 201585/primary<br>_02/L17 | Listing of All Grade 3-5 Adverse Events -<br>Maintenance Phase | Remove "Time Since Last Dose" from the column header. | IW24, W24 |
| 16 | 15 | Safety | 201585/primary<br>_02/L17 | Listing of All Adverse Events - Long-term Follow-up Phase | Remove "Time Since Last Dose" from the column header. | IW24, W24 |
| PK | | | | | | |
| 17 | NA | Pharmacokinetic | 201584/idmc_0<br>3/L4.3 | Listing of Plasma CAB PK Concentration-Time Data for Subjects with CAB Concentration <1.35 ug/mL (~8 X PAIC90) at Visits up to Week 16 | Change the first footnote to "Relative Time is calculated relative to the date and time of last previous dose. If the time of the last previous dose (e.g. oral lead-in/oral-bridging) is missing, then the relative time will be set to missing and the sample will not be considered 'evaluable'." Remove the second footnote. Change column header 'Visit' to 'Analysis Visit/Nominal Visit' to include both visits. | IW24 |

| Non-ICH | Non-ICH Listings | | | | | |
|---|---|---|---|---|---|---|
| No. in<br>IW24 | No. in<br>W24 | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 18 | NA | Pharmacokinetic | 201584/idmc_0<br>3/L4.4 | Listing of Plasma CAB PK Concentration-Time Data for Subjects with CAB Concentration <0.166 ug/mL (PAIC90) at Visits up to Week 16 | The same note as in Listing 17. | IW24 |
| 19 | NA | Pharmacokinetic | 201584/idmc_0<br>3/L4.5 | Listing of Plasma RPV PK Concentration-Time<br>Data for Subjects with RPV Concentration <12<br>ng/mL (PAIC90) at Visits up to Week 16 | The same note as in Listing 17. | IW24 |
| Virology | 1 | | | | | |
| 20 | 16 | Confirmed Virologic Failure | 201584/idmc_0<br>3/L7.1 | Listing of Genotypic Mutation Data at All Timepoints | | IW24, W24 |
| 21 | 17 | Confirmed Virologic Failure | 201584/idmc_0<br>3/L7.2 | Listing of Phenotypic Data at All Timepoints | | IW24, W24 |

# 15.14.5. List of Data Displays for Week 48/96/End-of-Study Planned Analyses

# 15.14.5.1. Study Population Tables

| Study P | opulation | n Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subject | Disposit | ion | | | | | |
| 1.1 | 1.1 | 1.1 | Randomized | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | 'No Treatment' column is not needed. | W48, W96, EOS |
| 1.2 | 1.2 | 1.2 | Screened | ES6 | Summary of Screening Status and Reasons for Screening Failures | | W48, W96, EOS |
| 1.3 | 1.3 | 1.3 | Intent-to-<br>Treat<br>Exposed | ES1 | Summary of Subject Accountability: Study Conclusion Record | | W48, W96, EOS |
| 1.4 | 1.4 | NA | Intent-to-<br>Treat<br>Exposed | ES1 | Summary of Subject Accountability: Maintenance Phase Conclusion Record | | HL, W48, W96 |
| NA | 1.5 | 1.4 | Intent-to-<br>Treat<br>Exposed | ES1 | Summary of Subject Accountability: Maintenance + Extension Phase Conclusion Record | For subject status, include 'ONGOING', 'COMPLETED MAINTENANCE PHASE', 'COMPLETED EXTENSION PHASE', 'WITHDRAWN FROM MAINTENANCE PHASE' and 'WITHDRAWN FROM EXTENSION PHASE'. | W96, EOS |
| 1.5 | 1.6 | 1.5 | Long-term<br>Follow-up | ES1 | Summary of Subject Accountability: Long-term Follow-up Phase Conclusion Record | | W48, W96, EOS |

| Study P | Study Population Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.6 | 1.7 | 1.6 | Intent-to-<br>Treat<br>Exposed | ES4 | Summary of Subject Disposition at Each Study Phase | Replace 'Epoch' with 'Phase' in column header. Screening Phase will not be included. Add a footnote "Note: Entry into Long-Term Follow-up is based on presence of a long-term follow-up visit in the eCRF (i.e. LTFU Month 1, LTFU Month 3, etc.) or evidence of filling out the long-term follow-up phase conclusion form." | W48, W96, EOS |
| 1.7 | 1.8 | 1.7 | Intent-to-<br>Treat<br>Exposed | ES5 | Summary of Reasons for Withdrawal at Each Study Phase | The same comment as above. | W48, W96, EOS |
| 1.8 | 1.9 | 1.8 | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T1.9 | Summary of Subject Accountability:<br>Withdrawals by Visit (Maintenance + Extension<br>Phase) | | W48, W96, EOS |
| 1.9 | 1.10 | 1.9 | Intent-to-<br>Treat<br>Exposed | ES1 | Summary of Study Drug Discontinuation | Update the row label to 'Primary Reason[1]/Subreason[2] for Study Drug Discontinuation'. | W48, W96, EOS |
| 1.10 | 1.11 | NA | Intent-to-<br>Treat<br>Exposed | DV1a | Summary of Important Protocol Deviations (Maintenance Phase) | | W48, W96 |
| NA | 1.12 | 1.10 | Intent-to-<br>Treat<br>Exposed | DV1a | Summary of Important Protocol Deviations (Maintenance + Extension Phase) | | W96, EOS |
| 1.11 | 1.13 | 1.11 | Intent-to-<br>Treat | IE1 | Summary of Inclusion/Exclusion Criteria | | W48, W96, EOS |

| Study P | opulation | 1 Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | Exposed | | Deviations | | |
| 1.12 | 1.14 | 1.12 | Screened | 201585/primar<br>y_02/T1.1 | Summary of Study Populations | Adjust the footnote as appropriate. | HL, W48, W96,<br>EOS |
| 1.13 | 1.15 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.14 | Summary of Protocol Deviations Leading to Exclusion from the Per-Protocol Population (through Maintenance Phase) | | W48, W96 |
| Demog | raphic an | d Baselir | e Characterist | ics | | | |
| 1.14 | 1.16 | 1.13 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.16 | Summary of Demographic Characteristics | | HL, W48, W96,<br>EOS |
| 1.15 | 1.17 | 1.14 | Randomized | DM11 | Summary of Age Ranges | Also refer to 201585/primary_02/T1.4. Follow the footnote in 201585/primary_02/T1.4. | W48, W96, EOS |
| 1.16 | 1.18 | 1.15 | Intent-to-<br>Treat<br>Exposed | DM5 | Summary of Race and Racial Combinations | | W48, W96, EOS |
| 1.17 | 1.19 | 1.16 | Intent-to-<br>Treat<br>Exposed | DM6 | Summary of Race and Racial Combinations Details | | W48, W96, EOS |
| 1.18 | 1.20 | 1.17 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.19 | Summary of Hepatitis Status at Entry | Add footnote as appropriate for subjects classified as Hepatitis B positive in analysis. | W48, W96, EOS |
| 1.19 | 1.21 | 1.18 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.20 | Summary of Derived Baseline CDC Stages of HIV Infection | | W48, W96, EOS |

| Study P | opulation | n Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.20 | 1.22 | 1.19 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.21 | Summary of Baseline Cardiovascular Risk<br>Assessments | | W48, W96, EOS |
| 1.21 | 1.23 | 1.20 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.22 | Distribution of CD4+ Cell Count Results at Screening and Baseline | | W48, W96, EOS |
| 1.22 | 1.24 | 1.21 | Intent-to-<br>Treat<br>Exposed | Shell POP_T1 | Summary of Prior Exposure to CAB+RPV | | W48, W96, EOS |
| 1.23 | 1.25 | 1.22 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.36 | Summary of HIV Risk Factors | | W48, W96, EOS |
| Medical | l Conditio | ns and N | ledications | | | | |
| 1.24 | 1.26 | 1.23 | Intent-to-<br>Treat<br>Exposed | MH1 | Summary of Current Medical Conditions | | W48, W96, EOS |
| 1.25 | 1.27 | 1.24 | Intent-to-<br>Treat<br>Exposed | MH1 | Summary of Past Medical Conditions | | W48, W96, EOS |
| 1.26 | 1.28 | 1.25 | Intent-to-<br>Treat<br>Exposed | MH4 | Summary of Current Cardiac, Gastrointestinal,<br>Metabolism and Nutrition, Psychiatric, Renal<br>and Urinary, Nervous System Conditions, and<br>Hepatobiliary Disorders | | W48, W96, EOS |
| 1.27 | 1.29 | 1.26 | Intent-to-<br>Treat<br>Exposed | MH4 | Summary of Past Cardiac, Gastrointestinal,<br>Metabolism and Nutrition, Psychiatric, Renal<br>and Urinary, Nervous System Conditions, and<br>Hepatobiliary Disorders | | W48, W96, EOS |

| Study P | opulation | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.28 | 1.30 | 1.27 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.28 | Summary of Prior ART Medications | Remove the footnote. Follow definitions in Section 6.2 to determine the prior ART medications. | W48, W96, EOS |
| 1.29 | 1.31 | NA | Intent-to-<br>Treat<br>Exposed | CM8 | Summary of Concomitant Non-ART Medication Ingredient Combinations (Maintenance Phase) | | W48, W96 |
| NA | 1.32 | 1.28 | Intent-to-<br>Treat<br>Exposed | CM8 | Summary of Concomitant Non-ART Medication Ingredient Combinations (Maintenance + Extension Phase) | | W96, EOS |
| 1.30 | 1.33 | 1.29 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.33 | Summary of Lipid Modifying Agent Use at Baseline | | W48, W96, EOS |
| 1.31 | 1.34 | 1.30 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.34 | Summary of Lipid Modifying Agent Use Started during the Maintenance Phase | | W48, W96, EOS |
| 1.32 | 1.35 | 1.31 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T1.35 | Summary of Substance Use at Entry | | W48, W96, EOS |

# 15.14.5.2. Efficacy Tables

**Note:** For subgroup analyses, include rederived randomization strata (i.e. prior exposure to CAB+RPV: 0, 1-24, >24 weeks), all demographic and baseline characteristic subgroups as mentioned in EMA Subgroup Category 2 in Section 5.4.2, unless otherwise specified. Not all subjects on Q8W arm are planned to have viral load data collected at Week 4 (Week 4A or 4B), so leave Week 4 data blank for Q8W arm in by-visit snapshot analysis.

| Efficacy | Efficacy Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Primary | Primary Efficacy Analyses | | | | | | |
| 2.1 | 2.1 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.1 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 48 (Maintenance Phase) – Snapshot Analysis – ITT-E | Adjust the footnotes as appropriate. For WK96, replace 'Week 48' with 'Week 96' in title. | HL, W48, W96 |
| 2.2 | 2.2 | NA | Per-<br>Protocol | 201584/primar<br>y_01/T2.2 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 48 (Maintenance Phase) – Snapshot Analysis – Per-Protocol | Adjust the footnotes as appropriate. For WK96, replace 'Week 48' with 'Week 96' in title. | HL, W48, W96 |
| 2.3 | 2.3 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.3 | Summary of Study Outcomes (50 c/mL Threshold) at Week 48 (Maintenance Phase) – Snapshot Analysis | For WK96, replace 'Week 48' with 'Week 96' in title. | HL, W48, W96 |
| 2.4 | 2.4 | NA | Intent-to-<br>Treat<br>Exposed | Shell EFF_T3 | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 48 (Maintenance Phase) - Snapshot Analysis | For WK96, replace 'Week 48' with 'Week 96' in title. | HL, W48, W96 |

| Efficacy | Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.5 | 2.5 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.5 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 48 by Subgroup (Maintenance Phase) - Snapshot Analysis | Adjust the footnote/column header label as appropriate. For WK96, replace 'Week 48' with 'Week 96' in title. Do not include rederived randomization strata in the table. | W48, W96 |
| 2.6 | 2.6 | NA | Intent-to-<br>Treat<br>Exposed | Shell EFF_T4 | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 48 among Subjects with >=1 Weeks Prior Exposure to CAB+RPV (Maintenance Phase) - Snapshot Analysis | For WK96, replace 'Week 48' with 'Week 96' in title. | W48, W96 |
| 2.7 | 2.7 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.6 | Summary of Study Outcomes (50 c/mL Threshold) at Week 48 by Subgroup (Maintenance Phase) – Snapshot Analysis | For WK96, replace 'Week 48' with 'Week 96' in title. | W48, W96 |
| Seconda | ary and E | xplorato | ry Efficacy An | alyses | | | |
| 2.8 | 2.8 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.7 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 (Maintenance Phase) – Snapshot Analysis – ITT-E | Adjust the footnotes as appropriate. For WK96, replace 'Week 48' with 'Week 96' in title. | HL, W48, W96 |
| 2.9 | 2.9 | NA | Per-<br>Protocol | 201584/primar<br>y_01/T2.8 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 (Maintenance Phase) – Snapshot Analysis – Per-Protocol | Adjust the footnotes as appropriate. For WK96, replace 'Week 48' with 'Week 96' in title. | HL, W48, W96 |

| Efficacy | Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.10 | 2.10 | NA | Intent-to-<br>Treat<br>Exposed | Shell EFF_T3 | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 (Maintenance Phase) - Snapshot Analysis | Replace 'Number of HIV-1<br>RNA >=50 c/mL' with 'Number<br>of HIV-1 RNA <50 c/mL' in<br>column header. For WK96,<br>replace 'Week 48' with 'Week<br>96' in title. | HL, W48, W96 |
| 2.11 | 2.11 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.10 | Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL at Week 48 by Subgroup (Maintenance Phase) - Snapshot Analysis | Adjust the footnote/column header label as appropriate. For WK96, replace 'Week 48' with 'Week 96' in title. Do not include rederived randomization strata in the table. | W48, W96 |
| 2.12 | 2.12 | NA | Intent-to-<br>Treat<br>Exposed | Shell EFF_T4 | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Week 48 among Subjects with >=1 Weeks Prior Exposure to CAB+RPV (Maintenance Phase) - Snapshot Analysis | Replace 'Number of HIV-1<br>RNA >=50 c/mL' with 'Number<br>of HIV-1 RNA <50 c/mL' in<br>column header. For WK96,<br>replace 'Week 48' with 'Week<br>96' in title. | W48, W96 |
| 2.13 | 2.13 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.11 | Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.14 | 2.14 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.12 | Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL by Subgroup and Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.15 | 2.15 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.15 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |

| Efficacy | Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.16 | 2.16 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.16 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Subgroup and Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.17 | 2.17 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.17 | Proportion of Subjects with Plasma HIV-1 RNA <200 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.18 | 2.18 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.17 | Proportion of Subjects with Plasma HIV-1 RNA >=200 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | Adjust column headers as appropriate. Keep one decimal place for proportion. | W48, W96 |
| 2.19 | 2.19 | NA | Intent-to-<br>Treat<br>Exposed | Shell EFF_T1 | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Failure at Week 48 - Treatment Related Discontinuation = Failure | Adjust the row labels and footnotes as appropriate. For WK96, replace 'Week 48' with 'Week96' in title. | W48, W96 |
| 2.20 | 2.20 | NA | Intent-to-<br>Treat<br>Exposed | Shell EFF_T2 | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Failure at Week 48 - Efficacy Related Discontinuation = Failure | Adjust the row labels and footnotes as appropriate. For WK96, replace 'Week 48' with 'Week96' in title. | W48, W96 |
| 2.21 | 2.21 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.19 | Proportion of Subjects with HIV-1 RNA >=50 c/mL at Week 48 (Snapshot) by Last Delay in IP Injection (Maintenance Phase) | Display both arms. Change the footnote to 'The last delay in IP injection will be the delay in IP injection at Week 48, or the delay in last IP injection prior to Week 48 if a participant did not receive Week 48 injection (i.e. missing visit or withdrawal)'. For WK96, replace 'Week 48' with 'Week96' in title. | W48, W96 |

| Efficacy | Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.22 | 2.22 | 2.1 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.20 | Summary of Plasma HIV-1 RNA (log10 c/mL) by Visit | | W48, W96,<br>EOS |
| 2.23 | 2.23 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.21 | Cumulative Proportion of Subjects Meeting<br>Confirmed Virology Failure Criteria by Visit during the<br>Maintenance Phase (Up to Week 48) | For WK96, replace 'Up to Week 48' with 'Up to Week 96' in title. | HL, W48, W96 |
| 2.24 | 2.24 | 2.2 | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.21 | Cumulative Proportion of Subjects Meeting<br>Confirmed Virology Failure Criteria (Maintenance +<br>Extension Phase) | | W48, W96,<br>EOS |
| 2.25 | 2.25 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.24 | Distribution of Quantitative Plasma HIV-1 RNA Results at Suspected and Confirmation of Confirmed Virologic Failure (Maintenance Phase) | | W48, W96 |
| 2.26 | 2.26 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.34 | Proportion of Subjects with Plasma HIV-1 RNA <2 c/mL by Visit (Maintenance Phase) | Change footnote to 'Note:<br>Data come from BioMontr low-<br>level assay. Only visits with<br>available data from this assay<br>are included.' | W48, W96 |
| 2.27 | 2.27 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.51 | Summary of Study Outcomes (200 c/mL Threshold) at Week 48 (Maintenance Phase) – Snapshot Analysis | For WK96, replace 'Week 48' with 'Week 96' in title. | W48, W96 |
| 2.28 | 2.28 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.37 | Summary of Subjects per Viral Load Category by Visit (Maintenance Phase) | Refer to 'Summary for Participants per Viral Load Category by Visit' in Section 15.6.3. Remove footnote [2]. Add a footnote "Note: The visit windows are based on snapshot analysis windows'. | W48, W96 |

| Efficacy | Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.29 | 2.29 | 2.3 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.25 | Summary of Change from Baseline in CD4+ Cell<br>Count (cells/mm^3) by Visit (Maintenance +<br>Extension Phase) | | W48, W96,<br>EOS |
| 2.30 | 2.30 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.38 | Summary of Change from Baseline in CD4+ Cell<br>Count (cells/mm^3) at Week 48 by Subgroup<br>(Maintenance Phase) | For WK96, replace 'Week 48' with 'Week 96' in title. | W48, W96 |
| 2.31 | 2.31 | 2.4 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.26 | Summary of CD4+ Cell Count (cells/mm^3) by Visit (Maintenance + Extension Phase) | | W48, W96,<br>EOS |
| 2.32 | 2.32 | 2.5 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.28 | Summary of Change from Baseline in CD8+ Cell<br>Count (cells/mm^3) by Visit (Maintenance +<br>Extension Phase) | | W48, W96,<br>EOS |
| 2.33 | 2.33 | 2.6 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.27 | Summary of CD8+ Cell Count (cells/mm^3) by Visit (Maintenance + Extension Phase) | | W48, W96,<br>EOS |
| 2.34 | 2.34 | 2.7 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.29 | Summary of CD4+/CD8+ Ratio Cell Count (cells/mm^3) by Visit (Maintenance + Extension Phase) | Ratio will be taken when both CD4+ and CD8+ are available on the same date. | W48, W96,<br>EOS |
| 2.35 | 2.35 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.30 | Summary of HIV-1 Associated Conditions Including Recurrences (Maintenance Phase) | | W48, W96 |
| NA | 2.36 | 2.8 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.30 | Summary of HIV-1 Associated Conditions Including Recurrences (Maintenance +Extension Phase) | | W96, EOS |
| 2.36 | 2.37 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.31 | Summary of HIV-1 Associated Conditions Excluding Recurrences (Maintenance Phase) | | W48, W96 |

| Efficacy | Efficacy Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| NA | 2.38 | 2.9 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T2.31 | Summary of HIV-1 Associated Conditions Excluding Recurrences (Maintenance +Extension Phase) | | W96, EOS |
| 2.37 | 2.39 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.47 | Summary of HIV-1 Disease Progression and/or Deaths (Maintenance Phase) | | W48, W96 |
| NA | 2.40 | 2.10 | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/T2.47 | Summary of HIV-1 Disease Progression and/or Deaths (Maintenance + Extension Phase) | | W96, EOS |

# 15.14.5.3. Efficacy Figures

**Note:** For subgroup analyses, include rederived randomization strata (i.e. prior exposure to CAB+RPV: 0, 1-24, >24 weeks), all demographic and baseline characteristic subgroups as mentioned in EMA Subgroup Category 2 in Section 5.4.2, unless otherwise specified. Not all subjects on Q8W arm are planned to have viral load data collected at Week 4 (Week 4A or 4B), so leave Week 4 data blank for Q8W arm in by-visit snapshot analysis.

| Efficacy | / Figures | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Primary | Efficacy | Analyses | | | | | |
| 2.1 | 2.1 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F2.1 | Proportion (95% CI) of Subjects with HIV-1 RNA<br>≥50 c/mL by Visit (Maintenance Phase) – Snapshot<br>Analysis | | HL, W48, W96 |
| 2.2 | 2.2 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primary<br>_01/F2.2 | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA ≥50 c/mL at Week 48 by Subgroup – Snapshot Analysis | Non-inferiority margin is 4%.<br>Adjust the footnotes,<br>reference line and labels as<br>appropriate. For WK96,<br>replace 'Week 48' with<br>'Week 96' in title. | W48, W96 |
| Second | ary and E | xploratory | Efficacy Ana | lyses | | | |
| 2.3 | 2.3 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F2.3 | Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | HL, W48, W96 |
| 2.4 | 2.4 | NA | Intent-to-<br>Treat<br>Exposed | 201584/primary<br>_01/F2.4 | Unadjusted Treatment Difference in Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL at Week 48 by Subgroup – Snapshot Analysis | Adjust the footnotes, reference line and labels as appropriate. For WK96, replace 'Week 48' with 'Week 96' in title. | W48, W96 |

| Efficacy | Figures | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.5 | 2.5 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F2.10 | Proportion (95% CI) of Subjects with HIV-1 RNA >=200 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.6 | 2.6 | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F2.5 | Proportion (95% CI) of Subjects with HIV-1 RNA <200 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | W48, W96 |
| 2.7 | 2.7 | 2.1 | Intent-to-<br>Treat<br>Exposed | 207966/idmc_0<br>3/F2.1 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit – for CVF subjects | | HL, W48, W96,<br>EOS |
| 2.8 | 2.8 | NA | Intent-to-<br>Treat<br>Exposed | 207966/idmc_0<br>3/F2.1 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit for subjects Who are in the Category of 'HIV-1 RNA >=50 c/mL' at Week 48 per Snapshot algorithm | For WK96, replace 'Week 48' with 'Week 96' in the title. | HL, W48, W96 |

# 15.14.5.4. Safety Tables

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Exposu | re | | | | | | • |
| 3.1 | 3.1 | 3.1 | Safety | 201585/primar<br>y_02/T3.1 | Summary of Extent of Exposure to Investigational Product (Maintenance Phase) | No need for the first two footnotes. Update the last footnote to be below: Note: The injection at nominal visit of Week 100 was not included in the summary of Exposure (No. of IP injections). | W48, W96,<br>EOS |
| NA | 3.2 | 3.2 | Safety | 201585/primar<br>y_02/T3.1 | Summary of Extent of Exposure to Investigational Product (Maintenance + Extension Phase) | Remove the footnotes. | W96, EOS |
| 3.2 | 3.3 | NA | Safety | 201585/primar<br>y_03/T3.102 | Summary of Needle Length and Gauge for CAB Injection (Maintenance Phase) | Display both arms. | W48, W96 |
| 3.3 | 3.4 | NA | Safety | 201585/primar<br>y_03/T3.103 | Summary of Needle Length and Gauge for RPV Injection (Maintenance Phase) | Display both arms. | W48, W96 |
| 3.4 | 3.5 | NA | Safety | 201585/primar<br>y_02/T3.6 | Summary of Adherence to CAB/RPV Injection Dosing Schedule (Maintenance Phase) | Display both arms. Adjust the footnotes as appropriate. | W48, W96 |
| Adverse | Events | | | | | | • |
| 3.5 | 3.6 | NA | Safety | 201585/primar<br>y_02/T3.7 | Summary of All Adverse Events by System Organ Class (Maintenance Phase) | | W48, W96 |
| 3.6 | 3.7 | NA | Safety | 201585/primar<br>y_02/T3.8 | Summary of All Adverse Events by System Organ Class and Maximum Toxicity (Maintenance Phase) | | HL, W48,<br>W96 |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| NA | 3.8 | 3.3 | Safety | 201585/primar<br>y_02/T3.8 | Summary of All Adverse Events by System Organ Class and Maximum Toxicity (Maintenance + Extension Phase) | | W96, EOS |
| 3.7 | 3.9 | NA | Safety | 201585/primar<br>y_02/T3.8 | Summary of All Adverse Events Excluding<br>Study Drug Injection Site Reactions by<br>System Organ Class and Maximum Toxicity<br>(Maintenance Phase) | | HL, W48,<br>W96 |
| NA | NA | 3.4 | Long-term<br>Follow-up | 201585/primar<br>y_02/T3.8 | Summary of All Adverse Events by System Organ Class and Maximum Toxicity (Longterm Follow-up Phase) | | EOS |
| 3.8 | 3.10 | NA | Safety | 201585/primar<br>y_02/T3.11 | Summary of All On-treatment Adverse<br>Events by System Organ Class and<br>Maximum Toxicity (Maintenance Phase) | | W48, W96 |
| 3.9 | NA | NA | Oral Lead-<br>in | 201585/primar<br>y_02/T3.13 | Summary of All Adverse Events by System Organ Class and Maximum Toxicity (Oral Lead-in Period during the Maintenance Phase) | Remove the footnote. Display both arms. | W48 |
| 3.10 | 3.11 | NA | Safety | 201585/primar<br>y_02/T3.14 | Summary of Common Adverse Events (>=5%) by Overall Frequency (Maintenance Phase) | | W48, W96 |
| 3.11 | 3.12 | NA | Safety | 201585/primar<br>y_02/T3.15 | Summary of Common Grade 2-5 Adverse<br>Events (>=1%) by Overall Frequency<br>(Maintenance Phase) | | W48, W96 |
| 3.12 | 3.13 | NA | Safety | 201585/primar<br>y_02/T3.16 | Summary of All Drug-related Adverse<br>Events by System Organ Class<br>(Maintenance Phase) | | W48, W96 |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.13 | 3.14 | NA | Safety | 201585/primar<br>y_02/T3.17 | Summary of All Drug-related Adverse<br>Events by System Organ Class and<br>Maximum Toxicity (Maintenance Phase) | | HL, W48,<br>W96 |
| NA | 3.15 | 3.5 | Safety | 201585/primar<br>y_02/T3.17 | Summary of All Drug-related Adverse Events by System Organ Class and Maximum Toxicity (Maintenance + Extension Phase) | | W96, EOS |
| 3.14 | 3.16 | NA | Safety | 201585/primar<br>y_02/T3.101 | Summary of All Drug-related Adverse<br>Events Excluding Study Drug Injection Site<br>Reactions by System Organ Class and<br>Maximum Toxicity (Maintenance Phase) | | HL, W48,<br>W96 |
| 3.15 | 3.17 | NA | Safety | 201585/primar<br>y_02/T3.20 | Summary of All Drug-Related Grade 2-5<br>Adverse Events by Overall Frequency<br>(Maintenance Phase) | | W48, W96 |
| Serious | and Other | r Significa | ant Adverse Ev | vents | | | |
| 3.16 | 3.18 | NA | Safety | 201585/primar<br>y_02/T3.21 | Summary of Serious Adverse Events by<br>System Organ Class (Maintenance Phase) | | HL, W48,<br>W96 |
| NA | 3.19 | 3.6 | Safety | 201585/primar<br>y_02/T3.21 | Summary of Serious Adverse Events by<br>System Organ Class (Maintenance +<br>Extension Phase) | | W96, EOS |
| 3.17 | 3.20 | 3.7 | Long-term<br>Follow-up | 201585/primar<br>y_02/T3.24 | Summary of Serious Adverse Events by<br>System Organ Class (Long-term Follow-up<br>Phase) | | W48, W96,<br>EOS |
| 3.18 | NA | NA | Oral Lead-<br>in | 201585/primar<br>y_02/T3.25 | Summary of Serious Adverse Events by<br>System Organ Class (Oral Lead-in Period<br>during the Maintenance Phase) | Display both arms. | W48 |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.19 | 3.21 | NA | Safety | 201585/primar<br>y_02/T3.26 | Summary of Drug-related Serious Adverse<br>Events by System Organ Class<br>(Maintenance Phase) | | W48, W96 |
| NA | 3.22 | 3.8 | Safety | 201585/primar<br>y_02/T3.26 | Summary of Drug-related Serious Adverse<br>Events by System Organ Class<br>(Maintenance + Extension Phase) | | W96, EOS |
| 3.20 | 3.23 | NA | Safety | 201585/primar<br>y_02/T3.29 | Summary of Non-Fatal Serious Adverse<br>Events by Overall Frequency (Maintenance<br>Phase) | | W48, W96 |
| 3.21 | 3.24 | NA | Safety | 201585/primar<br>y_02/T3.30 | Summary of Drug-related Non-Fatal Serious<br>Adverse Events by Overall Frequency<br>(Maintenance Phase) | | W48, W96 |
| 3.22 | 3.25 | NA | Safety | 201585/primar<br>y_02/T3.31 | Summary of Adverse Events Leading to<br>Withdrawal/Permanent Discontinuation of<br>Investigational Product by System Organ<br>Class (Maintenance Phase) | | HL, W48,<br>W96 |
| NA | 3.26 | 3.9 | Safety | 201585/primar<br>y_02/T3.31 | Summary of Adverse Events Leading to<br>Withdrawal/Permanent Discontinuation of<br>Investigational Product by System Organ<br>Class (Maintenance + Extension Phase) | | W96, EOS |
| 3.23 | NA | NA | Oral Lead-<br>in | 201585/primar<br>y_02/T3.34 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by System Organ Class (Oral Lead-in Period during the Maintenance Phase) | Remove the footnote. Display both arms. | W48 |
| 3.24 | 3.27 | NA | Safety | 201585/primar<br>y_02/T3.35 | Summary of Common (>=5%) Non-Serious Adverse Events (Maintenance Phase) | | W48, W96 |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.25 | 3.28 | NA | Safety | 201585/primar<br>y_02/T3.36 | Summary of Subjects and Number of<br>Occurrences of Common (>=5%) Non-<br>Serious Adverse Events by System Organ<br>Class (Maintenance Phase) | | W48, W96 |
| 3.26 | 3.29 | NA | Safety | 201585/primar<br>y_02/T3.37 | Summary of Subjects and Number of occurrences of SAEs, Fatal SAEs, and Drug-related SAEs (Maintenance Phase) | | W48, W96 |
| 3.27 | 3.30 | NA | Safety | 201585/primar<br>y_02/T3.38 | Summary of Cumulative Adverse Events by Visit (Maintenance Phase) | Note that this table only display AEs occurring >=5% subjects during Maintenance Phase. | W48, W96 |
| Study D | rug Injecti | ion Site R | eaction Adver | se Events (displa | y for both arms) | | |
| 3.28 | 3.31 | NA | Safety | 201585/primar<br>y_02/T3.40 | Summary of Study Drug Injection Site<br>Reaction Adverse Events (Event-level<br>Summary) - Maintenance Phase | | HL, W48,<br>W96 |
| NA | 3.32 | 3.10 | Safety | 201585/primar<br>y_02/T3.40 | Summary of Study Drug Injection Site<br>Reaction Adverse Events (Event-level<br>Summary) - Maintenance + Extension<br>Phase | | W96, EOS |
| 3.29 | 3.33 | NA | Safety | 201585/primar<br>y_02/T3.43 | Summary of Subject-level Characteristics of<br>Study Drug Injection Site Reaction Adverse<br>Events – Overall and Common<br>(Maintenance Phase) | | W48, W96 |
| NA | 3.34 | 3.11 | Safety | 201585/primar<br>y_02/T3.43 | Summary of Subject-level Characteristics of<br>Study Drug Injection Site Reaction Adverse<br>Events – Overall and Common<br>(Maintenance + Extension Phase) | | W96, EOS |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.30 | 3.35 | NA | Safety | 201585/primar<br>y_02/T3.46 | Summary of Study Drug Injection Site<br>Reaction Adverse Events by Visit and<br>Maximum Severity – Overall and Common<br>(Maintenance Phase) | Change the second footnote to 'Note: Common ISR includes pain, induration, nodules and any other ISR with >=5% subjects in either treatment arm.' Footnote may be adjusted for clarifications. | W48, W96 |
| 3.31 | 3.36 | NA | Safety | 201585/primar<br>y_02/T3.47 | Summary of Drug-related Study Drug<br>Injection Site Reaction Adverse Events<br>(Event-level Summary) - CAB (Maintenance<br>Phase) | | W48, W96 |
| 3.32 | 3.37 | NA | Safety | 201585/primar<br>y_02/T3.48 | Summary of Drug-related Subject-level<br>Characteristics of Study Drug Injection Site<br>Reaction Adverse Events (Maintenance<br>Phase) - Overall and Common (CAB) | | W48, W96 |
| 3.33 | 3.38 | NA | Safety | 201585/primar<br>y_02/T3.49 | Summary of Overall and Common Drug-<br>related Study Drug Injection Site Reaction<br>Adverse Events by Visit and Maximum<br>Severity (Maintenance Phase) - CAB | Footnote may be adjusted for clarifications. | W48, W96 |
| 3.34 | 3.39 | NA | Safety | 201585/primar<br>y_02/T3.50 | Summary of Maximum Drug-related Study<br>Drug Injection Site Reaction Adverse Event<br>Grade by Needle Length (Maintenance<br>Phase) – Common (CAB) | Update the needle length in column header to be "<=1.5 inches', '>1.5 to <2 inches' and '>=2 inches' respectively. Change the first footnote to 'Note: Common ISR includes pain, induration, nodules and any other ISR with >=5% subjects in either treatment arm.'. Remove the second footnote. | W48, W96 |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.35 | 3.40 | NA | Safety | 201585/primar<br>y_02/T3.51 | Summary of Drug-related Study Drug<br>Injection Site Reaction Adverse Events<br>(Event-level Summary) - RPV (Maintenance<br>Phase) | | W48, W96 |
| 3.36 | 3.41 | NA | Safety | 201585/primar<br>y_02/T3.52 | Summary of Drug-related Subject-level<br>Characteristics of Study Drug Injection Site<br>Reaction Adverse Events (Maintenance<br>Phase) - Overall and Common (RPV) | | W48, W96 |
| 3.37 | 3.42 | NA | Safety | 201585/primar<br>y_02/T3.53 | Summary of Overall and Common Drug-<br>related Study Drug Injection Site Reaction<br>Adverse Events by Visit and Maximum<br>Severity (Maintenance Phase) - RPV | Footnote may be adjusted for clarifications. | W48, W96 |
| 3.38 | 3.43 | NA | Safety | 201585/primar<br>y_02/T3.54 | Summary of Maximum Drug-related Study<br>Drug Injection Site Reaction Adverse Event<br>Grade by Needle Length (Maintenance<br>Phase) – Common (RPV) | Update the needle length in column header to be "<=1.5 inches', '>1.5 to < 2 inches' and '>=2 inches' respectively. Change the first footnote to 'Note: Common ISR includes pain, induration, nodules and any other ISR with >=5% subjects in either treatment arm.'. Remove the second footnote. | W48, W96 |
| Laborate | ory: Chem | istry and | Hematology | | | | |
| 3.39 | 3.44 | 3.12 | Safety | 201585/primar<br>y_02/T3.55 | Summary of Chemistry Changes from<br>Baseline by Visit (Maintenance + Extension<br>Phase) | Present GFR, lipids and glucose in both conventional and standard units. Change 'Post Baseline' to 'Postbaseline' in the footnote. | W48, W96,<br>EOS |
| 3.40 | 3.45 | 3.13 | Safety | 201585/primar<br>y_02/T3.59 | Summary of Chemistry Values by Visit (Maintenance + Extension Phase) | Present GFR, lipids and glucose in both conventional and standard units. Change 'Post Baseline' to 'Post- | W48, W96,<br>EOS |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| | | | | | | baseline' in the footnote. | |
| 3.41 | 3.46 | 3.14 | Safety | 201585/primar<br>y_02/T3.60 | Summary of Hematology Changes from Baseline by Visit (Maintenance + Extension Phase) | Change 'Post Baseline' to 'Post-baseline' in the footnote. | W48, W96,<br>EOS |
| 3.42 | 3.47 | 3.15 | Safety | 201585/primar<br>y_02/T3.59 | Summary of Hematology Values by Visit (Maintenance + Extension Phase) | Remove the first footnote. Change 'Post Baseline' to 'Post-baseline' in the footnote. | W48, W96,<br>EOS |
| 3.43 | 3.48 | NA | Safety | 201585/primar<br>y_02/T3.61 | Summary of Maximum Post-Baseline<br>Emergent Chemistry Toxicities<br>(Maintenance Phase) | Add "Emergent is relative to last toxicity up to and including baseline." to the end of the second footnote. | W48, W96 |
| NA | 3.49 | 3.16 | Safety | 201585/primar<br>y_02/T3.61 | Summary of Maximum Post-Baseline<br>Emergent Chemistry Toxicities<br>(Maintenance + Extension Phase) | Adjust the footnote similar to above. | W96, EOS |
| 3.44 | NA | NA | Oral Lead-<br>in | 201585/primar<br>y_02/T3.64 | Summary of Maximum Post-Baseline<br>Emergent Chemistry Toxicities - Oral Lead-<br>in Period during the Maintenance Phase | Display both arms. Adjust the footnote similarly to above. | W48 |
| 3.45 | 3.50 | NA | Safety | 201585/primar<br>y_02/T3.65 | Summary of Maximum Post-Baseline<br>Emergent Hematology Toxicities<br>(Maintenance Phase) | Adjust the footnote similarly to above. | W48, W96 |
| NA | 3.51 | 3.17 | Safety | 201585/primar<br>y_02/T3.65 | Summary of Maximum Post-Baseline<br>Emergent Hematology Toxicities<br>(Maintenance + Extension Phase) | Adjust the footnote similarly to above. | W96, EOS |
| 3.46 | NA | NA | Oral Lead-<br>in | 201585/primar<br>y_02/T3.68 | Summary of Maximum Post-Baseline Emergent Hematology Toxicities - Oral Lead-in Period during the Maintenance Phase | Display both arms. Adjust the footnote similarly to above. | W48 |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Laborat | ory: Urina | lysis | • | | | | |
| 3.47 | 3.52 | 3.18 | Safety | 201585/primar<br>y_02/T3.69 | Summary of Urinalysis Dipstick Results by Visit (Maintenance + Extension Phase) | Change 'Post Baseline' to 'Post-Baseline' in the footnote. | W48, W96,<br>EOS |
| 3.48 | 3.53 | 3.19 | Safety | 201585/primar<br>y_02/T3.70 | Summary of Urine Concentrations Changes from Baseline by Visit (Maintenance + Extension Phase) | Change 'Post Baseline' to 'Post-Baseline' in the footnote. | W48, W96,<br>EOS |
| 3.49 | 3.54 | NA | Safety | 201585/primar<br>y_02/T3.71 | Summary of Changes in Proteinuria Baseline Laboratory Result to Maximum Post-Baseline Laboratory Result (Maintenance Phase) | Change 'Post Baseline' to 'Post-Baseline' in the footnote. | W48, W96 |
| Laborat | ory: Lipid | | | | | | • |
| 3.50 | 3.55 | NA | Safety | 201585/primar<br>y_02/T3.72 | Summary of Changes in Baseline NCEP<br>Fasting Lipid Category to Maximum Post-<br>Baseline Category – Triglycerides<br>(Maintenance Phase) | | W48, W96 |
| 3.51 | 3.56 | NA | Safety | 201585/primar<br>y_02/T3.73 | Summary of Changes in Baseline NCEP<br>Fasting Lipid Category to Maximum Post-<br>Baseline Category – Total Cholesterol<br>(Maintenance Phase) | | W48, W96 |
| 3.52 | 3.57 | NA | Safety | 201585/primar<br>y_02/T3.74 | Summary of Changes in Baseline NCEP<br>Fasting Lipid Category to Minimum Post-<br>Baseline Category – HDL Cholesterol<br>(Maintenance Phase) | | W48, W96 |
| 3.53 | 3.58 | NA | Safety | 201585/primar<br>y_02/T3.75 | Summary of Changes in Baseline NCEP<br>Fasting Lipid Category to Maximum Post-<br>Baseline Category – LDL Cholesterol<br>(Maintenance Phase) | | W48, W96 |

| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.54 | 3.59 | NA | Safety | 201585/primar<br>y_02/T3.58 | Summary of Fasting Lipids Percentage<br>Changes from Baseline by Visit<br>(Maintenance Phase) - Lipids LOCF | Change 'Post Baseline' to 'Post-Baseline' in the footnote. | W48, W96 |
| 3.55 | 3.60 | NA | Safety | 201585/primar<br>y_02/T3.76 | Summary of Fasting TC/HDL ratio Changes from Baseline (Maintenance Phase) – Lipids LOCF | Change 'Post Baseline' to 'Post-<br>Baseline' in the footnote. | W48, W96 |
| Laborate | ory: Hepat | tobiliary (I | _iver) | | | | • |
| 3.56 | 3.61 | NA | Safety | 201585/primar<br>y_02/T3.80 | Summary of Liver Monitoring/Stopping<br>Event Reporting (Maintenance Phase) | | W48, W96 |
| 3.57 | 3.62 | NA | Safety | 201585/primar<br>y_02/T3.81 | Summary of Subjects Meeting Hepatobiliary<br>Abnormality Criteria (Maintenance Phase) | | W48, W96 |
| NA | 3.63 | 3.20 | Safety | 201585/primar<br>y_02/T3.81 | Summary of Subjects Meeting Hepatobiliary<br>Abnormality Criteria (Maintenance<br>+Extension Phase) | | W96, EOS |
| 3.58 | NA | NA | Oral Lead-<br>in | 201585/primar<br>y_02/T3.84 | Summary of Subjects Meeting Hepatobiliary<br>Abnormality Criteria – Oral Lead-in Period<br>during the Maintenance Phase | Display both arms. | W48 |
| ECG | | | | | | | • |
| 3.59 | 3.64 | 3.21 | Safety | 201585/primar<br>y_02/T3.85 | Summary of ECG Findings (Maintenance + Extension Phase) | Change 'Post Baseline' to 'Post-<br>Baseline' in the footnote. | W48, W96,<br>EOS |
| 3.60 | 3.65 | 3.22 | Safety | 201585/primar<br>y_02/T3.88 | Summary of Change from Baseline in ECG values by Visit (Maintenance + Extension Phase) | Change 'Post Baseline' to 'Post-Baseline' in the footnote. | W48, W96,<br>EOS |
| 3.61 | 3.66 | 3.23 | Safety | 201585/primar<br>y_02/T3.91 | Summary of QTc Values by Category (Maintenance + Extension Phase) | Change 'Post Baseline' to 'Post-<br>Baseline' in the footnote. | W48, W96,<br>EOS |
| Safety T | ables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.62 | 3.67 | 3.24 | Safety | 201585/primar<br>y_02/T3.94 | Summary of Change from Baseline QTc<br>Values by Category (Maintenance +<br>Extension Phase) | Change 'Post Baseline' to 'Post-<br>Baseline' in the footnote. | W48, W96,<br>EOS |
| Vital Sig | ns and eC | C-SSRS | | | | | |
| 3.63 | 3.68 | NA | Safety | 201585/primar<br>y_02/T3.97 | Summary of Change from Baseline in Vital Signs by Visit (Maintenance Phase) | Change 'Post Baseline' to 'Post-Baseline' in the footnote. | W48, W96 |
| 3.64 | 3.69 | NA | Safety | SAFE_T1 | Summary of BMI Shift from Baseline by Visit (Maintenance Phase) | | W48, W96 |
| 3.65 | 3.70 | NA | Safety | 201585/primar<br>y_02/T3.99 | Summary of Subjects with eC-SSRS<br>Suicidal Ideation or Behaviour<br>(Maintenance Phase) | Change 'post baseline' to 'post-<br>baseline' in the row header. | W48, W96 |
| Adverse | Event of | Special In | terest (AESI) | | | | |
| 3.66 | 3.71 | NA | Safety | 201585/primar<br>y_02/T3.100 | Summary of Depression, Anxiety and<br>Suicidal Ideation/Behaviour Adverse Events<br>by System Organ Class, Maximum DAIDS<br>Toxicity Grade, and Prior History of<br>Depression, Anxiety and Suicidal Ideation at<br>Screening (Maintenance Phase) | | W48, W96 |
| 3.67-<br>3.83 | 3.72-<br>3.88 | NA | Safety | 209522/iss_01/<br>T3.38-3.49,<br>T3.51-3.55 | Summary of XXX Adverse Events of<br>Special Interest by System Organ Class<br>and Preferred Term (Number of Subjects<br>and Occurrence) – Maintenance Phase | Only display data from this study, no need for showing study number. For 'XXX', refer to Table 4. | W48, W96 |
| 3.84 | 3.89 | NA | Safety | 209522/iss_01/<br>T3.62 | Summary of Characteristics of Common<br>Adverse Events of Special Interest –<br>Maintenance Phase | Only display data from this study, no need for showing study number. Present by individual common AESI. | W48, W96 |

# **15.14.5.5.** Safety Figures

**Note:** Unless otherwise specified, display both arms.

| Safety F | | | | aispiay oom air | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.1 | 3.1 | NA | Safety | 201585/primar<br>y_02/F3.1 | Plot of Common Adverse Events and Relative Risk - Q8W vs. Q4W (Maintenance Phase) – Excluding Study Drug ISRs | Remove the second footnote. | HL, W48, W96 |
| 3.2 | 3.2 | NA | Safety | 201585/primar<br>y_02/F3.1 | Plot of Common Study Drug Injection Site Reaction<br>Adverse Events and Relative Risk - Q8W vs. Q4W<br>(Maintenance Phase) | Remove the second footnote. | HL, W48, W96 |
| 3.3 | 3.3 | NA | Safety | 201585/primar<br>y_02/F3.5 | Plot of Onset, Duration, and Severity of Overall and Common Study Drug Injection Site Reaction AEs by Maximum Grade — CAB and/or RPV (Maintenance Phase) | | W48, W96 |
| 3.4 | 3.4 | NA | Safety | 201585/primar<br>y_02/F3.6 | Plot of Onset, Duration, and Severity of Overall and Common Drug-related Study Drug Injection Site Reaction AEs by Maximum Grade — CAB (Maintenance Phase) | | W48, W96 |
| 3.5 | 3.5 | NA | Safety | 201585/primar<br>y_02/F3.7 | Plot of Onset, Duration, and Severity of Overall and Common Drug-related Study Drug Injection Site Reaction AEs by Maximum Grade — RPV (Maintenance Phase) | | W48, W96 |
| 3.6 | 3.6 | NA | Safety | 201585/primar<br>y_02/F3.8 | Plot of Incidence of Maintenance Phase Study Drug<br>Injection Site Reaction Adverse Events by Visit<br>(Overall and Common) – CAB and/or RPV | Footnote may be adjusted for clarifications. | W48, W96 |
| 3.7 | 3.7 | NA | Safety | 201585/primar<br>y_02/F3.9 | Plot of Incidence of Maintenance Phase Drug-<br>Related Study Drug Injection Site Reaction Adverse<br>Events by Visit (Overall and Common) – CAB | Footnote may be adjusted for clarifications. | W48, W96 |

| Safety F | igures | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.8 | 3.8 | NA | Safety | 201585/primar<br>y_02/F3.10 | Plot of Incidence of Maintenance Phase Drug-<br>Related Study Drug Injection Site Reaction Adverse<br>Events by Visit (Overall and Common) – RPV | Footnote may be adjusted for clarifications. | W48, W96 |
| 3.9 | 3.9 | NA | Safety | 201585/primar<br>y_02/F3.11 | Plot of Incidence of Grade 3-5 Maintenance Phase<br>Study Drug Injection Site Reaction Adverse Events<br>by Visit (Overall and Common) - CAB and/or RPV | Footnote may be adjusted for clarifications. | W48, W96 |
| 3.10 | 3.10 | NA | Safety | 201585/primar<br>y_02/F3.12 | Plot of Incidence of Grade 3-5 Maintenance Phase<br>Drug-related Study Drug Injection Site Reaction<br>Adverse Events by Visit (Overall and Common) -<br>CAB | Footnote may be adjusted for clarifications. | W48, W96 |
| 3.11 | 3.11 | NA | Safety | 201585/primar<br>y_02/F3.13 | Plot of Incidence of Grade 3-5 Maintenance Phase<br>Drug-related Study Drug Injection Site Reaction<br>Adverse Events by Visit (Overall and Common) -<br>RPV | Footnote may be adjusted for clarifications. | W48, W96 |
| 3.12 | 3.12 | NA | Safety | 201585/primar<br>y_02/F3.2 | Scatter Plot of Maximum vs. Baseline for ALT (Maintenance Phase) | Display at log10 scale. | HL, W48, W96 |
| 3.13 | 3.13 | NA | Safety | 201585/primar<br>y_02/F3.3 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin (Maintenance Phase) | | HL, W48, W96 |
| 3.14 | 3.14 | NA | Safety | 201585/primar<br>y_02/F3.4 | Matrix Plot of Maximum Liver Chemistries during the Maintenance Phase | | HL, W48, W96 |
| 3.15 | 3.15 | NA | Safety | 201585/primar<br>y_02/F3.14 | Bar Chart of Lipid NCEP Categories at Week 48 vs. Baseline – Triglycerides, Total Cholesterol, LDL Cholesterol | For WK96, replace 'Week 48' with 'Week 96' in the title. | W48, W96 |
| 3.16 | 3.16 | NA | Safety | 201585/primar<br>y_02/F3.15 | Bar Chart of Lipid NCEP Categories at Week 48 vs. Baseline - HDL Cholesterol | For WK96, replace 'Week 48' with 'Week 96' in the title. | W48, W96 |

2019N406358\_00 207966

| Safety F | Safety Figures | | | | | |
|---|---|---|---|---|---|---|
| No. in W48 No. in No. in Ros Population IDSL / Example Shell Title Programming Notes Deliveration Deliveration Deliveration Deliveration Programming Notes Deliveration Deliveration | | | | | | Deliverable |
| 3.17 | 3.17 | NA | Safety | SAFE_F1 | Histogram of Timeliness of Injections (Maintenance Phase) | W48, W96 |

# 15.14.5.6. Pharmacokinetic Tables

**Note:** For WK48 deliverable, data from visits up to Week 48 are included.

| Pharma | cokinetic | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 4.1 | 4.1 | NA | Pharmacokinetic | 201585/primary_<br>02/T4.1 | Summary of Plasma CAB PK Concentration (ug/mL) -Time Data by Treatment and Visit – Including Log-transformed Statistics | Remove the first footnote. | W48, W96 |
| 4.2 | 4.2 | NA | Pharmacokinetic | 201585/primary_<br>02/T4.2 | Summary of Plasma RPV PK Concentration (ng/mL) -Time Data by Treatment and Visit – Including Log-transformed Statistics | Remove the first footnote. | W48, W96 |
| 4.3 | 4.3 | NA | Pharmacokinetic | 201585/primary_<br>02/T4.3 | Summary of Evaluable Plasma CAB PK<br>Concentration (ug/mL) -Time Data by Treatment and<br>Visit – Including Log-transformed Statistics | Remove the first footnote. | W48, W96 |
| 4.4 | 4.4 | NA | Pharmacokinetic | 201585/primary_<br>02/T4.4 | Summary of Evaluable Plasma RPV PK Concentration (ng/mL) -Time Data by Treatment and Visit – Including Log-transformed Statistics | Remove the first footnote. | W48, W96 |
| 4.5 | 4.5 | NA | Pharmacokinetic | 201585/primary_<br>02/T4.3 | Summary of Evaluable Plasma CAB PK Concentration (ug/mL) -Time Data by Strata and Treatment and Visit – Including Log-transformed Statistics | Display by rederived randomization strata and add footnote for strata. | W48, W96 |
| 4.6 | 4.6 | NA | Pharmacokinetic | 201585/primary_<br>02/T4.4 | Summary of Evaluable Plasma RPV PK Concentration (ng/mL) -Time Data by Strata and Treatment and Visit – Including Log-transformed Statistics | Display by rederived randomization strata and add footnote for strata. | W48, W96 |
| 4.7 | 4.7 | NA | Pharmacokinetic | 201585/primary_<br>02/T4.6 | Summary of Results of Steady State Assessment by Strata for Q8W Arm- Evaluable Concentration | Display by rederived randomization strata and add footnote for strata. For Q8W arm only. | W48 |

# 15.14.5.7. Pharmacokinetic Figures

**Note:** Unless otherwise specified, display both arms.

| Pharma | cokinetic | Figures | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 4.1 | 4.1 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.1 | Individual Plasma CAB Concentration-<br>Time Plots (Linear and Semi-Log) | Also include prior exposure to CAB+RPV (e.g. 0, 1-24, >24 weeks) for each subject. | W48, W96 |
| 4.2 | 4.2 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.2 | Individual Plasma RPV Concentration-<br>Time Plots (Linear and Semi-Log) | Also include prior exposure to CAB+RPV (e.g. 0, 1-24, >24 weeks) for each subject. | W48, W96 |
| 4.3 | 4.3 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.3 | Mean (SD) Plasma CAB Concentration-<br>Time Plots (Linear and Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.4 | 4.4 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.5 | Mean (SD) Plasma RPV Concentration-<br>Time Plots (Linear and Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.5 | 4.5 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.7 | Mean (SD) Evaluable Plasma CAB<br>Concentration-Time Plots (Linear and<br>Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.6 | 4.6 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.9 | Mean (SD) Evaluable Plasma RPV<br>Concentration-Time Plots (Linear and<br>Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.7 | 4.7 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.7 | Mean (SD) Evaluable Plasma CAB<br>Concentration-Time Plots by Strata<br>(Linear and Semi-Log) | Display by rederived randomization strata and add footnote for strata. For WK48, data from visits up to Week 48 are included. | W48, W96 |

| Pharma | cokinetic | Figures | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 4.8 | 4.8 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.9 | Mean (SD) Evaluable Plasma RPV<br>Concentration-Time Plots by Strata<br>(Linear and Semi-Log) | Display by rederived randomization strata and add footnote for strata. For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.9 | 4.9 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.4 | Median (5th and 95th Percentile) Plasma<br>CAB Concentration-Time Plots (Linear<br>and Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.10 | 4.10 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.6 | Median (5th and 95th Percentile) Plasma<br>RPV Concentration-Time Plots (Linear<br>and Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.11 | 4.11 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.8 | Median (5th and 95th Percentile) Evaluable Plasma CAB Concentration- Time Plots (Linear and Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.12 | 4.12 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.10 | Median (5th and 95th Percentile) Evaluable Plasma RPV Concentration- Time Plots (Linear and Semi-Log) | For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.13 | 4.13 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.8 | Median (5th and 95th Percentile) Evaluable Plasma CAB Concentration- Time Plots by Strata (Linear and Semi- Log) | Display by rederived randomization strata and add footnote for strata. For WK48, data from visits up to Week 48 are included. | W48, W96 |
| 4.14 | 4.14 | NA | Pharmacokinetic | 201585/primary_02/<br>F4.10 | Median (5th and 95th Percentile) Evaluable Plasma RPV Concentration- Time Plots by Strata (Linear and Semi- Log) | Display by rederived randomization strata and add footnote for strata. For WK48, data from visits up to Week 48 are included. | W48, W96 |

# 15.14.5.8. Pharmacokinetic / Pharmacodynamic Tables

**Note:** Unless otherwise specified, display by treatment arm.

| Pharma | Pharmacokinetic / Pharmacodynamic Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| PK / PD | Efficacy | | | | | | |
| 5.1 | 5.1 | NA | Pharmacokinetic | 201584/primary_0<br>1/T5.1 | Univariable Logistic Regression Analysis of Snapshot 'HIV-1 RNA ≥50 c/mL' at Week 48 by Trough PK Concentration and Subgroup for Subjects without Prior Exposure to CAB + RPV | For WK96, replace 'Week 48' with 'Week 96' in title. Do not display by treatment arm. | W48, W96 |
| 5.2 | 5.2 | NA | Pharmacokinetic | 201584/primary_0<br>1/T5.2 | Multivariable Logistic Regression Analysis of Predictors of Snapshot 'HIV-1 RNA ≥50 c/mL' at Week 48 for Subjects without Prior Exposure to CAB + RPV | For WK96, replace 'Week 48' with 'Week 96' in title. Adjust the footnote as appropriate. Do not display by treatment arm. | W48, W96 |
| 5.3 | 5.3 | NA | Pharmacokinetic | 201584/primary_0<br>1/T5.5 | Summary of Week 8 Trough CAB PK concentration by Snapshot 'HIV-1 RNA ≥50 c/mL' (Yes vs. No) at Week 48 for Subjects without Prior Exposure to CAB + RPV – Including Log-transformed Statistics | For WK96, replace 'Week 48' with 'Week 96' in title. | W48, W96 |
| 5.4 | 5.4 | NA | Pharmacokinetic | 201584/primary_0<br>1/T5.6 | Summary of Week 8 Trough RPV PK concentration by Snapshot 'HIV-1 RNA ≥50 c/mL' (Yes vs. No) at Week 48 for Subjects without Prior Exposure to CAB + RPV – Including Log-transformed Statistics | For WK96, replace 'Week 48' with 'Week 96' in title. | W48, W96 |

# 15.14.5.9. Pharmacokinetic / Pharmacodynamic Figures

| Pharma | Pharmacokinetic / Pharmacodynamic Figures | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| PK / PD | Efficacy A | nalyses | | | | | |
| 5.1 | 5.1 | NA | Pharmacokinetic | 201585/primary_<br>02/F5.3 | Scatter Plot of Week 8 Trough CAB PK Concentration by Snapshot 'HIV-1 RNA ≥50 c/mL' (Yes vs. No) at Week 48 for Subjects without Prior Exposure to CAB + RPV | For WK96, replace 'Week 48' with 'Week 96' in title. Display by treatment arm. | W48, W96 |
| 5.2 | 5.2 | NA | Pharmacokinetic | 201585/primary_<br>02/F5.4 | Scatter Plot of Week 8 Trough RPV PK<br>Concentration by Snapshot 'HIV-1 RNA ≥50<br>c/mL' (Yes vs. No) at Week 48 for Subjects<br>without Prior Exposure to CAB + RPV | For WK96, replace 'Week 48' with 'Week 96' in title. Display by treatment arm. | W48, W96 |
| 5.3 | 5.3 | NA | Pharmacokinetic | 201585/primary_<br>02/F5.7 | Individual CAB Trough Concentration-time Profiles for Subjects with Snapshot 'HIV-1 RNA ≥50 c/mL' at Week 48 and Median, 5th & 95th Percentile of CAB Conc-Time Profiles for Other Subjects (Semi-Log) | For WK96, replace 'Week 48' with 'Week 96' in title. Display by treatment arm. | W48, W96 |
| 5.4 | 5.4 | NA | Pharmacokinetic | 201585/primary_<br>02/F5.8 | Individual RPV Trough Concentration-time Profiles for Subjects with Snapshot 'HIV-1 RNA ≥50 c/mL' at Week 48 and Median, 5th & 95th Percentile of RPV Conc-Time Profiles for Other Subjects (Semi-Log) | For WK96, replace 'Week 48' with 'Week 96' in title. Display by treatment arm. | W48, W96 |
| 5.5 | 5.5 | NA | Pharmacokinetic | 201585/primary_<br>02/F5.10 | Scatter Plot of Week 8 Trough Concentration of CAB and RPV in Relation to Occurrence of Snapshot 'HIV-1 RNA ≥50 c/mL' at Week 48 for Subjects without Prior Exposure to CAB + RPV | For WK96, replace 'Week 48' with 'Week 96' in title. Display by treatment arm. | W48, W96 |

| Pharma | Pharmacokinetic / Pharmacodynamic Figures | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| PK / PD | PK / PD Safety Analyses | | | | | | |
| 5.6 | 5.6 | NA | Pharmacokinetic | 201585/primary_<br>02/F5.13 | Scatter Plot of Maximum Change from<br>Baseline in ALT versus Last Trough CAB<br>PK Concentrations by Strata and Treatment<br>during the Maintenance Phase | Display by strata and treatment arm. Add footnote for rederived randomization strata. | W48, W96 |
| 5.7 | 5.7 | NA | Pharmacokinetic | 201585/primary_<br>02/F5.14 | Scatter Plot of Maximum Change from Baseline in ALT versus Last Trough RPV PK Concentrations by Strata and Treatment during the Maintenance Phase | Display by strata and treatment arm. Add footnote for rederived randomization strata. | W48, W96 |
| 5.8 | 5.8 | NA | Pharmacokinetic | 201585/primary_<br>02/F5.15 | Scatter Plot of Maximum Change from Baseline in Total Bilirubin versus Last Trough CAB PK Concentrations by Strata and Treatment during the Maintenance Phase | Display by strata and treatment arm. Add footnote for rederived randomization strata. | W48, W96 |
| 5.9 | 5.9 | NA | Pharmacokinetic | 201585/primary_<br>02/F5.16 | Scatter Plot of Maximum Change from<br>Baseline in Total Bilirubin versus Last<br>Trough RPV PK Concentrations by Strata<br>and Treatment during the Maintenance<br>Phase | Display by strata and treatment arm. Add footnote for rederived randomization strata. | W48, W96 |
| 5.10 | 5.10 | NA | Pharmacokinetic | 201585/primary_<br>02/F5.17 | Box Plot of Maximum Toxicity Grades of<br>Most Frequently Reported Study Drug ISR<br>Adverse Events versus Last Trough CAB<br>PK Concentrations during the Maintenance<br>Phase by Strata and Treatment | Display by strata and treatment arm. Add footnote for rederived randomization strata. Adjust the footnotes as appropriate. | W48, W96 |

| Pharma | Pharmacokinetic / Pharmacodynamic Figures | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 5.11 | 5.11 | NA | Pharmacokinetic | 201585/primary_<br>02/F5.18 | Box Plot of Maximum Toxicity Grades of<br>Most Frequently Reported Study Drug ISR<br>Adverse Events versus Last Trough RPV<br>PK Concentrations during the Maintenance<br>Phase by Strata and Treatment | Display by treatment arm. Adjust the footnotes as appropriate. | W48, W96 |

# 15.14.5.10. Health Outcomes Tables

| Health ( | Health Outcomes Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Percept | ion of Inje | ection (PI | N) | | | | |
| 6.1 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.1 | Proportion of Subjects with Each Individual Item<br>Score in PIN by Visit –LOCF (Maintenance<br>Phase) | Display both arms. | W48 |
| 6.2 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.2 | Summary of PIN in Domain Scores (CCI and Individual Items Scores (CCI by Individual Items Scor | Display both arms. | W48 |
| 6.3 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.3 | Summary and Statistical Analysis of PIN in Domain Scores (CCI) and CCI) and Individual Items Scores (CCI) by Visit - LOCF (Maintenance Phase) | Display both arms. Adjust the first half of the footnote to "[1] Week 24/48 was compared with the 1st visit (Week 8) based on Wilcoxon signed-rank test, respectively." | W48 |
| 6.4 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.4 | Summary of PIN Change from Week 8 in Domain Scores (Columbia) and Individual Items Scores (Columbia) by Visit (Maintenance Phase) | Display both arms. Adjust the footnote to "Note: Actual values are shown at Week 8." | W48 |

| Health C | Outcomes | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.5 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.5 | Summary of PIN Change from Week 8 in Domain Scores (CCI and CCI ) and Individual Items Scores (CCI ) by Visit – LOCF (Maintenance Phase) | Display both arms. Adjust the footnote to "Note: Actual values are shown at Week 8." | W48 |
| 6.6 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.11 | Statistical Analysis of PIN Change from Week 8 in Domain Scores (PCI and CCI and Individual Items Scores (PCI by Visit – LOCF (Maintenance Phase) | Adjust the column header and the footnote as appropriate. | W48 |
| Health-r | elated Qu | uality of L | ife (HAT-QoL) | ) | | | _ |
| 6.7 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.6 | Proportion of Subjects with Each Individual Questionnaire Item Score in HAT-QoL by Visit - LOCF (Maintenance Phase) | | W48 |
| 6.8 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.7 | Summary of Quality of Life (HAT-QoL) Score in<br>Life Satisfaction, HIV Medication, and Disclosure<br>worries by Visit (Maintenance phase) | | W48 |
| 6.9 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.8 | Summary of Quality of Life (HAT-QoL) Score in Life Satisfaction, HIV Medication, and Disclosure worries by Visit - LOCF (Maintenance phase) | | W48 |
| 6.10 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.9 | Summary of Quality of Life Score (HAT-QoL)-<br>Change from Baseline in Life Satisfaction, HIV<br>Medication, and Disclosure Worries by Prior<br>Exposure to CAB+RPV (0 vs. >=1 Weeks) and<br>Visit (Maintenance Phase) | | W48 |

| Health ( | Outcomes | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.11 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.10 | Summary of Quality of Life Score (HAT-QoL)-<br>Change from Baseline in Life Satisfaction, HIV<br>Medication, and Disclosure Worries by Prior<br>Exposure to CAB+RPV (0 vs. >=1 Weeks) and<br>Visit – LOCF (Maintenance Phase) | | W48 |
| 6.12 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.11 | Statistical Analysis of Quality of Life Score (HAT-QoL)- Change from Baseline in Life Satisfaction, HIV Medication, and Disclosure Worries by Visit for Subjects without Prior Exposure to CAB+RPV – LOCF (Maintenance Phase) | Adjust the column header and the footnote as appropriate. | W48 |
| 6.13 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.11 | Statistical Analysis of Quality of Life Score (HAT-QoL)- Change from Baseline in Life Satisfaction, HIV Medication, and Disclosure Worries by Visit for Subjects with Prior Exposure to CAB+RPV – LOCF (Maintenance Phase) | Adjust the column header and the footnote as appropriate. | W48 |
| HIV Trea | atment Sa | tisfaction | n Questionnai | re Status Versior | n (HIVTSQs) | | |
| 6.14 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.18 | Proportion of Subjects with HIVTSQs - Individual Item Scores by Visit - LOCF (Maintenance Phase) | | W48 |
| 6.15 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.19 | Proportion of Subjects with HIVTSQs - Individual Item Scores by Visit and Subgroup - LOCF (Maintenance Phase) | The subgroup includes: prior exposure to CAB+RPV (0, 1-24, >=24 weeks), sex at birth, age (<35, 35 - <50, >=50), race (white, non-white), Baseline CD4+ cell count (<350, 350 - <500, >=500) | W48 |

| Health ( | Outcomes | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.16 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.20 | Summary of HIVTSQs - Total Treatment<br>Satisfaction Score by Visit (Maintenance Phase) | | W48 |
| 6.17 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.21 | Summary of HIVTSQs - Total Treatment<br>Satisfaction Score by Visit – LOCF (Maintenance<br>Phase) | | W48 |
| 6.18 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.22 | Summary of HIVTSQs - Change from Baseline in Total Treatment Satisfaction Score by Prior Exposure to CAB+RPV (0 vs. >=1 Weeks) and Visit (Maintenance Phase) | | W48 |
| 6.19 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.23 | Summary of HIVTSQs - Change from Baseline in Total Treatment Satisfaction Score by Prior Exposure to CAB+RPV (0 vs. >=1 Weeks) and Visit – LOCF (Maintenance Phase) | | W48 |
| 6.20 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_03/T7.41 | Summary of HIVTSQs - Change from Baseline in Individual Item Score by Prior Exposure to CAB+RPV (0 vs. >=1 Weeks) and Visit – LOCF (Maintenance Phase) | | W48 |
| 6.21 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.24 | Statistical Analysis of HIVTSQs - Change from<br>Baseline in Total Treatment Satisfaction Score by<br>Visit for Subjects without Prior Exposure to<br>CAB+RPV - LOCF (Maintenance Phase) | Adjust column header and footnote as appropriate. | W48 |
| 6.22 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.24 | Statistical Analysis of HIVTSQs - Change from<br>Baseline in Total Treatment Satisfaction Score by<br>Visit for Subjects with Prior Exposure to<br>CAB+RPV - LOCF (Maintenance Phase) | Adjust column header and footnote as appropriate. | W48 |

| Health ( | Outcomes | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| HIV Trea | atment Sa | atisfaction | n Questionnai | re Change Version | on (HIVTSQc) | | |
| 6.23 | NA | NA | Q4W<br>ATLAS | 201584/primar<br>y_01/T6.25 | Proportion of Subjects with HIVTSQc - Individual Item Change Score at Week 48 (Maintenance Phase) for Subjects from Q4W ATLAS | | W48 |
| 6.24 | NA | NA | SOC | 201584/primar<br>y_01/T6.25 | Proportion of Subjects with HIVTSQc - Individual Item Change Score at Week 48 (Maintenance Phase) for Subjects from SOC | | W48 |
| 6.25 | NA | NA | Q4W<br>ATLAS | 201584/primar<br>y_01/T6.26 | Summary of HIVTSQc – Total Treatment<br>Satisfaction Change Score at Week 48<br>(Maintenance Phase) for Subjects from Q4W<br>ATLAS | | W48 |
| 6.26 | NA | NA | SOC | 201584/primar<br>y_01/T6.26 | Summary of HIVTSQc – Total Treatment<br>Satisfaction Change Score at Week 48<br>(Maintenance Phase) for Subjects from SOC | | W48 |
| 6.27 | NA | NA | Q4W<br>ATLAS | 201584/primar<br>y_02/T6.41 | Summary of HIVTSQc – Individual Item Change<br>Score at Week 48 (Maintenance Phase) for<br>Subjects from Q4W ATLAS | | W48 |
| 6.28 | NA | NA | SOC | 201584/primar<br>y_02/T6.41 | Summary of HIVTSQc – Individual Item Change<br>Score at Week 48 (Maintenance Phase) for<br>Subjects from SOC | | W48 |
| 6.29 | NA | NA | Q4W<br>ATLAS | 201584/primar<br>y_01/T6.27 | Statistical Analysis of HIVTSQc – Total Treatment<br>Satisfaction Change Score at Week 48 for<br>Subjects from Q4W ATLAS | Adjust column header and footnote as appropriate. | W48 |
| 6.30 | NA | NA | SOC | 201584/primar<br>y_01/T6.27 | Statistical Analysis of HIVTSQc – Total Treatment<br>Satisfaction Change Score at Week 48 for<br>Subjects from SOC | Adjust column header and footnote as appropriate. | W48 |

| Health ( | Outcomes | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Treatme | ent Accep | tance (A | CCEPT) | | | | |
| 6.31 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.28 | Proportion of Subjects with ACCEPT - Individual Item Score by Visit - LOCF (Maintenance Phase) | | W48 |
| 6.32 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.29 | Summary of Acceptance/General Dimension<br>Score (ACCEPT Questionnaire) by Visit<br>(Maintenance Phase) | | W48 |
| 6.33 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.30 | Summary of Acceptance/General Dimension<br>Score (ACCEPT Questionnaire) by Visit - LOCF<br>(Maintenance Phase) | | W48 |
| 6.34 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.31 | Summary of Change from Baseline in<br>Acceptance/General Dimension Score (ACCEPT<br>Questionnaire) by Prior Exposure to CAB+RPV (0<br>vs. >=1 Weeks) and Visit (Maintenance Phase) | | W48 |
| 6.35 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.32 | Summary of Change from Baseline in<br>Acceptance/General Dimension Score (ACCEPT<br>Questionnaire) by Prior Exposure to CAB+RPV (0<br>vs. >=1 Weeks) and Visit - LOCF (Maintenance<br>Phase) | | W48 |
| 6.36 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.33 | Statistical Analysis of Change from Baseline in Acceptance/General Dimension Score (ACCEPT Questionnaire) by Visit for Subjects without Prior Exposure to CAB+RPV – LOCF (Maintenance Phase) | Adjust column header and footnote as appropriate. | W48 |

| Health ( | Outcomes | Tables | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.37 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/T7.33 | Statistical Analysis of Change from Baseline in Acceptance/General Dimension Score (ACCEPT Questionnaire) by Visit for Subjects with Prior Exposure to CAB+RPV – LOCF (Maintenance Phase) | Adjust column header and footnote as appropriate. | W48 |
| Prefere | nce | | | | | | |
| 6.38 | NA | NA | Q4W<br>ATLAS | Shell HO_T1 | Proportion of Subjects with Response to Each Individual Question in Preference Questionnaire at Week 48 (Maintenance Phase) for Subjects from Q4W ATLAS to Q8W ATLAS-2M | Only display Q8W arm. | HL, W48 |
| 6.39 | NA | NA | Intent-to-<br>Treat<br>Exposed | Shell HO_T1 | Proportion of Subjects with Response to Each Individual Question in Preference Questionnaire by Prior Exposure to CAB+RPV (0 vs. >=1 Weeks) at Week 48 for Subjects in Q8W ATLAS-2M (Maintenance Phase) | Only display Q8W arm. | W48 |
| 6.40 | NA | NA | Intent-to-<br>Treat<br>Exposed | Shell HO_T1 | Proportion of Subjects with Response to Each Individual Question in Preference Questionnaire at Week 48 for Subjects in Q4W ATLAS-2M (Maintenance Phase) | Only display Q4W arm. | W48 |
| Reason | s for Swit | ch/Conti | nuation | | | | |
| 6.41 | NA | NA | SOC | 201585/primar<br>y_02/T7.40 | Reasons for Switch at Baseline for Subjects from SOC | Remove columns 'Analysis Visit' and 'Total'. For percentages, use the format 'xx / xx (xx%)' where the denominator is the number of subjects with available valid data from the questionnaire. | W48 |

| Health C | Health Outcomes Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 6.42 | NA | NA | Q4W<br>ATLAS | 201585/primar<br>y_02/T7.40 | Reasons for Continuation at Baseline for Subjects from Q4W ATLAS | Remove columns 'Analysis Visit' and 'Total'. For percentages, use the format 'xx / xx (xx%)' where the denominator is the number of subjects with available valid data from the questionnaire. | W48 |

# 15.14.5.11. Health Outcomes Figures

| Health C | Outcomes | Figures | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 6.1 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.1 | Line Plot of Adjusted Mean (95% CI) Change from Baseline in HIVTSQs Total Treatment Satisfaction Score over Time(ANCOVA) for Subjects without Prior Exposure to CAB+RPV - LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |
| 6.2 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.1 | Line Plot of Adjusted Mean (95% CI) Change from Baseline in HIVTSQs Total Treatment Satisfaction Score over Time(ANCOVA) for Subjects with Prior Exposure to CAB+RPV - LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |
| 6.3 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.2 | Line Plot of Difference (95% CI) in Adjusted Mean<br>Change from Baseline in HIVTSQs Total Treatment<br>Satisfaction Score over Time (ANCOVA) for<br>Subjects without Prior Exposure to CAB+RPV -<br>LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |
| 6.4 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.2 | Line Plot of Difference (95% CI) in Adjusted Mean<br>Change from Baseline in HIVTSQs Total Treatment<br>Satisfaction Score over Time (ANCOVA) for<br>Subjects with Prior Exposure to CAB+RPV - LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |
| 6.5 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.5 | Line Plot of Adjusted Mean (95% CI) Change from Baseline in HAT-QoL (Life Satisfaction, HIV medication, and Disclosure Worries) by Visit (ANCOVA) for Subjects without Prior Exposure to CAB+RPV - LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |

| Health C | Outcomes | Figures | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 6.6 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.5 | Line Plot of Adjusted Mean (95% CI) Change from Baseline in HAT-QoL (Life Satisfaction, HIV medication, and Disclosure Worries) by Visit (ANCOVA) for Subjects with Prior Exposure to CAB+RPV - LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |
| 6.7 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.6 | Line Plot of Difference in Adjusted Mean (95% CI) Change from Baseline in HAT-QoL (Life Satisfaction, HIV Medication, and Disclosure Worries) by Visit (ANCOVA) for Subjects without Prior Exposure to CAB+RPV - LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |
| 6.8 | NA | NA | Intent-to-<br>Treat<br>Exposed | 201585/primary<br>_02/F7.6 | Line Plot of Difference in Adjusted Mean (95% CI) Change from Baseline in HAT-QoL (Life Satisfaction, HIV Medication, and Disclosure Worries) by Visit (ANCOVA) for Subjects with Prior Exposure to CAB+RPV - LOCF | Adjust footnotes as appropriate. Include Baseline as a timepoint in x axis. | W48 |

# **15.14.5.12. Virology Tables**

| Virology | y Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Genoty | ре | | | | | | |
| 7.1 | 7.1 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.1 | Summary of the Prevalence of Known INI Resistance<br>Mutations at time of CVF (Maintenance Phase) –<br>Plasma Sample | | W48, W96 |
| 7.2 | 7.2 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.2 | Summary of the Prevalence of Major Resistance<br>Mutations of NRTI, NNRTI and PI Class at time of<br>CVF (Maintenance Phase) - Plasma Sample | | W48, W96 |
| 7.3 | 7.3 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.4 | Summary of Genotypic Susceptibility at time of CVF (Maintenance Phase) - Plasma Sample | | W48, W96 |
| Phenoty | уре | | | | | | |
| 7.4 | 7.4 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.3 | Summary of Phenotype Susceptibility at time of CVF (Maintenance Phase) - Plasma Sample | | W48, W96 |
| 7.5 | 7.5 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.6 | Summary of Phenotype: Number of Drugs to Which<br>Subject is Phenotypic Resistant or Partial Sensitive<br>or Sensitive at Time of CVF (Maintenance Phase) -<br>Plasma Sample | | W48, W96 |
| 7.6 | 7.6 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.7 | Summary of Fold Change to CAB and RPV at Time of CVF (Maintenance Phase) - Plasma Sample | | W48, W96 |
| 7.7 | 7.7 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.5 | Summary of Net Assessment at time of CVF (Maintenance Phase) - Plasma Sample | | W48, W96 |

| Virology | Virology Tables | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Miscella | neousne | SS | | | | | |
| 7.8 | 7.8 | NA | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.8 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure Criteria during the Maintenance Phase | Remove columns for 'ARTs',<br>'FC for ARTs'. Adjust the<br>footnotes as appropriate. | HL, W48,<br>W96 |
| NA | 7.9 | 7.1 | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/T8.8 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure Criteria during the Extension Phase | Remove columns for 'ARTs',<br>'FC for ARTs'. Adjust the<br>footnotes as appropriate. | W96, EOS |
| 7.9 | 7.10 | 7.2 | Safety | 201585/primar<br>y_02/T8.8 | Summary of Viral load, Genotypic and Phenotypic data for Non-CVF Subjects with Genotypic and/or Phenotypic Data | Remove columns for 'ARTs',<br>'FC for ARTs'. Adjust the<br>footnotes as appropriate. | W48, W96,<br>EOS |

# 15.14.5.13. ICH Listings

**Note:** Unless otherwise specified, both unique subject ID and latest subject ID for a subject will be included in the listings; display by prior exposure to CAB+RPV (0, 1-24, >24 weeks, refer to Section 15.6.2 for calculation details) for all listings except for study population listings.

| ICH List | ings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Study P | opulation | 1 | | | | | |
| 1 | 1 | 1 | Randomized | 201585/prima<br>ry_02/L1 | Listing of Subjects Randomized but Not Treated | | W48, W96, EOS |
| 2 | 2 | 2 | Randomized | 201585/prima<br>ry_02/L2 | Listing of Randomized and Actual<br>Strata and Treatment Assignment | Randomized and Actual Treatments will include oral lead-in information (e.g. Oral followed by Q4W). Change the footnote # for column 'Dev.' to be [2]. Add a footnote for actual strata: [1] Actual strata are derived using the prior exposure to CAB+RPV in Study 201585, collected from eCRF. | W48, W96, EOS |
| 3 | 3 | 3 | Screened | 201585/prima<br>ry_02/L3 | Listing of Reasons for Screen Failure | | W48, W96, EOS |
| 4 | 4 | 4 | Intent-to-<br>Treat<br>Exposed | ES2 | Listing of Reasons for Study<br>Withdrawal | | HL, W48, W96,<br>EOS |
| 5 | 5 | 5 | Intent-to-<br>Treat<br>Exposed | 201585/prima<br>ry_02/L5 | Listing of Reasons for Study Drug<br>Discontinuation | | W48, W96, EOS |

| ICH List | ICH Listings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 6 | 6 | 6 | Intent-to-<br>Treat<br>Exposed | 201585/prima<br>ry_02/L6 | Listing of Important Protocol Deviations | | W48, W96, EOS |
| 7 | 7 | 7 | Intent-to-<br>Treat<br>Exposed | 201585/prima<br>ry_02/L7 | Listing of Protocol Deviations<br>Leading to Exclusion from the Per-<br>Protocol Population | | HL, W48, W96,<br>EOS |
| 8 | 8 | 8 | Intent-to-<br>Treat<br>Exposed | 201585/prima<br>ry_02/L8 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | W48, W96, EOS |
| 9 | 9 | 9 | Intent-to-<br>Treat<br>Exposed | 201585/prima<br>ry_02/L9 | Listing of Demographic<br>Characteristics | | W48, W96, EOS |
| 10 | 10 | 10 | Intent-to-<br>Treat<br>Exposed | 201585/prima<br>ry_02/L10 | Listing of Race | | W48, W96, EOS |
| Efficacy | | | | | | | |
| 11 | 11 | 11 | Intent-to-<br>Treat<br>Exposed | 201585/prima<br>ry_02/L11 | Listing of Study Outcome (50 c/mL<br>Threshold) at Week 48 – Snapshot<br>Analysis | | HL, W48, W96,<br>EOS |
| Safety: I | Exposure | ) | | | | | |
| 12 | 12 | 12 | Safety | 201585/prima<br>ry_02/L12 | Listing of Investigational Product Exposure Data | | W48, W96, EOS |

| ICH List | ICH Listings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Safety: | Adverse | Events | | | | | |
| 13 | 13 | 13 | Safety | 201585/prima<br>ry_02/L13 | Listing of Subject Numbers for Individual Adverse Events (Maintenance + Extension Phase) | | W48, W96, EOS |
| 14 | 14 | 14 | Safety | 201585/prima<br>ry_02/L14 | Listing of Reasons for Considering as a Serious Adverse Event (Maintenance + Extension Phase) | | W48, W96, EOS |
| 15 | 15 | 15 | Safety | 201585/prima<br>ry_02/L15 | Listing of Fatal Adverse Events (Maintenance + Extension Phase) | Add Study Period to the 5 <sup>th</sup> Column from the left. | W48, W96, EOS |
| 16 | 16 | 16 | Safety | 201585/prima<br>ry_02/L16 | Listing of Non-Fatal Serious<br>Adverse Events (Maintenance +<br>Extension Phase) | Add Study Period to the 5 <sup>th</sup> Column from the left. | W48, W96, EOS |
| 17 | 17 | 17 | Safety | 201585/prima<br>ry_02/L17 | Listing of Adverse Events Leading<br>to Withdrawal/Permanent<br>Discontinuation of Investigational<br>Product (Maintenance + Extension<br>Phase) | Add Study Period to the 5 <sup>th</sup> Column from the left. | HL, W48, W96,<br>EOS |
| 18 | 18 | 18 | Safety | 201585/prima<br>ry_02/L18 | Listing of Changes in Intensity/Grades of Study Drug Injection Site Adverse Events (Maintenance + Extension Phase) | | W48, W96, EOS |
| 19 | 19 | 19 | Safety | 201585/prima<br>ry_03/L30 | Listing of All Adverse Events (Maintenance + Extension Phase) | Add Study Period to the 5 <sup>th</sup> Column from the left. | W48, W96, EOS |

| ICH List | ICH Listings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Safety: I | Pregnanc | у | | | | | |
| 20 | 20 | 20 | Safety | 201585/prima<br>ry_02/L19 | Listing of Subjects Who Became Pregnant during the Study (Maintenance + Extension Phase) | | W48, W96, EOS |

| ICH List | ICH Listings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Safety: I | Hepatobi | liary (Liv | er) | | | | |
| 21 | 21 | 21 | Safety | 201585/prima<br>ry_02/L20 | Listing of Medical Conditions for Subjects with Liver stopping Events | | W48, W96, EOS |
| 22 | 22 | 22 | Safety | 201585/prima<br>ry_02/L21 | Listing of Substance Use for Subjects with Liver Stopping Events | | W48, W96, EOS |
| Safety: I | ECG | | | | | | |
| 23 | 23 | 23 | Safety | 201584/prima<br>ry_01/L24 | Listing of ECG Values for Subjects with a Value of Potential Clinical Importance | Remove Phase Treatment from the column header. Add change from baseline values for each of QTc assessment. Adjust the footnote as appropriate. A footnote may be added to clarify the classification of PCI values. | W48, W96, EOS |
| 24 | 24 | 24 | Safety | 201584/prima<br>ry_01/L23 | Listing of ECG Findings | | W48, W96, EOS |
| Safety: 6 | C-SSRS | | | | | | |
| 25 | 25 | 25 | Safety | 201585/prima<br>ry_02/L24 | Listing of Possible Suicidality-<br>Related Adverse Event Data: Event<br>and Description (Section 1-Section<br>2) | | W48, W96, EOS |
| 26 | 26 | 26 | Safety | 201585/prima<br>ry_02/L25 | Listing of Possible Suicidality-<br>Related Adverse Event Data:<br>Possible Cause(s) (Section 3) | | W48, W96, EOS |
| 27 | 27 | 27 | Safety | 201585/prima<br>ry_02/L26 | Listing of Possible Suicidality-<br>Related Adverse Event Data<br>(Section 4) | | W48, W96, EOS |

| ICH List | ICH Listings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 28 | 28 | 28 | Safety | 201585/prima<br>ry_02/L27 | Listing of Possible Suicidality-<br>Related Adverse Event Data<br>(Section 5-Section 8) | | W48, W96, EOS |
| PK | | | | | | | |
| 29 | 29 | 29 | Pharmacokin etic | 201584/prima<br>ry_01/L30 | Listing of Plasma CAB PK Concentration-Time Data | Remove 'Phase Treatment' from the column header. | W48, W96, EOS |
| 30 | 30 | 30 | Pharmacokin etic | 201584/prima<br>ry_01/L31 | Listing of Plasma RPV PK Concentration-Time Data | Remove 'Phase Treatment' from the column header. | W48, W96, EOS |

# **15.14.5.14. Non-ICH Listings**

**Note:** Unless otherwise specified, both unique subject ID and latest subject ID for a subject will be included in the listings; display by prior exposure to CAB+RPV (0, 1-24, >24 weeks, refer to calculation details in Section 15.6.2) for all listings except for study population listings.

| Non-ICH | Non-ICH Listings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Study P | Study Population | | | | | | |
| 31 | 31 | 31 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/L30 | Listing of Reasons for Maintenance Phase Withdrawal | | W48, W96, EOS |
| 32 | 32 | 32 | Oral Lead-<br>in | 201585/primar<br>y_02/L31 | Listing of Reasons for Oral Lead-in Period<br>Withdrawal | | W48, W96, EOS |
| NA | 33 | 33 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/L32 | Listing of Reasons for Extension Phase<br>Withdrawal | | W96, EOS |
| 33 | 34 | 34 | Long-term<br>Follow-up | 201585/primar<br>y_02/L33 | Listing of Reasons for Long-term Follow-up Phase Withdrawal | | W48, W96, EOS |
| 34 | 35 | 35 | Screened | Shell POP_L2 | Listing of Subjects Who were Rescreened | | W48, W96, EOS |
| 35 | 36 | 36 | Intent-to-<br>Treat<br>Exposed | Shell POP_L1 | Listing of Prior ART Medications | Remove the column 'Phase during Which Concomitant' | W48, W96, EOS |
| 36 | 37 | 37 | Intent-to-<br>Treat<br>Exposed | Shell POP_L1 | Listing of Concomitant ART Medications | In case the same medication is concomitant during both maintenance and extension phases, list each of them in two separate rows. | W48, W96, EOS |

| Non-ICH | l Listings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 37 | 38 | 38 | Intent-to-<br>Treat<br>Exposed | Shell POP_L1 | Listing of ART Medications Received during Long-term Follow-up Phase | Remove the column 'Phase during Which Concomitant' | W48, W96, EOS |
| 38 | 39 | 39 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/L39 | Listing of Investigational Product Accountability - Oral Regimens | | W48, W96, EOS |
| 39 | 40 | 40 | Intent-to-<br>Treat<br>Exposed | 201584/primar<br>y_01/L43 | Listing of Medical History of Seizure | | W48, W96, EOS |
| Efficacy | | | | | | | |
| 40 | 41 | 41 | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/L40 | Listing of All Plasma HIV-1 RNA data for subjects with Confirmed Virologic Failure | In column headers, replace 'Period' with 'Phase', replace 'Sample Day' with 'Study Day'. | W48, W96, EOS |
| 41 | 42 | 42 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/L41 | Listing of All Plasma HIV-1 RNA data for subjects with viral load >=50 c/mL during the Maintenance Phase | In column headers, replace 'Period' with 'Phase', replace 'Sample Day' with 'Study Day'. | HL, W48, W96,<br>EOS |
| 42 | NA | NA | Oral Lead-<br>in | 201585/primar<br>y_02/L41 | Listing of All Plasma HIV-1 RNA data for subjects with viral load >=50 c/mL during the Maintenance Oral Lead-in Period | In column headers, replace 'Period' with 'Phase', replace 'Sample Day' with 'Study Day'. | W48 |
| 43 | 43 | 43 | Intent-to-<br>Treat<br>Exposed | 201585/primar<br>y_02/L43 | Listing of HIV-1 Associated Conditions (Maintenance + Extension Phase) | | W48, W96, EOS |
| Safety (I | list data d | during Ma | aintenance an | d Extension Phas | ses, unless otherwise specified) | | |
| 44 | 44 | 44 | Safety | ABC_HSR_EX<br>PO2 | Listing of Abacavir Hypersensitivity Reaction<br>Record - Exposure to Abacavir | | W48, W96, EOS |

| Non-ICH | Non-ICH Listings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 45 | 45 | 45 | Safety | ABC_HSR_DR<br>UG2 | Listing of Abacavir Hypersensitivity Reaction Record - Subject History of Drug Allergies | | W48, W96, EOS |
| 46 | 46 | 46 | Safety | ABC_HSR_CO<br>ND2 | Listing of Abacavir Hypersensitivity Reaction Record - Subject and Family Conditions | | W48, W96, EOS |
| 47 | 47 | 47 | Safety | ABC_HSR_RA<br>SH2 | Listing of Abacavir Hypersensitivity Reaction Record - Skin Rash Details | | W48, W96, EOS |
| 48 | 48 | 48 | Safety | ABC_HSR_SY<br>MP4 | Listing of Abacavir Hypersensitivity Reaction Record - Symptoms | | W48, W96, EOS |
| 49 | 49 | 49 | Safety | VS4 | Listing of Abacavir Hypersensitivity Reaction Record - Vital Signs | | W48, W96, EOS |
| 50 | 50 | 50 | Safety | ABC_HSR<br>_SYMP6 | Listing of Abacavir Hypersensitivity Reaction<br>Record - Individual Symptoms and Diagnostic<br>Category Assignments (Excluding Other<br>Symptoms) | | W48, W96, EOS |
| 51 | 51 | 51 | Safety | ABC_HSR_SY<br>MP7 | Listing of Abacavir Hypersensitivity Reaction<br>Record - Individual Symptoms and Diagnostic<br>Category Assignments (Other Symptoms) | | W48, W96, EOS |
| 52 | 52 | 52 | Safety | 201585/primar<br>y_02/L52 | Listing of Liver monitoring/stopping Event Reporting | | W48, W96, EOS |
| 53 | 53 | 53 | Safety | 201585/primar<br>y_02/L53 | Listing of Liver Event Information for RUCAM Score | | W48, W96, EOS |
| 54 | 54 | 54 | Safety | 201585/primar<br>y_02/L54 | Listing of Liver Biopsy Details | | W48, W96, EOS |
| 55 | 55 | 55 | Safety | 201585/primar<br>y_02/L55 | Listing of Liver Imaging Details | | W48, W96, EOS |

| Non-ICH | Non-ICH Listings | | | | | | |
|---|---|---|---|---|---|---|---|
| No. in<br>W48 | No. in<br>W96 | No. in<br>EOS | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 56 | 56 | 56 | Safety | 201585/primar<br>y_02/L59 | Listing of Subjects Meeting Hepatobiliary Lab<br>Criteria (Maintenance + Extension Phase) | | W48, W96, EOS |
| 57 | 57 | 57 | Safety | 201585/primar<br>y_02/L57 | Listing of Potential QTc Interval Prolonging<br>Events of Interest | Add Study Period to the 5 <sup>th</sup> Column from the left. | W48, W96, EOS |
| 58 | 58 | 58 | Safety | 201585/primar<br>y_02/L58 | Listing of ECG values for Subjects with<br>Potential QTc Interval Prolonging Events of<br>Interest | | W48, W96, EOS |
| 59 | 59 | 59 | Safety | 201584/primar<br>y_01/L64 | Listing of ALT, AST, Bilirubin (including Total and Direct Bilirubin), INR, and ALP for Subjects Meeting Hepatobiliary Lab Abnormality Criteria | Remove 'Only Q4W IM Subjects are presented in this listing.' from the footnote. | HL, W48, W96,<br>EOS |
| 60 | 60 | 60 | Safety | 201585/primar<br>y_02/L63 | Listing of Investigational Product Exposure Data for Subject Receiving Oral Bridging | | W48, W96, EOS |
| 61 | 61 | 61 | Safety | 201584/primar<br>y_01/L66 | Listing of Dosing Errors and IP Device Malfunctions | | W48, W96, EOS |
| Virology | Virology | | | | | | |
| 62 | 62 | 62 | Confirmed<br>Virologic<br>Failure | 201585/primar<br>y_02/64 | Listing of Replication Capacity in IN and PR/RT Region | Remove 'of Maintenance Phase' from the column header 'Study Day of Maintenance Phase'. | W48, W96, EOS |

# 15.15. Appendix 15: Example Mock Shells for Data Displays

Available upon request